## CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 12-0021 Study Title:

A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Trial to Assess the Safety and Efficacy of 5% Monolaurin Vaginal Gel Administered Intravaginally for the Treatment of Bacterial Vaginosis

Version 1.0

**DATE: 02 NOVEMBER 2017** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

## **Study Title**

| <b>Protocol Number Code:</b> | DMID Protocol: 12-0021 |
|---|---|
| <b>Development Phase:</b> | Phase II |
| Products: | 5% Monolaurin Vaginal Gel |
| Form/Route: | Intravaginally |
| Indication Studied: | Bacterial Vaginosis |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | |
| Clinical Trial Completion Date: | |
| Date of the Analysis Plan: | 02 November 2017 |
| Version Number: | 1.0 |

This study is performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

## TABLE OF CONTENTS

| TABLE OF C | CONTENTS | iii |
|---|---|---|
| LIST OF ABI | BREVIATIONS | vi |
| 1. PREFAC | CE | 8 |
| 2. INTROI | DUCTION | 8 |
| 2.1. Purp | ose of the Analyses | 9 |
| 3. STUDY | OBJECTIVES AND ENDPOINTS | 9 |
| 3.1. Stud | y Objectives | 9 |
| 3.2. End | points | 10 |
| 3.2.1. | Primary Efficacy Outcomes | 10 |
| 3.2.2. | Secondary Efficacy Outcomes | 10 |
| 3.2.3. | Exploratory Efficacy Outcomes | 10 |
| 3.2.4. | Primary Safety Outcomes | 10 |
| 3.2.5. | Secondary Safety Outcomes | 11 |
| 3.3. Stud | y Definitions and Derived Variables | 11 |
| 3.3.1. | Amsel Criteria | 11 |
| 3.3.2. | Bacteriological Cure | 11 |
| 3.3.3. | Clinical Cure | 11 |
| 3.3.4. | Therapeutic cure | 12 |
| 3.3.5. | Recurrent BV | 12 |
| 3.3.6. | First Time BV | 12 |
| 3.3.7. | Baseline Value | 13 |
| 3.3.8. | Test of Cure Visit | 13 |
| 3.3.9. | Treatment Compliance | 13 |
| 4. INVEST | IGATIONAL PLAN | 13 |
| 4.1. Over | rall Study Design and Plan | 13 |
| 4.2. Disc | ussion of Study Design, Including the Choice of Control Groups | 16 |
| 4.3. Sele | ction of Study Population | 16 |
| 4.4. Trea | tments | 19 |
| 4.4.1. | Treatments Administered | 19 |
| 4.4.2. | Method of Assigning Subjects to Treatment Groups (Randomization) | 19 |
| 4.4.3. | Blinding | 20 |

## TABLE OF CONTENTS (continued)

| 4.5. | Effic | cacy and Safety Variables | 20 |
|---|---|---|---|
| 5. S | AMPL | E SIZE CONSIDERATIONS | 21 |
| 6. ( | SENER | AL STATISTICAL CONSIDERATIONS | 22 |
| 6.1. | Gen | eral Principles | 22 |
| | 6.1.1. | Pseudo Code | 23 |
| 6.2. | Tim | ing of Analyses | 23 |
| 6.3. | Ana | lysis Populations | 24 |
| | 6.3.1. | Intent-to-Treat Analysis (ITT) Population | 24 |
| | 6.3.2. | Safety Analysis Population | 24 |
| | 6.3.3. | Modified Intention-to-Treat (mITT) Population | 24 |
| | 6.3.4. | Evaluable Population | 24 |
| | 6.3.5. | Per Protocol Population | 24 |
| 6.4. | Cov | ariates and Subgroups | 25 |
| 6.5. | Miss | sing Data | 25 |
| 6.6. | Inte | im Analyses and Data Monitoring | 26 |
| 6.7. | Mul | ticenter Studies | 26 |
| 6.8. | Mul | tiple Comparisons/Multiplicity | 27 |
| 7. S | TUDY | SUBJECTS | 27 |
| 7.1. | Sub | ect Disposition | 27 |
| 7.2. | Prot | ocol Deviations | 27 |
| 8. E | EFFICA | CY EVALUATION | 27 |
| 8.1. | Prin | nary Efficacy Analysis | 28 |
| 8.2. | Seco | ondary Efficacy Analyses | 28 |
| 8.3. | Exp | loratory Efficacy Analyses | 29 |
| 9. S | AFET | Y EVALUATION | 30 |
| 9.1. | Den | nographic and Other Baseline Characteristics | 30 |
| | 9.1.1. | Concurrent Illnesses and Medical Conditions | 30 |
| 9.2. | Mea | surements of Treatment Compliance | 30 |
| 9.3. | Adv | erse Events | 31 |
| | 9.3.1. | Solicited Events and Symptoms | 32 |
| | 9.3.2. | Unsolicited Adverse Events | 33 |
| 9.4. | Dea | ths, Serious Adverse Events and other Significant Adverse Events | 34 |

## TABLE OF CONTENTS (continued)

| 9.5. Pregnancies | 34 |
|---|---|
| 9.6. Clinical Laboratory Evaluations | 35 |
| 9.7. Physical Evaluations | 36 |
| 9.8. Concomitant Medications | 36 |
| 10. OTHER ANALYSES | 36 |
| 11. REPORTING CONVENTIONS | 36 |
| 12. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED A | ANALYSES37 |
| 13. TECHNICAL DETAILS | 37 |
| 14. REFERENCES | 37 |
| 15. LISTING OF TABLES, FIGURES, AND LISTINGS | 38 |
| 16. APPENDICES | 39 |
| Appendix I: Table Mock-Ups | 39 |
| Section 14.1 Demographic Data | 44 |
| Section 14.2 Efficacy Data | 69 |
| Section 14.3 Safety Data | 85 |
| Section 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events | 107 |
| Appendix II: Figure Mock-Ups | 120 |
| Appendix III: Listings Mock-Ups | 137 |
| Appendix IV: Clinical Lab Reference Ranges | 166 |

## LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|-------------------------------------------------------------------|
| AGUS | Atypical glandular cells of uncertain significance |
| ALT | Alanine Aminotransferase |
| ASCUS | Atypical squamous cells of undetermined significance HPV negative |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Classification |
| BV | Bacterial Vaginosis |
| CDC | Centers for Disease Control and Prevention |
| CI | Confidence Interval |
| CIN | Cervical intraepithelial neoplasia |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| EDC | Electronic Data Capture |
| ER | Emergency Room |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| GML | Glycerol monolaurate |
| HEENT | Head, Ears, Eyes, Nose, and Throat |
| HIV | Human Immunodeficiency Virus |
| HSIL | High grade Squamous Intraepithelial Lesion |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| ITT | Intention to Treat |
| kg | kilogram |
| КОН | Potassium Hydroxide |
| L | Liter |
| LLN | Lower Limit of Normal |
| LOCF | Last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |

## LIST OF ABBREVIATIONS (continued)

| mg | Milligram |
|------|------------------------------------------|
| mITT | Modified Intention to Treat |
| mL | Milliliter |
| N | Number (typically refers to subjects) |
| NAAT | Nucleic Acid Amplification Test |
| NF | National Formulary |
| NIH | National Institutes of Health |
| pН | Potential of Hydrogen |
| PI | Principal Investigator |
| PP | Per Protocol |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamate pyruvate transaminase |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| TOC | Test of Cure |
| U | Units |
| ug | microgram |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cell |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Trial to Assess the Safety and Efficacy of 5% Monolaurin Vaginal Gel Administered Intravaginally for the Treatment of Bacterial Vaginosis" (Division of Microbiology and Infectious Diseases (DMID) Protocol 12-0021) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA) and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for efficacy and safety outcomes, and (4) a list of proposed tables and figures. Any deviation from this SAP will be described and justified in the CSR. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Bacterial Vaginosis (BV) is a disorder of the chemical and biological balance of the normal vaginal flora [1]. In women of childbearing age, BV is the most common cause of vaginitis accounting for 22-50% of women who have symptoms of vaginitis [2]. In a cohort of young healthy women, nearly 30% had been treated for BV [3]. The diagnosis of BV has been based clinically on Amsel and Nugent scoring criteria using direct Gram stain of vaginal secretions. The Centers for Disease Control and Prevention (CDC) recommends metronidazole 500 mg orally twice daily for 7 days, intravaginal metronidazole gel 0.75% once daily for 5 days or clindamycin cream 2% intravaginally once daily for 7 days as first line therapy for BV [1]. However, up to 30% of women will have recurrent BV within 3 months of therapy [4]. Given BV's high recurrence rates and the risks for antimicrobial resistance, additional treatment options are desirable.

Monolaurin, also commonly referred to as glycerol monolaurate (GML), is a monoglyceride surfactant. It is an ester formed from glycerol and lauric acid. This formulation promotes rapid drug distribution, as well as adequate coverage, throughout the vaginal cavity. The acidic pH keeps monolaurin in its non-ionized form in the vagina. Monolaurin, which is practically insoluble in water, is highly soluble in this formulation. Laboratory studies have shown that Monolaurin has antibacterial, antifungal and antiviral properties. Monolaurin's mechanism of

action of blocking signals at the pathogen's plasma membrane provides an advantage over other antibiotics with regard to the development of resistance [5, 6]. Information on dosage forms can be found in Section 6 of the protocol.

New therapies for BV are needed and 5% Monolaurin Vaginal Gel has the potential to eradicate flora associated with BV while maintaining some of the normal flora that is considered protective for vaginal health, and with the added potential of preventing the emergence of vaginal candidiasis. This phase II study is designed to evaluate the safety of 5% Monolaurin Vaginal Gel compared to placebo gel and provide an early assessment of efficacy in treatment of women with BV. The July 2016 FDA draft guidance was used in the development of the study design.

## 2.1. Purpose of the Analyses

The analyses contained in this Statistical Analysis Plan will assess the safety and efficacy of 5% Monolaurin Vaginal Gel in comparison with Vehicle Placebo Gel and will be included in the clinical study report.

The protocol for DMID 12-0021 calls for a planned interim analysis to reassess the adequacy of the sample size based on subjects meeting eligibility for the Modified Intent-to-Treat (mITT) population. After eighty subjects have been enrolled and have available baseline test results for Nugent score, Human Immunodeficiency Virus (HIV), chlamydia and gonorrhea, the fraction of subjects enrolled to date who are eligible for the mITT cohort will be estimated. The tables and figures for the interim analysis are contained in the Data Safety Monitoring Board (DSMB) Interim Analysis Safety Summary Report Table and Figure Shells. The goal of the interim analysis is to review aggregate enrollment data in order to recommend whether an extension to the trial is necessary, while it is still possible to do so without halting enrollment and losing momentum in subject accrual.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

## 3.1. Study Objectives

**Primary Objectives** 

- To assess the safety and tolerability of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel (excipients only).
- To assess the efficacy by clinical cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visit 2.

#### Secondary Objectives

- To evaluate the therapeutic cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visits 2 and 3.
- To evaluate the clinical cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visit 3.
- To evaluate the changes in Nugent's criteria of vaginal bacterial flora at Visits 2 and 3.

#### **Exploratory Objectives**

- To evaluate the clinical and therapeutic cure rates of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel for each subgroup (first episode BV and recurrent BV) at Visits 2 and 3.
- To evaluate quantitative changes in selected bacterial species at Visits 2 and 3.
- To evaluate the quantitative changes of *Candida spp*. (in subjects with *Candida spp*. identified at screening) at Visits 2 and 3.

## 3.2. Endpoints

## 3.2.1. Primary Efficacy Outcomes

The primary efficacy outcome is assessed overall and in both treatment arms and is as follows:

1. Proportion of subjects with clinical cure in each study arm at Visit 2 (Day 8-15).

See Section 3.3 for definition of clinical cure.

#### 3.2.2. Secondary Efficacy Outcomes

- 1. Proportion of subjects with therapeutic cure in each study arm at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31).
- 2. Proportion of subjects with Nugent score of 3 or less (negative for BV) and 4-6 (intermediate) in each study arm at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31).
- 3. Proportion of subjects with clinical cure in each study arm at Visit 3 (Day 22-31).

See section 3.3 for definition of therapeutic cure.

#### 3.2.3. Exploratory Efficacy Outcomes

- 1. Proportion of subjects with clinical cure in each study arm by subgroup (first time or recurrent infection) by Visit 2 (Day 8-15) and by Visit 3 (Day 22-31).
- 2. Proportion of subjects with therapeutic cure in each study arm by subgroup (first time or recurrent infection) by Visit 2 (Day 8-15) and by Visit 3 (Day 22-31).
- 3. Mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.*, respectively, in each study arm at baseline, Visit 2 (Day 8-15) and at Visit 3 (Day 22-31).
- 4. Mean fungal colony count in vaginal secretions in each study arm at baseline, at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31).

See Section 3.3 for cure definitions.

#### 3.2.4. Primary Safety Outcomes

- 1. Number of subjects reporting solicited urogenital adverse events (AEs) following the first dose of the study product through Visit 2 (Day 8-15).
- 2. Number of subjects reporting serious adverse events (SAEs) considered product-related following the first dose of the study product through Visit 3 (Day 22-31).

#### 3.2.5. Secondary Safety Outcomes

- 1. Number of subjects experiencing non-laboratory, non-solicited AEs following the first dose of the study product through Visit 3 (Day 22-31).
- 2. Number of subjects experiencing laboratory AEs following the first dose of the study product through Visit 2 (Day 8-15).

## 3.3. Study Definitions and Derived Variables

#### 3.3.1. Amsel Criteria

During gynecologic examination, any three of the following will be used for the clinical diagnosis of BV by Amsel Criteria:

- a. Off-white (milky or gray), thin, homogenous discharge with minimal or absent pruritus or inflammation of the vulva or vagina.
- b. ≥20% "Clue" cells of total epithelial cells on microscopic examination of saline wet mount.
- c. Vaginal secretion pH >4.5.
- d. Positive "whiff test."

#### 3.3.2. Bacteriological Cure

A vaginal swab for bacteriological assessment of BV by Nugent criteria will be performed. The Nugent score utilizes a 10-point scale for evaluation of vaginal flora. The Nugent score can range from 0 to 10. A score of 7 to 10 is consistent with BV while 4-6 is considered intermediate and 0-3 is negative for BV. Bacteriological cure of BV is defined as a normal Nugent score of 0-3. Laboratory examination of vaginal smears and the determination of the Nugent score is as follows:

| N Score = The sum of the scores for each bacterial morphotype listed below. (Note: Number of Organisms seen/high power field as determined by averaging a representative field by two independent evaluators) | | | | | | |
|---|---|---|---|---|---|---|
| Lactobacilli | SCORE | Gardnerella,<br>Bacteroides | SCORE | Curved gram-negative<br>bacilli | SCORE | Sum=<br>*N SCORE |
| ≥30 | 0 | 0 | 0 | 0 | 0 | 0 |
| <30-5 | 1 | <1 | 1 | <1 | 1 | 3 |
| <5-1 | 2 | 1 to <5 | 2 | 1 to <5 | 1 | 5 |
| <1 | 3 | 5 to <30 | 3 | 5 to <30 | 2 | 8 |
| 0 | 4 | ≥30 | 4 | ≥30 | 2 | 10 |

#### 3.3.3. Clinical Cure

A clinical cure is defined by normal Amsel criteria. Normal Amsel criteria are defined as: normal physiological vaginal discharge, whiff test negative for any amine "fishy" odor, saline wet mount

less than 20% for clue cells, and vaginal pH is <=4.5. All four criteria must be normal and none of the clinical failure criteria listed below can be met to be considered a clinical cure.

A clinical failure is defined by at least one of the following:

- a. one or more abnormal Amsel criteria,
- b. early discontinuation of study therapy due to lack of treatment effect,
- c. use of any vaginosis therapy or systemic antimicrobial therapy other than study product during the study, or
- d. in the investigator's opinion, requires additional treatment for vaginosis.

Subjects who do not have enough information to determine a clinical cure or clinical failure status will not be evaluable for clinical cure.

#### 3.3.4. Therapeutic cure

Therapeutic cure is defined as both a clinical cure and a bacteriological cure.

Subjects who were clinical failures, or have a Nugent score >3 are therapeutic failures.

All other subjects will be considered not evaluable for therapeutic cure. See the table below for therapeutic cure outcome determinations.

| If the clinical cure outcome is | and the Nugent<br>(bacteriological)<br>score result is | then the overall<br>therapeutic cure<br>outcome is |
|---|---|---|
| Cure | 0-3 | Cure |
| Cure | >3 | Failure |
| Cure | Not Evaluable | Not Evaluable |
| Failure | 0-3 | Failure |
| Failure | >3 | Failure |
| Failure | Not Evaluable | Failure |
| Not Evaluable | 0-3 | Not Evaluable |
| Not Evaluable | >3 | Failure |
| Not Evaluable | Not Evaluable | Not Evaluable |

All cure related outcomes are assessed at follow-up Visits 2 and 3.

#### 3.3.5. Recurrent BV

Recurrent BV infection is defined as 2 or more episodes of BV in the previous 12 months, including the subject's current episode, as reported by the subject in the sexual history interview.

#### 3.3.6. First Time BV

First time BV infection is defined as one episode of BV in the previous 12 months including the subject's current episode, as reported by the subject in the sexual history interview.

#### 3.3.7. Baseline Value

The baseline value is defined as the last value obtained prior to the first dose of study product.

#### 3.3.8. Test of Cure Visit

The Test of Cure (TOC) visit is Visit 2, Day 8-15. For the ITT, mITT, and Evaluable analysis populations, if a subject is evaluable for clinical cure, even if they return outside of the 8 to 15-day window, their results will be included in the Test of Cure Visit 2 efficacy analyses. Subjects who return outside of the 8 to 15-day window will be excluded from the Per-Protocol analysis population. Similarly, if a subject does not have an assessment at Visit 2, but returns for an unscheduled Visit 2, the data collected at the unscheduled visit will be used for Visit 2 assessments. This applies for all tables that present data by study visit. See Section 6.3 for more details.

#### 3.3.9. Treatment Compliance

Compliance is assessed by the study coordinator's count of used/unused applicators in each returned subject kit. If a kit is not returned, compliance will be assessed by the subject's self-report on the memory aid. If an incomplete kit is returned, the subject's self-report will be used in conjunction with the count of used/unused applicators to determine subject compliance. In addition to the count of used/unused applicators, the timing of dosing will be considered. Subjects are instructed to administer study product twice daily (morning and evening) with at least 8 hours between doses. If the subject received her first dose after 3 pm, she will be instructed to administer the next dose the following morning. A subject is compliant if she uses at least 5 of 6 doses and they were administered within 72 hours from the first dose, at least 8 hours apart, and if no more than 2 doses in a 24 hour period are taken.

#### 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

This is a Phase 2, double-blind, randomized, placebo-controlled, multi-center trial comparing 5% Monolaurin Vaginal Gel to Vehicle Placebo Gel as outpatient therapy. A total of 120 eligible subjects with BV will be enrolled. Treatment assignments will be randomly allocated in a 2:1 ratio of test article to placebo, with the randomization stratified by clinical site. Each subject will receive intravaginal gel twice daily for three successive days for a total of 6 doses. There will be 3 clinic visits over 31 days.

The primary study objectives are to compare 5% Monolaurin Vaginal Gel with vehicle placebo gel (excipients only) with respect to safety and tolerability, and efficacy by clinical, bacteriological, and therapeutic cure. Treatment response is evaluated at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31).

The DSMB met after 30 subjects received at least one dose of study drug and completed Visit 2. The DSMB may also review study progress and subject safety data at other specified times during the course of the study and hold a study closeout meeting, as defined in the DSMB Charter.

Additionally, a single, fully blinded interim analysis occurred to reassess the adequacy of the sample size based on subjects meeting eligibility for the mITT population. After eighty subjects had been enrolled and had available baseline test results for Nugent score, HIV, chlamydia and gonorrhea, the fraction of subjects enrolled to date who were eligible for the mITT cohort was estimated. See Section 6.6 for more details.

The figure below presents the schematic of the study design.



Baseline clinical information is collected on all subjects at the screening/enrollment visit (Day 1). This information consists of demographics, medical and sexual history, including number of episodes of BV in the past year, concomitant medications review, and a physical exam including a gynecological exam.

Vaginal swabs are taken to perform a KOH test, vaginal pH, and to review a wet prep. Vaginal swabs for Gram stain of vaginal smear, and assessment for *Candida spp.*, selected bacterial species, *Trichomonas vaginalis, Chlamydia trachomatis*, and *Neisseria gonorrhoeae* are collected.

Blood samples are collected for safety assessments (HIV, White Blood Cell [WBC] count, hemoglobin, platelets, neutrophil count, creatinine, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, random glucose).

All subjects are provided with a 5-day memory aid to aid in their recall of local solicited events. **Table 1** below presents the schedule of events at each visit.

**Table 1:** Schedule of Events

| | Visit 1 | Visit 2 | Visit 3 | rly<br>nation | duled |
|---|---|---|---|---|---|
| | Day 1 | 8<br>(Window Days<br>8-15) | 28<br>(Window Days<br>22-31) | Early X X X X X X X X X X X X X X X X X X X | Unscheduled |
| Informed Consent | X | | | | |
| Inclusion/Exclusion | X | | | | |
| Demographics | X | | | | |
| Medical History | X | | | | |
| Concomitant Medication | X | X | X | X | X |
| Intercurrent Medical History | 71 | X | X | ł | X |
| Physical Exam | X | | | | |
| Targeted Physical Exam | | {X} | {X} | {X} | |
| Urine Pregnancy Test | X | | | | |
| Gynecological Exam 3 | X | X | X | X | $X^{\dagger}$ |
| Vaginal Swabs for Nugent Score, bacterial/fungal cultures, trichomonas testing and appropriate samples for gonorrhea, | X | X | X | X | $\chi^{\dagger}$ |
| Chlamydia testing Vaginal Swab for Future Use (if subject consents to future use sample collection) | X | X | X | X | |
| Randomization | X | | | | |
| Study Drug Administration <sup>5</sup> | X | | | | |
| Distribute Memory Aid and Study Drug Kit | X | | | | |
| Counsel on intravaginal products, objects, sexual intercourse, and pregnancy avoidance | X | X | | | |
| Safety Labs <sup>6</sup> | X | X | X^ | X | |
| Telephone Contact to Stop Study Treatment | [X] | | | | |
| Review Vaginal Symptomology | X | X | X | X | X |
| Review for insertion of intravaginal products, objects, and sexual intercourse | | X | X | X | |
| Review Memory Aid and Collect Study Drug Kit | | X | $\chi^{+}$ | X | |
| Assessment of Clinical Cure | | X | X | X | |
| Assessment of Therapeutic Cure | | X | X | X | |
| AE/SAE | X | X | X | X* | X |

<sup>&</sup>lt;sup>1</sup> Include menstrual, contraceptive, sexual history and history of previous episodes of vaginitis.

<sup>&</sup>lt;sup>2</sup> Include use of intravaginal products or objects, sexual intercourse, treatment for vaginitis (other than the study product).

<sup>&</sup>lt;sup>3</sup> Evaluate cervix, vagina, and vulva. Perform Vaginal pH, Saline Wet Mount, KOH Wet Mount, "Whiff Test".

<sup>&</sup>lt;sup>4</sup> Collect vaginal swabs for study specific tests (gram stain, cultures for bacterial flora and yeast) and trichomonas OSOM testing (if saline wet mount is negative, Visit 1 only) and institution specific samples for culture or molecular testing for *Chlamydia*, *Neisseria* gonorrheae. (Visit 1 only). Samples for gonorrhea and chlamydia testing will be consistent with standard of care at the institution).

<sup>&</sup>lt;sup>5</sup> Provide instructions on proper use of study drug applicator and observe first dose. Remaining 5 doses will be administered by the subject at home on Day 2 and Day 3.

<sup>&</sup>lt;sup>6</sup> Safety Laboratories Include: White blood cell count, hemoglobin, platelet count, absolute neutrophil count, creatinine, ALT, AST, total bilirubin, random glucose, HIV test (*Visit 1 only*).

<sup>{ }</sup> Targeted physical examination if indicated based on review of symptoms.

## 4.2. Discussion of Study Design, Including the Choice of Control Groups

Subjects are randomized at a ratio of 2:1 to receive 5% Monolaurin Vaginal Gel or Vehicle Placebo Gel, which has the same formulation except not containing 5% GML, administered vaginally morning and night for 6 consecutive doses (3 days). The July 2016 FDA draft guidance was used in the development of the study design.

## 4.3. Selection of Study Population

Subjects may have asymptomatic BV, but must meet any three of the four Amsel criteria for BV as defined in Section 3.3.

Subjects must meet all of the following inclusion criteria to participate in this study:

- 1. Non-pregnant, non-breastfeeding females between the ages of 18 and 50 years, inclusive.
- 2. Women of childbearing potential\* must agree to practice reliable contraception\*\* for the 28-day period before enrollment through 30 days following treatment.
  - \*(not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy, or who have not been postmenopausal for  $\geq 1$  year)
  - \*\*Acceptable birth control methods for the purposes of this study may include, but are not limited to, abstinence from intercourse with a male partner, monogamous relationship with vasectomized partner, barrier methods to include condoms and diaphragms, intrauterine devices, and licensed hormonal methods. NuvaRing® contraceptive use will be prohibited from this study since the device can alter vaginal secretions.
- 3. Presenting with signs of BV (as per Amsel Criteria). Subjects must meet any three of the four criteria for enrollment\*
  - \*Presence of discharge, greater than or equal to 20% clue cells on wet prep, positive "whiff test" on KOH prep, vaginal pH of greater than 4.5.
- 4. Not currently menstruating or expected to in the next 4 days.
- 5. Able to understand and comply with planned study procedures.
- 6. Willing to abstain from sexual intercourse, insertion of tampons, douches, or other intravaginal medications or objects between Visit 1 and Visit 2 and 48 hours prior to Visit 3.

<sup>[]</sup> Subjects will be called regarding grade 3 laboratory abnormalities within 24 hours of receipt of results and told to discontinue study product. Subjects with positive HIV, chlamydia or gonorrhea tests will be contacted as soon as possible after results are available and referred to their primary care provider for appropriate treatment.

<sup>&</sup>lt;sup>+</sup> Memory Aid will be reviewed *only* if solicited events continued at Visit 2. Study Drug Kit returned *only* if not returned at Visit 2.

<sup>\*</sup> If subject declines to return for an in-person visit, the study personnel will ask to contact the subject by telephone to assess for AE/SAEs on Day 22-31.

<sup>†</sup> Evaluate cervix, vagina, and vulva. Collect appropriate clinical samples for genital infectious pathogens.

<sup>&</sup>lt;sup>#</sup> Assess for vaginal discharge (quantity, color, odor, and consistency) and record presence or absence of objective signs of inflammation of cervix, vagina, and vulva (edema, erythema, excoriation).

<sup>^</sup> Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 should be repeated until resolved or has stabilized. Further testing beyond Visit 3 is at the discretion of the PI or study investigator.

- 7. Provide written informed consent before initiation of any study procedures and be available for all study visits.
- 8. No known history of HIV.

Subjects are not able to participate if they meet any of the following exclusion criteria:

- 1. Signs or symptoms of vaginal/cervical/pelvic infection on screening or clinical diagnosis of vaginal/cervical/pelvic infection in the past 14 days.
  - \*(including but not limited to yeast vulvovaginitis, chlamydia, gonorrhea, trichomonas, genital ulcer disease, pelvic inflammatory disease). Self-treatment for presumed yeast vaginitis is not an exclusion if treatment was discontinued 7 days or greater prior to enrollment.
- 2. Treatment for BV within the past 14 days.
- 3. Cervical or vaginal high grade squamous intraepithelial dysplasia (HSIL), atypical glandular cells of uncertain significance (AGUS) or cervical intraepithelial neoplasia grade 2 (CIN2) or higher\*
  - \*Atypical squamous cells of undetermined significance (ASCUS), low grade squamous intraepithelial lesion (LSIL) or cervical intraepithelial neoplasia grade 1 (CIN1) are acceptable. Individuals with a history of atypical glandular cells of uncertain significance (AGUS), HSIL or CIN2 and who have received subsequent evaluation and/or treatment with follow up normal PAP smear are eligible. Patient report will be accepted.
- 4. History of undiagnosed vaginal bleeding.
- 5. Use of a systemic, vaginal, or perineal antibiotic within 7 days prior to enrollment in this study.
- 6. Use of an immunosuppressive or immunomodulatory drug\* for two or more consecutive weeks within 6 months prior to enrollment
  - \*such as >0.5 mg/kg/day or  $\ge 20$  mg total dose/day of prednisone orally or > 800  $\mu g$  of inhaled beclomethasone (nasal and non-genital topical steroids are allowed).
- 7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Monolaurin Vaginal Gel.
- 8. Uncontrolled concurrent illness\*. Subjects with a history of organ or marrow transplant are excluded.
  - \*Including, but not limited to, ongoing or active infection, active liver, kidney or autoimmune diseases (a history of thyroid disease will be permitted as long as the thyroid disease is now stable), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 9. Acute illness within 3 days before receipt of study product (per investigator's discretion).
- 10. Pregnant women and women who are planning to become pregnant within 30 days after the final study dose, or women who are breastfeeding.
- 11. Immunosuppression as a result of an underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.

- 12. Active neoplastic disease\* or a history of any hematologic malignancy. Active neoplastic disease is defined as neoplastic disease or treatment for neoplastic disease within the past 5 years.
  - \*(excluding non-melanoma skin cancer)
- 13. Received an experimental agent\* within 30 days before receipt of study product or expect to receive an experimental agent during the 1-month study period.
  - \*(vaccine, drug, biologic, device, blood product, or medication)
- 14. Any condition that would place the subject at an unacceptable risk of injury, render her unable to meet the requirements of the protocol, or that may interfere with successful completion of the study.
- 15. A history of alcohol or drug abuse\* during the previous 1 year that in the opinion of the site investigator would interfere with study procedures
  - \*For example, daily excessive alcohol use or frequent binge drinking as determined by the investigator, or daily marijuana use.

Any enrolled subject may withdraw or be withdrawn from the study for the following reasons:

- The subject withdraws consent.
- The study is terminated.
- For any reason that, in the opinion of the investigator, precludes the subject's participation in the study.
- The subject no longer meets inclusion/exclusion criteria.
- The subject develops an SAE that warrants withdrawal.
- Other safety-related reasons at the discretion of the Principal Investigator (PI), DMID Medical Monitor, DSMB, or the subject.

Any subject who has received at least one dose of study drug is continued in efficacy and safety follow-up, if the subject agrees.

Subjects who test positive for chlamydia, gonorrhea, HIV, or are incidentally found to have a PAP result consistent with AGUS or HSIL, or have a Grade 3 laboratory abnormality are discontinued from receiving study product if the result is available within the 3 days of study drug administration. They are continued in follow up for safety and efficacy if they have received one dose of study drug. (PAP smears are not part of the study protocol, but may have been done outside of the study protocol by the subject's provider. Patient report of PAP smear abnormalities may be accepted as a criterion for discontinuation of study product).

If a subject develops a grade 3 laboratory abnormality while still receiving study product, they are contacted and asked to discontinue study product and are continued in safety and efficacy follow up. If any subject experiences a severe AE related to the study product, further doses are discontinued. Additionally, subjects who experience a new or worsening solicited reactogenicity symptom that is grade 2 or higher are asked to contact the study site to confirm the severity. A determination is made whether to continue or discontinue the study product by a licensed study clinician. A subject who withdraws voluntarily from or has been discontinued from receiving

further treatment is encouraged to permit continued follow-up of AEs and to follow scheduled visits. If the subject agrees, study procedures (e.g., blood sampling for safety and vaginal sampling) are continued.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

#### 5% Monolaurin Vaginal Gel

Monolaurin Vaginal Gel is a clear and colorless non-sterile glycol-based gel for vaginal administration. Monolaurin Vaginal Gel is comprised of 5% monolaurin and the following excipients:

Active test article is comprised of 5% monolaurin prepared as pre-filled vaginal gel applicators of identical likeness to placebo. The components of the applicator are biocompatible and latex-free.

#### Vehicle Placebo Gel

The Vehicle Placebo Gel is a clear to opaque, colorless to light gray, non-sterile glycol-based gel for vaginal administration and contains the following:

. The Vehicle Placebo Gel contains the same excipients as the active product.

The Vehicle Placebo Gel is comprised of the identical vehicle contained in the active test article prepared as pre-filled vaginal gel applicators of identical likeness to active test article. The components of the applicator are biocompatible and latex-free.

The first dose of Monolaurin Vaginal Gel or Vehicle Placebo Gel is administered by the subject while the subject is still in clinic. The remaining 5 doses are administered twice daily (morning and evening), with at least 8 hours between doses by the subject at home. If the subject receives her first dose after 3 p.m., she is instructed to administer the next dose the following morning.

#### 4.4.2. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment of subjects is done online using the enrollment module of AdvantageEDC<sup>SM</sup>. Subjects are randomly assigned to active drug or placebo in a 2:1 ratio. The study uses a stratified, permuted blocked randomization scheme. Permuted block randomization is used to avoid the potential for serious imbalance in the number of subjects assigned to each group during the study, an imbalance that can occur in the simple randomization procedures. Stratification is by clinical site.

The randomization is prepared by statisticians at the Statistical and Data Coordinating Center (SDCC) and included in the enrollment module for the trial. AdvantageEDC assigns each subject to a treatment group after the demographic and eligibility data have been entered into the system.

The vaginal gel applicators are packaged as a kit sufficient for twice daily administration for 3 consecutive days (six applicators). Random kit numbers are provided to Fisher, the investigational product distributor, in order to ensure the associated sets of applicators are filled with the same contents (placebo or active) without unblinding the sites to what treatment is in

each kit once the shipments arrive. Each vaginal gel dispensing kit is individually labeled with the kit number. Once a subject is assigned a randomization number, a kit corresponding to the assigned treatment is distributed to the subject.

#### 4.4.3. Blinding

A designated individual at each site is provided with a treatment key, which links the treatment code to the actual treatment assignment, which is kept in a secure place.

The applicators of vaginal gels are selected by the unmasked Site Research Pharmacist or designated unmasked study personnel and are distributed to masked study personnel with no labels that identify the product or applicators to the site as Monolaurin Vaginal Gel or Vehicle Placebo Gel.

The volunteers, the study personnel who perform study assessments after administration, data entry personnel at the sites, and laboratory personnel are masked to treatment assignment. The DSMB may receive data in aggregate and presented by treatment group. The DSMB may be unmasked to individual study treatment assignments, as needed, to adequately assess safety issues.

For the interim analysis, the blind was maintained when reporting results prepared for the DSMB meeting.

## 4.5. Efficacy and Safety Variables

Subject assessment of solicited urogenital adverse events constitutes a primary safety endpoint. Solicited event assessments were captured on a memory aid starting on Day 1, the first day of therapy and continuing for 5 days. The subject was to record the presence and intensity of vulvovaginal solicited events on the memory aid. Any symptom that was present at the time that the subject was screened should have been considered as baseline and not reported as a solicited urogenital AE. However, if the symptom deteriorated at any time during the study, it was to be recorded as an AE. If a symptom was reported that was not present at baseline, it too was to be recorded as an AE. Any symptoms still present on Day 5 were continued to be followed by subject memory aid notations until symptom resolution. Solicited events include vaginal odor, vaginal pain, vaginal tenderness, vulvar/vaginal itching, vaginal dryness, vaginal discharge, and vulvar inflammation. Severity of solicited events symptoms are graded according to the table in Appendix C in the protocol. Symptoms not specifically mentioned will be graded using the following scale:

- Grade 1: Mild (does not interfere with activity)
- Grade 2: Moderate (interferes with activity)
- Grade 3: Severe (prevents daily activity)

Clinical laboratory evaluations constitute a secondary safety endpoint. Hematology includes: WBC count, hemoglobin, platelets, and neutrophil count. Clinical chemistry includes: creatinine, AST (SGOT), ALT (SGPT), total bilirubin, and glucose (random). Grade 3 abnormal laboratory values were to be repeated within 10 days. Laboratory abnormalities that were stable at Visit 2 were not repeated at Visit 3. Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 were repeated at Visit 3. A laboratory abnormality is considered an

adverse event if there was a worsening of the laboratory value at Visit 2 from the baseline value and it increased in laboratory toxicity grading from the baseline toxicity grading. For laboratory abnormalities repeated at Visit 3, if there was a worsening of the laboratory value at Visit 3 from the Visit 2 value and it increased in laboratory toxicity grading, it was considered an additional adverse event.

Multiple observations within a specific visit period are accepted. In the case of multiple observations within a specific window, the assessment value that is closest to the scheduled visit window will be used in the analyses for the post-baseline records. For screening and baseline visits, the last assessment value prior to first dose will be used as the baseline measurement. All the recorded data will be listed. If observations have the same distance to the scheduled assessment, the latest one will be used.

Culture counts for following bacterial and yeast species will be collected: Lactobacillus, Gardnerella, Mobiluncus, and Candida. Nugent score and Budding yeast will be reported from the Gram Stain. Budding yeast will be categorized as Few, Moderate, Many, or No organisms seen

See Section 3.3 for efficacy variable definitions.

#### 5. SAMPLE SIZE CONSIDERATIONS

The statistical informational goal for the study is 90 subjects eligible for the primary efficacy analysis of clinical cure in the modified Intent-to-Treat (mITT) efficacy population. This is an ad-hoc sample size determined by logistical and feasibility considerations, as there is insufficient pilot data upon which to base more formal sample size calculations.

Subjects who did not meet all inclusion/exclusion criteria, who have a Nugent score <4 at Visit 1 or are positive for other concomitant vulvovaginal infections at baseline which may interfere with the efficacy assessment will be excluded from the mITT population.

Based on observed rates of these outcomes at the participating clinics, it is anticipated that a total of 120 subjects will be enrolled to reach this target. However, enrollment will be continued past 120 subjects to a maximum of 150, if necessary, to reach the informational goal of 90 eligible subjects.

The table below shows the statistical power conferred by this sample size for a two-sided significance level 5% Fisher's exact test comparing binomial proportions, under different assumed proportions.

Power to compare binomial proportions using a two-sided significance level 0.05 Fisher's Exact Test with a sample size of N = 90 (60 subjects in the 5% Monolaurin Vaginal Gel arm, 30 subjects in the Vehicle Placebo Gel arm) is shown below. Conditions in which Power is  $\geq$ .80 are highlighted.

| | | | | 5% | 6 Monol | aurin Va | ginal G | el (N=60 | )) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | .05 | .10 | .20 | .30 | .40 | .50 | .60 | .70 | .80 | .90 | .95 |
| | .05 | .02 | .04 | .38 | .82 | .97 | >.99 | >.99 | >.99 | >.99 | >.99 | >.99 |
| (=30) | .10 | .13 | .03 | .15 | .52 | .85 | .98 | >.99 | >.99 | >.99 | >.99 | >.99 |
| el (N | .20 | .53 | .22 | .03 | .12 | .42 | .78 | .96 | >.99 | >.99 | >.99 | >.99 |
| Vehicle Placebo Gel (N=30) | .30 | .86 | .61 | .15 | .03 | .12 | .41 | .76 | .95 | >.99 | >.99 | >.99 |
| lacel | .40 | .98 | .89 | .47 | .13 | .04 | .13 | .41 | .76 | .96 | >.99 | >.99 |
| le P | .50 | >.99 | .98 | .79 | .42 | .13 | .04 | .13 | .42 | .79 | .98 | >.99 |
| ehic | .60 | >.99 | >.99 | .96 | .76 | .41 | .13 | .04 | .13 | .47 | .89 | .98 |
| > | .70 | >.99 | >.99 | >.99 | .95 | .76 | .41 | .12 | .03 | .15 | .61 | .86 |
| | .80 | >.99 | >.99 | >.99 | >.99 | .96 | .78 | .42 | .12 | .03 | .22 | .53 |
| | .90 | >.99 | >.99 | >.99 | >.99 | >.99 | .98 | .85 | .52 | .15 | .03 | .13 |
| | .95 | >.99 | >.99 | >.99 | >.99 | >.99 | >.99 | .97 | .82 | .38 | .04 | .02 |

With respect to the safety objectives, for a sample size of 60 subjects in the treatment arm with no observed SAEs related to study product, the 95% confidence interval (CI) for the estimated proportion is (.00,.06) (Clopper-Pearson interval).

In actuality, the safety analysis cohort will be larger than the mITT cohort, and the CI will be more precise than this.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

## **6.1.** General Principles

Tabulations will be used extensively to summarize the data. All continuous variables will be summarized using the following descriptive statistics: n (sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the sample size) of observed levels will be reported for all categorical measures. Wilson confidence intervals for binomial proportions and differences in binomial proportions will be computed for efficacy variables. Clopper-Pearson confidence intervals for binomial proportions and differences in binomial proportions will be computed for safety variables. In general, all data will be listed by treatment group and/or subject, and when appropriate by visit number within subject.

All summary tables will be structured with a column/sub-table for each treatment group (5% Monolaurin Vaginal Gel, Placebo Gel, and All Subjects). The total population size relevant to that table/column if applicable, including any missing observations will be displayed in the tables.

Note that in the data listings, Subject ID is the unique subject identifier, not the Study ID used on study and dates will not be included, only Study Day. Study Day 1 will be the day of the first dose of treatment.

#### 6.1.1. Pseudo Code

The following SAS® peudo code will be used to calculate the following:

Fisher's Exact test:

```
proc freq;
  Table treatment*analysis variable / exact;
   ods output FishersExact=outputdsn1;
run;
95% Wilson CI for proportions/percents:
Proc freq;
  Table treatment*analysisvariable / binomial(wilson);
   ods output binomialcls=outputdsn2;
Run;
95% Wilson CI for difference in proportions (produces Newcombe CI):
Proc freq;
  Table treatment*analysisvariable / riskdiff(cl=Wilson);
  Exact Riskdiff;
   ods output pdiffcls=outputdsn3;
Run;
95% Clopper-Pearson CI for proportions/percents:
Proc freq;
  Table treatment*analysisvariable / binomial(clopperpearson);
   ods output binomialcls=outputdsn2;
Run;
95% Exact CI for difference in proportions:
Proc freq;
 Table treatment*analysisvariable / riskdiff(cl=Exact);
 Exact Riskdiff;
  ods output pdiffcls=outputdsn3;
Run;
```

## **6.2.** Timing of Analyses

The fully blinded interim analysis will be performed when 80 subjects have been enrolled and have available baseline test results for Nugent score, HIV, Chlamydia, and gonorrhea.

The final analysis will be performed after database lock when all subjects have been followed through Visit 3, the final study visit, at Day 28 (Window: Days 22-30).

## 6.3. Analysis Populations

A tabular listing of all subjects, visits, and observations excluded from the efficacy analysis will be provided in the CSR (Listing 4). Five analysis populations will be used in the analyses, the Intent-to-Treat (ITT), Safety, mITT, Evaluable, and Per Protocol (PP). A listing of subjects whose assigned treatment group does not match their randomized treatment group will be provided in Listing 20.

#### 6.3.1. Intent-to-Treat Analysis (ITT) Population

The ITT population includes all randomized subjects, regardless of whether or not they received study treatment. In the unlikely event of an error in randomization or study product administration (i.e., incorrect product), subjects will be grouped by their intended randomized assignment.

#### **6.3.2.** Safety Analysis Population

The safety population includes all randomized subjects who received at least one dose of study treatment. In the unlikely event of an error in randomization or study product administration (i.e., incorrect product), subjects will be grouped by the product they actually received.

#### 6.3.3. Modified Intention-to-Treat (mITT) Population

The mITT population includes all randomized subjects who met all inclusion/exclusion criteria, excluding those who have a Nugent score <4 at Visit 1 or a positive Visit 1 HIV, Chlamydia, or Neisseria gonorrhoeae test. A review of medical history and concomitant medications will be performed to identify any other infections that may interfere with the efficacy assessment. Subjects with these identified infections will be excluded from the mITT population. In the unlikely event of an error in randomization or study product administration (i.e., incorrect product), subjects will be grouped by their intended randomized assignment. The mITT population will be used as the primary analysis population for the primary efficacy endpoint test of 5% Monolaurin Vaginal Gel to Vehicle Placebo Gel.

#### **6.3.4.** Evaluable Population

The Evaluable population includes all subjects in the mITT population who received study treatment and returned for at least one post-baseline visit that includes an assessment of efficacy.

In the unlikely event of an error in randomization or study product administration (i.e., incorrect product), subjects will be grouped by the product they actually received.

#### 6.3.5. Per Protocol Population

The Per Protocol (PP) population for all endpoints measured at Visit 2 includes all randomized subjects who met all inclusion/exclusion criteria, did not have sexual intercourse including receptive oral sex or insertion of substances or objects intravaginally between Visit 1 and Visit 2, complied with the assigned study treatment, returned to the study site for the Test of Cure visit within the specified window (Visit 2 Study Day 8 relative to the first day of treatment [Window: Days 8-15]), or discontinued study product early due to lack of treatment effect or received vaginosis or systemic antimicrobial therapy other than study drug before Visit 2. Subjects with

Visit 1 test results including a grade 3 laboratory abnormality, a positive Visit 1 HIV, Chlamydia, or *Neisseria gonorrhoeae* test, are found to have a PAP result consistent with HSIL, AGUS, or CIN2 or greater, or a Visit 1 Nugent score < 4 will be excluded from the PP population. A review of medical history and concomitant medications will be performed to identify any other infections that may interfere with the efficacy assessment. Subjects with these identified infections will be excluded from the PP population.

The PP population for all endpoints measured at Visit 3 includes all randomized subjects who met all inclusion/exclusion criteria, did not have sexual intercourse including receptive oral sex or insertion of substances or objects intravaginally between Visit 1 and Visit 2 or 48 hours before Visit 3, complied with the assigned study treatment, returned to the study site for Visit 2 and Visit 3 within the specified windows (Visit 2 Study Day 8 relative to the first day of treatment [Window: Days 8-15]), Visit 3 Study Day 28 relative to the first day of treatment [Window: Days 22-31]), or discontinued study product early due to lack of treatment effect or received vaginosis or systemic antimicrobial therapy other than study drug between Visits 1 and 3. Subjects with Visit 1 test results including a grade 3 laboratory abnormality, a positive Visit 1 HIV, Chlamydia, or Neisseria gonorrhoeae test, are found to have a PAP result consistent with HSIL, AGUS, or CIN2 or greater, or a Visit 1 Nugent score < 4 will be excluded from the PP population. A review of medical history and concomitant medications will be performed to identify any other infections that may interfere with the efficacy assessment. Subjects with these identified infections will be excluded from the PP population.

See Section 9.2 for measurements of compliance.

In the unlikely event of an error in randomization or study product administration (i.e., incorrect product), subjects will be grouped by the product they actually received.

## 6.4. Covariates and Subgroups

Clinical and therapeutic cure will be analyzed by subgroup. Subgroups will be defined by first time or recurrent BV infection as defined in Section 3.3. Additionally, subjects with *Candida spp.* identified at screening will be analyzed to evaluate quantitative changes of *Candida spp.* See Section 8.3 for more details on the exploratory efficacy analyses.

## 6.5. Missing Data

Subjects who are non-evaluable for clinical cure at the TOC visit will be excluded from the PP population. Non-evaluable therapeutic cures will be handled similarly for the PP population. For the mITT, ITT, and Evaluable analysis populations, the cure status of subjects whose status cannot be determined at the TOC visit for any reason will be considered 'not cured' or failure for all cure-related endpoints. The cure status of subjects whose status cannot be determined at Visit 3 for any reason will be imputed using Last Observation Carried Forward (LOCF). Note this differs from what is stated in Section 11.3 of the protocol. See Section 12 for more details.

A sensitivity analysis will be performed to assess the impact of missing results on the primary efficacy outcome. The primary analysis will be repeated in which subjects in the 5% Monolaurin Vaginal Gel arm who are not evaluable for clinical cure will have their cure status imputed as a clinical failure and subjects in the placebo arm who are not evaluable for clinical cure will have their cure status imputed as a clinical cure. See **Table 56**.

## 6.6. Interim Analyses and Data Monitoring

The study is monitored to determine if any of the safety halting rules are met.

Enrollment will be halted for DSMB review/recommendation if any of the following are reported:

- 1. One or more subjects experiences a treatment-related SAE.
- 2. One or more subjects experiences vulvar and/or vaginal ulceration, abscess, or necrosis associated with study product administration.
- 3. Two or more subjects experience a treatment-related severe (Grade 3) unsolicited adverse event
- 4. Three or more subjects who received at least one treatment dose experience the same severe (Grade 3) solicited AE as evaluated by a licensed clinician.
- 5. Three or more subjects who received at least one treatment dose experience a severe (Grade 3) study-related laboratory abnormality in the same laboratory parameter.
- 6. An overall pattern of symptomatic, clinical, or laboratory events that the DMID, Medical Monitor, or DSMB consider associated with study product and that may collectively represent a serious potential concern for safety.

If any of the halting rules are met, the study will not continue with the remaining enrollments or study treatments without a review by and recommendation from the DSMB to proceed. A summary of halting rules is provided in **Table 85.** 

The DSMB met after 30 subjects received at least one dose of study drug and completed Visit 2. The DSMB will also review study progress and subject safety data at least annually during the course of the study and will hold a study closeout meeting 6 to 8 months after database lock, as defined in the DSMB Charter. The DSMB may also meet for an ad hoc review in response to a safety issue.

Additionally, a single, fully blinded interim analysis took place to reassess the adequacy of the sample size based on subjects meeting eligibility for the mITT population. After eighty subjects were enrolled and had available baseline test results for Nugent score, HIV, chlamydia and gonorrhea, the fraction of subjects enrolled to date who were eligible for the mITT cohort was estimated. Based on this calculation, the enrollment target was not increased from 120 subjects. The study sponsor and investigators had access to the data shared in fully blinded reports issued to the DSMB. The tables and figures for the interim analysis are contained in the DSMB Interim Analysis Safety Summary Report.

#### 6.7. Multicenter Studies

Safety and efficacy data will be pooled across all clinical sites. Center effects are not anticipated because treatment is self-administered, the sites are using standardized procedures for assessment of unsolicited adverse events, and the study relies on a central laboratory for Gram stain Nugent scoring. See Sections 8.3 and 9.3 for more details.

## 6.8. Multiple Comparisons/Multiplicity

No adjustments for multiplicity are planned.

#### 7. STUDY SUBJECTS

## 7.1. Subject Disposition

The disposition of subjects in the study will be tabulated by randomized treatment group and all subjects. Table 2 shows the number of subjects who are screen failures and the number of subjects that met each inclusion/exclusion criterion. Table 3 summarizes the ITT and mITT population eligibilities by randomized treatment group and reasons excluded and Table 4 summarizes the safety, Evaluable and PP analysis population eligibilities by actual treatment group and reasons excluded. Subjects will be included in the count for a particular reason for Exclusion if they met that criterion. As subjects may meet more than one criterion for exclusion, the "Excluded from..." counts may be less than the sum of the individual reason counts. A listing of the subjects excluded from each of the analysis populations and the reasons for exclusion will be provided (Listing 4). The number of enrolled subjects in the study completing study milestones will be tabulated separately by randomized treatment group. Table 5 shows the total number of subjects enrolled, randomized, treated, complying with treatment, completing Visits 2, and 3, and completing Visits 2 and 3 and in the PP population by randomized treatment group. A listing of subjects who completed the study, terminated early from study, or discontinued treatment and the reason for early termination or treatment discontinuation is included in Listing 1.

**Figure 1** is a flowchart showing the disposition of study subjects in the primary efficacy analysis, adapted from the CONSORT statement. It shows the number of subjects eligible, enrolled and randomized, lost to follow-up, and analyzed for the primary efficacy analysis, overall and by treatment group.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category, the type of deviation, and randomized treatment group for all enrolled subjects (**Table 6**). All subject-specific protocol deviations and non-subject-specific protocol deviations will be included in Appendix III as data listings (**Listings 2** and **3**, respectively).

#### 8. EFFICACY EVALUATION

All efficacy variables will be listed by subject and summarized by analysis population and treatment group. Continuous efficacy variables will use some or all of the following: N, Mean, Standard Deviation, Median, Minimum and Maximum, whereas Number and Percent will summarize categorical efficacy variables. Confidence intervals for binomial proportions and difference in binomial proportions will be computed using the Wilson confidence limits.

## 8.1. Primary Efficacy Analysis

The primary efficacy endpoint is the proportion of subjects with clinical cure in each study arm at Visit 2 (Day 8-15), TOC.

A test of hypothesis comparing the proportion of subjects who achieve clinical cure at the Test of Cure Visit, Visit 2 (Day 8-15), will be conducted in the mITT population using the randomized treatment, and repeated as a secondary analysis using the actual treatment received in the PP population and the Evaluable analysis population, and using the randomized treatment in the Intent-to-Treat population. The null hypothesis for each comparison is that there is no difference in proportions of clinical cure between treatment groups, with a two-sided alternative that considers the possibility of a difference in either direction. Fisher's exact test at the 5% two-sided level of significance will be used without adjustment for multiplicity. The number of subjects, the proportion of subjects who achieved clinical cure (clinical cure rate), and the 95% Wilson confidence interval for the proportion of subjects achieving clinical cure will be presented for each analysis population and treatment group. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented. See **Table 29**. See Section 6.1 for pseudocode to fit the above analyses.

A subject listing of individual Amsel criteria will be provided in **Listing 22**. A summary of Amsel criteria is provided for subjects by visit and site in **Table 33**. The number of Amsel criteria present (0,1,2,3,4), pH (> 4.5,  $\leq$ 4.5), Clue cells ( $\geq$ 20%, <20%), Amine ("whiff") test on KOH wet mount (Positive, Negative), and discharge (yes/no) will be summarized. A summary of Amsel criteria is provided for subjects by visit and treatment group for each analysis population in **Tables 34-37**. Individual efficacy response data is presented in **Listing 10**. Reasons for clinical failure are provided in **Listing 24**.

## 8.2. Secondary Efficacy Analyses

Secondary efficacy analyses will be performed in the mITT, ITT, Evaluable and PP populations. The mITT and ITT populations will be summarized by randomized treatment and the Evaluable and PP populations will be summarized by actual treatment received.

**Table 30** presents the proportion of subjects with clinical cure in each treatment group at Visit 3 (Day 22-31). The number of subjects, the proportion of subjects who achieved clinical cure (clinical cure rate), and the 95% Wilson confidence interval for the proportion of subjects achieving clinical cure will be presented for each analysis population and treatment group. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented.

**Tables 31 and 32** present the proportion of subjects with therapeutic cure in each treatment group at Test of Cure Visit, Visit 2 (Day 8-15) and at Visit 3 (Day 22-31), respectively. The number of subjects, the proportion of subjects who achieved therapeutic cure (therapeutic cure rate), and the 95% Wilson confidence interval for the proportion of subjects achieving therapeutic cure will be presented for each analysis population, treatment group, and study visit. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented.

**Tables 38-41** presents the number and proportion of subjects with Nugent scores falling in negative BV (3 or less), intermediate (4-6), and BV (7-10) range by analysis population, study visit, and site. The 95% Wilson confidence intervals for the proportion of subjects falling in each category will also be presented. **Tables 42-43** presents the proportion of subjects with Nugent score of 3 or less (negative for BV), 4-6 (intermediate), and 7-10 (positive for BV) in each treatment group at Visit 1, at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31). The number and proportion of subjects with Nugent scores falling in negative, intermediate, and BV range is presented by analysis population, study visit, and treatment group. The 95% Wilson confidence intervals will also be presented. Mean Nugent scores will also be presented by analysis population, study visit, and treatment group in **Table 44.** A subject listing of Nugent scores and bacterial morphotypes will be presented in **Listing 23**. Raw Nugent scores are displayed graphically by visit, treatment group, and analysis population in **Figures 2-5**. Categorical and Continuous Nugent Score characteristics are presented by study visit, clinical cure status, and treatment group for subjects in the ITT population in **Tables 45 and 46**. See Section 6.1 for pseudocode to use in calculating the 95% CIs.

## 8.3. Exploratory Efficacy Analyses

Exploratory efficacy analyses will be performed in the mITT, ITT, Evaluable and PP populations. The mITT and ITT populations will be summarized by randomized treatment and the Evaluable and PP populations will be summarized by actual treatment received.

The first exploratory efficacy endpoint is the proportion of subjects with clinical cure in each treatment group by subgroup (first time or recurrent infection) at the Test of Cure Visit, Visit 2 (Day 8-15) and at Visit 3 (Day 22-31). The number of subjects, the proportion of subjects who achieved clinical cure (clinical cure rate), and the 95% Wilson confidence interval for the proportion of subjects achieving clinical cure will be presented for each analysis population, treatment group, and infection type (first time or recurrent). In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented. See **Tables 47-50**. A listing of subjects BV infection status (first time or recurrent) will be provided in **Listing 25.** See Section 6.1 for pseudocode to use in calculating the 95% CIs.

The second exploratory efficacy endpoint is the proportion of subjects with therapeutic cure in each study arm by subgroup (first time or recurrent infection) at the Test of Cure Visit, Visit 2 (Day 8-15) and at Visit 3 (Day 22-31). The number of subjects, the proportion of subjects who achieved therapeutic cure (therapeutic cure rate), and the 95% Wilson confidence interval for the proportion of subjects achieving therapeutic cure will be presented for each analysis population, treatment group, and infection type (first time or recurrent). In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented. See **Tables 51-54**.

The third exploratory efficacy endpoint is the mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.*, respectively, in each treatment group at Visit 1, at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31). Mean count and standard deviation of each specimen type will be presented by study visit, analysis population, and treatment group. Additionally, mean change from baseline and corresponding standard deviation will be presented for Visit 2 and Visit 3. See **Tables 57-60**.

The fourth exploratory efficacy endpoint is the mean fungal colony count of *Candida spp*. in vaginal secretions in each study arm at baseline, at Visit 2 (Day 8-15) and at Visit 3 (Day 22-31). Mean count and standard deviation will be presented by study visit, analysis population, and treatment group for subjects with *Candida spp*. identified by either positive culture counts or presence of budding yeast organisms at screening. Additionally, mean change from baseline and corresponding standard deviation will be presented for Visit 2 and Visit 3. See **Table 61**.

#### 9. SAFETY EVALUATION

#### 9.1. Demographic and Other Baseline Characteristics

Ethnicity and race will be summarized by site in **Table 7** and by randomized treatment group in **Table 9**. Ethnicity is categorized as Hispanic or Latino, or Not Hispanic or Latino. Race is categorized as American Indian or Alaska Native, Asian, Native Hawaiian or Other Pacific Islander, Black or African American, White, Multi-Racial or Unknown In accordance with NIH reporting policy. Subjects may self-designate as belonging to more than one race (Multi-Racial) or may refuse to identify a race (Unknown), the latter reflected in the Case Report Form (CRF) as "No" to each racial option. Age and episodes of BV (including current episode) in the previous 12 months (from the sexual history questionnaire) will be summarized by site in **Table 8** and by randomized treatment in **Table 10**.

Baseline sexual history will be presented by site in **Table 11** and by randomized treatment group in **Table 12** for all enrolled subjects.

Baseline clinical assessment of BV will be presented by sign/symptom, maximum severity, and site for subjects in the Safety population in **Table 13.** Baseline clinical assessment of BV will be presented by sign/symptom, maximum severity, and actual treatment group for subjects in the Safety population in **Table 14**.

Individual subject listings will be presented for all demographics (**Listing 5**); sexual history (**Listings 7-8**).

#### 9.1.1. Concurrent Illnesses and Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA® dictionary version 20.1 or higher. Summaries of subjects' pre-existing medical conditions will be presented by randomized treatment group overall and by each site (**Tables 15-18**).

Individual subject listings will be presented for all medical conditions (Listing 6).

## 9.2. Measurements of Treatment Compliance

All subjects are to receive a total of six doses of study product (twice daily for three consecutive days). The first dose is administered in clinic and the remaining 5 doses will be administered by the subject at home. Subjects record the timing of all remaining doses on a memory aid, which is reviewed with clinic staff at Visit 2. Compliance is assessed by the study coordinator's count of used/unused applicators in each returned subject kit. If a kit is not returned, compliance will be

assessed by the subject's self-report on the memory aid. If an incomplete kit is returned, the subject's self-report will be used in conjunction with the count of used/unused applicators to determine subject compliance. In addition to the count of used/unused applicators, the timing of dosing will be considered. Subjects are instructed to administer study product twice daily (morning and evening) with at least 8 hours between doses. If the subject received her first dose after 3 pm, she will be instructed to administer the next dose the following morning. A subject is compliant if she uses at least 5 of 6 doses and they were administered within 72 hours from the first dose, at least 8 hours apart, and if no more than 2 doses in a 24 hour period are taken.

If a subject is found to have a positive test for HIV, chlamydia or gonorrhea or a Grade 3 laboratory abnormality from Visit 1, she will be notified of the results, withdrawn from receiving further study product, but will be followed for safety and efficacy. All subjects who were randomized will be followed for safety and efficacy. If any subject experiences a severe AE related to the study product, further doses will be discontinued.

The dates of first treatment are presented for subjects in the Safety population by site in **Table 19** and actual treatment group in **Table 20**. The number of subjects not compliant with study treatment will be presented by treatment group as part of the subject disposition table (**Table 5**). The number of doses administered as scheduled and out of window is summarized for subjects in the Safety population by site in **Table 21** and by actual treatment in **Table 23**.

Administration schedule is categorized as either "as scheduled" or "out of window." As scheduled is defined as twice daily (morning and evening) with at least 8 hours between doses as reported on the memory aid. **Tables 22 and 24** show the number and percentage of subjects who received the dose as scheduled, received the dose out of window, or missed the dose, for each of the 6 doses, by site and actual treatment group, respectively for subjects in the Safety population.

**Table 25** displays product administration position by site and number of doses administered and **Table 27** displays product administration position by actual treatment group and number of doses administered for the subjects in the Safety population. Product administration position is categorized as either "Recumbent" or "Not Recumbent." A subject contributes to the "Recumbent" rows if they administer each of the specified number of doses in the recumbent position. If a subject was not recumbent for at least one of the specified number of doses or is missing product administration position, they will appear in the "Not Recumbent" rows. **Tables 26 and 28** show the number and percentage of subjects who received the dose and remained in the recumbent position, received the dose and did not remain in the recumbent position, or did not enter the position they were in for the dose, for each of the 6 doses, by site and actual treatment group, respectively for subjects in the Safety population.

Individual subject listings of treatment compliance assessment will be presented (**Listing 9**).

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total safety population size and population within actual treatment group. All adverse events reported will be included in the summaries and analyses. All analyses in Section 9.3 will be performed in the safety analysis population using the actual treatment received.

#### 9.3.1. Solicited Events and Symptoms

Solicited urogenital symptoms were collected before study product administration, and then daily for 5 days and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Urogenital symptoms include: vaginal odor, vaginal pain, vaginal tenderness, vulvar/vaginal itching, vaginal dryness, vaginal discharge, and vulvar inflammation. Any symptom that is present at the time that the subject is screened should be considered as baseline and not reported as a solicited urogenital AE. However, if it deteriorates at any time during the study, it will be recorded as a solicited urogenital AE. If a symptom is reported that was not present at baseline, it too will be recorded as a solicited urogenital AE. Treatment emergent solicited urogenital adverse events will be identified by comparing the severity of the baseline solicited urogenital symptoms with the severity of the post-baseline solicited urogenital symptoms. If the severity increases post-baseline or the symptoms appears post-baseline when it was 'None' at baseline, then the symptom will be considered to be treatment-emergent.

The first primary safety endpoint is the number of subjects reporting treatment-emergent solicited urogenital AEs following the first dose of the study product through Visit 2 (Day 8-15).

The number and percent of subjects reporting at least one treatment-emergent solicited urogenital adverse event will be summarized for each solicited adverse event and any solicited adverse event along with the 95% Clopper-Pearson CI and presented in **Table 62**. **Table 63** will present the proportion of subjects experiencing any solicited urogenital event and each specific urogential solicited event, along with the 95% Clopper-Pearson CI of the proportion, the difference in the proportions of subjects experiencing a solicited event between 5% Monolaurin Vaginal Gel and Placebo Gel, the 95% Exact CI of the difference and the p-value for a Fisher's exact test. A Fisher's exact test will be performed to test for the difference in the proportion of subjects reporting a treatment emergent solicited urogenital adverse event. The null hypothesis is that there is no difference in proportions of subjects reporting solicited urogenital AEs between treatment groups, with a two-sided alternative which considers the possibility of a difference in either direction. Section 6.1 provides pseudo SAS code to use for the analyses.

For each treatment-emergent solicited urogenital adverse event and any solicited adverse events, the maximum severity over 5 days after the first dose will be summarized for the Safety population. The number and percentage of subjects reporting each treatment-emergent solicited adverse event will be summarized by the maximum severity and actual treatment group along with the 95% Clopper-Pearson CIs. For each event the denominator is the number of subjects with non-missing data for the specific solicited urogenital adverse event. See **Table 64** and **Figure 6**.

**Table 64** and **Figure 7** will summarize any reported solicited symptom (treatment-emergent and non treatment-emergent) and each solicited symptom by maximum severity over 5 days after the first dose along with the 95% Clopper-Pearson CI for the Safety population. The number and percentage of subjects reporting each symptom will be summarized by the maximum severity and actual treatment group. For each event, the denominator is the number of subjects with non-missing data for the specific symptom. Maximum severity of solicited symptoms is displayed by study day and treatment group in **Figure 8**.

The number of subjects reporting a solicited symptom will be summarized for each day for all subjects and separately for each treatment group (**Tables 66-68**) and graphically in a bar chart (**Figure 7**).

Solicited symptoms by subject will be presented in Listing 12.

#### 9.3.2. Unsolicited Adverse Events

The first secondary safety endpoint is the number of subjects experiencing non-laboratory, non-solicited AEs following the first dose of the study product through Visit 3 (Day 22-31). Laboratory events are defined as WBC count, hemoglobin, platelets, neutrophil count, creatinine, AST (SGOT), ALT (SGPT), and total bilirubin, and glucose (random). Events involving laboratory parameters that are not collected as part of the protocol will be counted as non-laboratory, non-solicited adverse events. The number of subjects, the proportion of subjects who experienced non-laboratory, non-solicited AEs following the first dose of the study product through Visit 3 (Day 22-31), and the 95% Clopper-Pearson CIs for the proportion of subjects who experienced non-laboratory, non-solicited AEs through Visit 3 will be presented for the safety population and actual treatment group. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Exact CIs will be presented in **Table 69**.

The proportion of subjects reporting at least one non-laboratory, non-solicited adverse event will be summarized by MedDRA® system organ class and preferred term for all subjects and each actual treatment group. Denominators for percentages are the number of subjects who received the study product being summarized. A 95% Clopper-Pearson CI will be presented for each MedDRA® system organ class and preferred term (**Table 70**). Adverse events by subject will be presented in **Listing 13**.

The following summaries for non-solicited, non-laboratory adverse events will be presented by MedDRA® system organ class, preferred term, and treatment group:

- Subject level summary of severity and relationship to study product (**Tables 71-73**);
- Subject level summary of severity by related AEs (**Tables 74-76**);
- Subject incidence of adverse events over time (**Tables 77-79**). AEs will be categorized as occurring from Visit 1 through the TOC, Visit 2, from the TOC, Visit 2 through Visit 3, and anytime during the study;
- Total frequency of adverse events over time (**Tables 80-82**). AEs will be categorized as occurring from Visit 1 through the TOC, Visit 2, from the TOC, Visit 2 through Visit 3, and anytime during the study.
- Subject listing of non-serious adverse events of moderate or greater severity (**Table 88**);
- Bar chart of total frequency of adverse events by severity and MedDRA® system organ class (**Figure 9**);
- Bar chart of subject incidence of adverse events by severity and MedDRA® system organ class (**Figure 10**);

- Bar chart of total frequency of adverse events by severity and treatment group (Figure 11);
- Bar chart of subject incidence of adverse events by severity and treatment group (**Figure 12**):
- Bar chart of total frequency of adverse events by relationship to study product and MedDRA® system organ class (**Figure 13**);
- Bar chart of subject incidence of adverse events by relationship to study product and MedDRA® system organ class (Figure 14):
- Bar chart of total frequency of adverse events by relationship to study product (**Figure 15**).
- Bar chart of subject incidence of adverse events by relationship to study product (**Figure 16**).
- The number of adverse events occurring in 5% of subjects in any treatment group will be presented by MedDRA® system organ class, preferred term, and treatment group in **Table 83.**
- The number of subjects reporting adverse events occurring in 5% of subjects in any treatment group presented by MedDRA® system organ class, preferred term and treatment group in **Table 84.**

## 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The second primary safety outcome is the number of subjects reporting serious adverse events (SAEs) considered product related following the first dose of the study product through Visit 3 (Day 22-31). The number of subjects, the proportion of subjects who experienced product-related SAEs, and the 95% Clopper-Pearson confidence interval for the proportion of subjects who experienced product-related SAEs will be presented for each analysis population, treatment group, and study visit. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Exact confidence intervals will be presented. The proportion of subjects in each treatment group who experience product-related SAEs following the first dose of the study product through Visit 3 (Day 22-31) will be tested using a Fisher's exact test at the 5% two-sided level of significance level without adjustment for multiplicity in the safety analysis population (**Table 86**). See Section 6.1 for pseudocode for calculating p-values and CIs.

A listing of deaths and serious adverse events will be presented, including Subject ID, treatment group, Adverse Event Description, Study Day the Event became Serious, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event in days (**Table 87**).

## 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome,

including information regarding any complications with pregnancy and/or delivery. A listing of the total pregnancies, number of live births, and number of spontaneous abortions, elective abortions or still births will be presented (**Listings 26-29**).

## 9.6. Clinical Laboratory Evaluations

Safety clinical laboratory data includes: WBC count, hemoglobin, platelets, neutrophil count, creatinine, AST (SGOT), ALT (SGPT), total bilirubin, and glucose (random). These hematology and chemistry parameters will be collected at Visit 1 and Visit 2. Laboratory abnormalities that were stable at Visit 2 will not be repeated at Visit 3. Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 will be repeated at Visit 3. A laboratory abnormality is considered an adverse event if there is a worsening of the laboratory value at Visit 2 from the baseline value and it increases in laboratory toxicity grading from the baseline toxicity grading. For laboratory abnormalities repeated at Visit 3, if there is a worsening of the laboratory value at Visit 3 from the Visit 2 value and it increases in laboratory toxicity grading, it is considered an additional adverse event. Toxicity grading can be found in Appendix B of the protocol. All analyses in Section 9.6 will be performed in the safety analysis population.

The second secondary safety endpoint is number of subjects experiencing laboratory AEs following the first dose of the study product through Visit 2 (Day 8-15). The number of subjects reporting at least one laboratory measurement at the visit, the proportion of subjects who experienced laboratory AEs, and the 95% Clopper-Pearson confidence interval for the proportion of subjects who experienced laboratory AEs will be presented by treatment group. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Exact confidence intervals will be presented in **Table 89**.

The proportion of subjects with laboratory results meeting toxicity grading criteria will be presented for each parameter in **Tables 90 and 92** by severity, study day and treatment group. The proportion of subjects with laboratory results related to study product meeting toxicity grading criteria will be presented for each parameter in **Tables 91 and 93** by severity, study day and treatment group. Descriptive statistics including mean, standard deviation, median, mean change from baseline and associated standard deviation by study day, for each laboratory parameter, will be summarized in **Table 94** by treatment group. Laboratory values will be presented by parameter, severity and visit in **Figures 17-19.** Mean changes in laboratory values will be presented in **Figures 20-28**.

The denominator for proportions is the number of subjects with each specific laboratory value at the visit.

Laboratory abnormalities are those that meet toxicity grading. When the site-specific laboratory normal range is available, if there is a discrepancy between the laboratory value in Appendix B of the protocol and the site-specific laboratory normal range, the value in Appendix B of the protocol will take precedence in determining Grade 1 adverse events. Otherwise, all laboratory tests will be graded per the toxicity table in Appendix B of the protocol. Unscheduled or repeated follow-up laboratory tests for medical or safety reasons will be listed, but excluded from tabular and graphical summaries.

A listing of laboratory tests with toxicity Grade >=1 will also be provided. If a subject meets this criterion, the listing will provide data from all visits for the particular lab test that meet the criteria

so that the time course for the particular lab parameter can be observed. See **Tables 95-96.** A listing of all clinical laboratory values will be generated in **Listings 14 and 15.** 

## 9.7. Physical Evaluations

A physical exam including a gynecological exam will be performed at Visit 1. A gynecological exam and a targeted physical exam based on symptoms will be performed at Visit 2 and Visit 3. The change in physical examination data from Day 1 will be summarized for each visit by treatment group for subjects in the Safety population. The following body systems will be assessed: Abdomen, Cardiovascular/Heart Extremities, General Appearance, Head, Eyes, Ears, Nose, and Throat (HEENT), Lymph nodes, Musculoskeletal, Neck, Neurological, Pulmonary/Chest, and Skin (Listing 16). Findings from the pelvic exam which includes signs of inflammation in the cervix, vagina, and vulva, as well as vaginal discharge, will be presented in Listing 17. Other gynecological test results including saline wet mount, Trichomonas, and KOH wet mount will be presented in Listing 18. Clinical assessment of BV symptoms will be presented in Listing 11.

#### 9.8. Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing as well as medications that were starting during dosing or during follow up will be presented by WHO Drug Anatomical codes (ATC) level 1 and level 2 and actual treatment group for subjects in the Safety population (**Tables 97-100**).

Individual subject listings will be presented for all concomitant medications (Listing 19).

#### 10. OTHER ANALYSES

During the course of the study, the product administration form was updated to capture whether or not the subject remained in a recumbent position for 5 minutes after administration of study treatment. The primary efficacy analysis will be repeated as an exploratory, supplementary analysis of the primary outcome in **Table 55.** This analysis will be performed in the PP population, with the additional stipulation that the subject remain in the recumbent position for 5 of 6 doses to be considered compliant with study product. The number of subjects, the proportion of subjects who achieved clinical cure, and the 95% Wilson confidence interval for the proportion of subjects achieving clinical cure will be presented for each analysis population and treatment group. In addition, the difference in proportions between the 5% Monolaurin Vaginal Gel arm and the Placebo gel arm and 95% Wilson confidence intervals will be presented. A listing of subjects' product administration position for each dose is provided in **Listing 21.** 

## 11. REPORTING CONVENTIONS

P-values  $\ge$ 0.001 and  $\le$ 0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001"; p-values greater than 0.999 will be reported as ">0.999". The mean, median, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles other than the median will use the same number of decimal places as the original data. Proportions will be presented as two decimal
places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values < 1% will be presented as "<1". Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

# 12. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Protocol version 5.0 (August 31, 2016) changed the criterion requiring all four Amsel criteria for inclusion to any 3 of 4 Amsel criteria; changed the allowable interval between a previous vaginal/cervical/pelvic infection or episode of BV from 60 days prior to enrollment to 14 days and removed the prohibition of systemic, vaginal or perineal immunosuppressant or antiinflammatory medications within 14 days of treatment; and changed the procedure for review of the Gram stain when two independent reviewers have different Nugent scores. Protocol version 6.0 (November 29, 2016) included the addition of a clinical site, Duke University, and clarification of temperature range for specimen storage. Protocol version 7.0 (May 11, 2017) removed the criterion requiring subjects over age 21 to report a normal PAP smear within the past 3 years, revised the exclusion for HPV and cervical or vaginal dysplasia to exclude only HSIL, AGUS, or CIN2 or higher, changed exclusions for previous self-treatment for yeast vaginitis and systemic, vaginal, or perineal antibiotics from 14 days to 7 days, and removed exclusion for 6 or more episodes of vaginitis within the past year, clarified that subjects found to have HSIL or AGUS at visit 1 will have study treatment discontinued and subjects found to have HSIL, AGUS, or CIN2 or higher at visit 1 will be excluded from the PP analysis population, and corrected protocol deviation plan such that sexual intercourse 48 hours prior to Visit 3 will not exclude subjects from the Per-Protocol data analysis population definition. Protocol version 8.0 (May 23, 2017) removed exclusion for diabetes.

Protocol Section 11.3 states Last Observation Carried Forward (LOCF) will be used as a sensitivity analysis. Section 6.5 of this analysis plan clarifies that LOCF will be used to impute the cure status of subjects whose status cannot be determined at Visit 3 for any reason. Subjects whose status cannot be determined at the TOC visit, will be considered 'not cured' for all cure-related endpoints.

#### 13. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

#### 14. REFERENCES

- Workowski KA, Berman S. Sexually transmitted diseases treatment guidelines, 2010. MMWR Recommendations and reports: Morbidity and mortality weekly report Recommendations andreports / Centers for Disease Control 2010; 59:1-110
- 2. ACOG Practice Bulletin. Clinical management guidelines for obstetrician-gynecologists, Number 72, May 2006: Vaginitis. Obstetrics and gynecology **2006**; 107:1195-206.

- 3. McCormack WM, Jr., Zinner SH, McCormack WM. The incidence of genitourinary infections in a cohort of healthy women. Sexually transmitted diseases **1994**; 21:63-4.
- 4. Wilson J. Managing recurrent bacterial vaginosis. Sex Transm Infect 2004; 80:8-11.
- 5. Pechous R, Ledala N, Wilkinson BJ, Jayaswal RK. Regulation of the expression of cell wall stress stimulon member gene msrA1 in methicillin-susceptible or -resistant Staphylococcus aureus. Antimicrobial agents and chemotherapy **2004**; 48:3057-63.
- 6. Schlievert PM, Peterson ML. Glycerol monolaurate antibacterial activity in broth and biofilm cultures. PloS one **2012**; 7:e40350.

#### 15. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices I, II, and III.

#### 16. APPENDICES

## **Appendix I: Table Mock-Ups**

This document includes examples mock-ups of tables to present efficacy and safety data.

Sites that are activated after the SAP has been drafted will not appear in the table, figure, or listing shells, but will appear in the final CSR.

Instructional text is included in brackets [Instruction or Implementation Note:].

### LIST OF TABLES

| Table 1: | Schedule of Events |
|---|---|
| Table 2: | Ineligibility Summary of Screen Failures |
| Table 3: | Intent-to-Treat and Modified Intent-to-Treat Analysis Populations by Treatment Group . 45 |
| Table 4: | Safety, Evaluable, and Per-Protocol Analysis Populations by Treatment Group |
| Table 5: | Subject Disposition by Treatment Group - All Enrolled Subjects |
| Table 6: | Distribution of Protocol Deviations by Category, Type, and Treatment Group - All Enrolled |
| Subjects | 48 |
| Table 7: | Summary of Categorical Demographic and Baseline Characteristics by Site - ITT |
| Population | 50 |
| Table 8: | Summary of Continuous Demographic and Baseline Characteristic by Site - ITT Population |
| | 51 |
| Table 9: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - |
| ITT Population | |
| Table 10: | Summary of Continuous Baseline Characteristics by Treatment Group - ITT Population $53$ |
| Table 11: | Baseline Sexual History by Site - ITT Population |
| Table 12: | Baseline Sexual History by Treatment Group - ITT Population |
| Table 13: | Summary of Baseline Clinical Assessment of BV by Site - Safety Population56 |
| Table 14: | Summary of Baseline Clinical Assessment of BV by Treatment Group - Safety Population |
| | 57 |
| Table 15: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ |
| Class and Trea | tment Group - ITT Population - All Sites |
| Table 16: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ |
| | tment Group -ITT Population- Cincinnati Children's Hospital |
| Table 17: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ |
| | tment Group -ITT Population- University of Iowa |
| Table 18: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ |
| | tment Group -ITT Population- Duke University |
| Table 19: | Dates of First Treatment by Site - Safety Population |
| Table 20: | Dates of First Treatment by Treatment Group - Safety Population |
| Table 21: | Dose Administration Schedule by Site and Number of Doses Administered - Safety |
| Population | 61 |
| Table 22: | Dose Administration Schedule by Site and Dose Number - Safety Population |
| Table 23: | Dose Administration Schedule by Treatment Group and Number of Doses Administered - |
| Safety Populati | |
| Table 24: | Dose Administration Schedule by Treatment Group and Dose Number - Safety Population |
| | 64 |

| Table 25: | Product Administration Position by Site and Number of Doses Administered - Safety |
|---|---|
| Population | 65 |
| Table 26: | Product Administration Position by Site and Dose Number - Safety Population |
| Table 27: | Product Administration Position and Number of Doses Administered - Safety Population 67 |
| Table 28: | Product Administration Position by Treatment Group and Dose Number - Safety Population $68$ |
| Table 29: | Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment |
| Group | 69 |
| Table 30: | Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group70 |
| Table 31: | Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and |
| | up71 |
| Table 32: | Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group71 |
| Table 33: | Summary of Amsel Criteria by Site and Study Visit - All Enrolled Subjects |
| Table 34: | Summary of Amsel Criteria by Treatment Group and Study Visit - ITT Population 73 |
| Table 35: | Summary of Amsel Criteria by Treatment Group and Study Visit - mITT Population 73 |
| Table 36: | Summary of Amsel Criteria by Treatment Group and Study Visit - Evaluable Population 73 |
| Table 37: | Summary of Amsel Criteria by Treatment Group and Study Visit - PP Population73 |
| Table 38: | Nugent Scores by Category, Study Visit, Analysis Population, and Site – All Subjects 74 |
| Table 39: | Nugent Scores by Category, Study Visit, Analysis Population, and Site-Cincinnati |
| Children's Hos | spital |
| Table 40: | Nugent Scores by Category, Study Visit, Analysis Population, and Site—University of Iowa 74 |
| Table 41: | Nugent Scores by Category, Study Visit, Analysis Population, and Site—Duke University 74 |
| Table 42: | Nugent Scores by Category, Study Visit, Analysis Population, and Treatment Group - 5% |
| Monolaurin Va | aginal Gel75 |
| Table 43: | Nugent Scores by Category, Study Visit, Analysis Population, and Treatment Group - |
| Placebo Gel | 75 |
| Table 44: | Continuous Nugent Score Characteristics by Study Visit, Analysis Population, and |
| Treatment Gro | up76 |
| Table 45: | Nugent Scores by Category, Study Visit, Clinical Cure Status, and Treatment Group -ITT |
| Population | 77 |
| Table 46: | Continuous Nugent Score Characteristics by Study Visit, Clinical Cure Status, and |
| Treatment Gro | up- ITT Population |
| Table 47: | Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment |
| Group - First T | Time BV |
| Table 48: | Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment |
| Group - Recurr | rent BV |
| Table 49: | Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group - First Time |
| BV | 79 |
| Table 50:<br>BV | Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group - Recurrent 79 |
| Table 51: | Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and |
| Treatment Gro | up - First Time BV80 |
| Table 52: | Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and |
| Treatment Gro | up - Recurrent BV80 |
| Table 53:<br>Time BV | Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group - First 80 |

| Table 54: | Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group - |
|---|---|
| Recurrent BV | 80<br>CV: 1 C P 1 |
| Table 55: | Clinical Cure Results at the Test of Cure Visit, Visit 2 by Treatment Group- Recumbent |
| • | Population |
| Table 56: | Clinical Cure Results at the Test of Cure Visit, Visit 2 by Treatment Group Using Imputation |
| | tion |
| Table 57: | Mean count of Lactobacillus spp., Gardnerella spp., and Mobiluncus spp. by Study Visit, |
| Table 58: | Group - ITT Population |
| Table 59: | Group - mITT Population |
| | Group - Evaluable Population |
| Table 60: | Mean count of Lactobacillus spp., Gardnerella spp., and Mobiluncus spp. by Study Visit, |
| | Group - PP Population |
| Table 61: | Mean fungal colony count of Candida Spp. by Study Visit, Analysis Population, and |
| | up in Subjects with Candida spp. Identified at Screening |
| Table 62: | Number and Percentage of Subjects Experiencing Treatment Emergent Solicited Urogenital |
| | s with 95% Confidence Intervals by Symptom and Treatment Group - Safety Population 85 |
| Table 63: | Comparison of the Proportion of Subjects Experiencing Treatment Emergent Solicited |
| | verse Events through the Test of Cure Visit, Visit 2 by Treatment Group - Safety Population |
| Orogenital Au | 86 |
| Table 64: | Number and Percentage of Subjects Experiencing Treatment Emergent Solicited Urogenital |
| | s by Symptom, Maximum Severity, and Treatment Group - Safety Population |
| Table 65: | Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, |
| | erity, and Treatment Group - Safety Population |
| Table 66: | Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, |
| | Day, and Treatment Group - All Treatment Groups - Safety Population |
| Table 67: | Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, |
| | Day, and Treatment Group-5% Monolaurin Vaginal Gel - Safety Population |
| Table 68: | Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, |
| | Day, and Treatment Group-Placebo Gel - Safety Population 94 |
| Table 69: | Proportion of Subjects Reporting Non-Solicited Non-Laboratory Adverse Events Following |
| | of Study Product through Visit 3 by Treatment Group - Safety Population95 |
| Table 70: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Events |
| with 95% Con | fidence Intervals by MedDRA System Organ Class, and Preferred Term, and Treatment |
| | Population96 |
| Table 71: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| Events by Me | dDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and |
| | up - Safety Population 97 |
| Table 72: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| Events by Me | dDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and |
| | up - 5% Monolaurin Vaginal Gel - Safety Population |
| Table 73: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| Events by Me | dDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and |
| Treatment Gro | up-Placebo Gel - Safety Population |
| Table 74: | Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory |
| Adverse Event | s by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment |
| Group - Safety | Population - All Subjects |
| Table 75: | Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory |
| Adverse Event | s by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment |
| Group-5% Mor | nolaurin Vaginal Gel - Safety Population98 |

| Table 76: | Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory |
|---|---|
| Adverse Event | s by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment |
| Group-Placebo | Gel - Safety Population98 |
| Table 77: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| Events by Med | dDRA System Organ Class and Preferred Term, Study Day, and Treatment Group - Safety |
| Population - A | ll Subjects |
| Table 78: | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| | dDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-5% |
| | aginal Gel - Safety Population |
| | Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse |
| | dDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-Placebo |
| | opulation99 |
| Table 80: | Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| | erred Term, Study Day, and Treatment Group - Safety Population - All Subjects 100 |
| Table 81: | Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| | ferred Term, Study Day, and Treatment Group-5% Monolaurin Vaginal Gel - Safety |
| Population | 100 |
| Table 82: | Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| | erred Term, Study Day, and Treatment Group-Placebo Gel - Safety Population |
| | Number of Non-Solicited Non-Laboratory Adverse Events Occurring in 5% of Subjects in |
| | Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety |
| Population | 101 |
| Table 84: | Subjects Reporting Non-Solicited Non-Laboratory Adverse Events occurring in 5% of |
| | y Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment |
| | Population |
| Table 85: | Summary of Halting Rules - Safety Population |
| Table 86: | Number and Percentage of Subjects Experiencing Serious Adverse Events Related to Study |
| | 5% Confidence Intervals by Treatment Group - Safety Population |
| Table 87: | Listing of Serious Adverse Events - Safety Population |
| Table 88: | Listing of Non-Serious, Non-Solicited, Non-Laboratory, Moderate or Severe Adverse |
| | Population |
| Table 89: | Proportion of Subjects Reporting Laboratory Adverse Events Following the First Dose of |
| | through the Test of Cure Visit, Visit 2 by Treatment Group - Safety Population |
| Table 90: | Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group - |
| | Safety Population |
| Table 91: | Laboratory Results Related to Study Product by Parameter, Maximum Severity, Study Visit, |
| | Group - Hematology - Safety Population |
| Table 92: | Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group – |
| | Safety Population |
| Table 93: | Laboratory Results Related to Study Product by Parameter, Maximum Severity, Study Visit, |
| | Group - Biochemistry - Safety Population |
| Table 94: | Laboratory Summary Statistics by Parameter, Study Visit, and Treatment Group - Safety |
| Population | 114 |
| Table 95: | Listing of Abnormal Laboratory Results - Hematology - Safety Population |
| Table 96: | Listing of Abnormal Laboratory Results - Biochemistry - Safety Population |
| Table 90. | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug |
| | and Treatment Group - Safety Population - All Subjects |
| Table 98: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug |
| | and Treatment Group-Safety Population-Cincinnati Children's Hospital |
| Table 99: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug |
| | and Treatment Group-Safety Population-University of Iowa |
| × // (0.000 10.00 10.00 | and required a virtual-particly regulation-commediate Of IOWa |

| Statistical Anal | ysis Plan |
|------------------|-----------|
| DMID Protocol | 112-0021 |

## **Section 14.1 Demographic Data**

**Table 2:** Ineligibility Summary of Screen Failures

| Inclusion/Exclusion<br>Category | Inclusion/Exclusion Criterion | Number of Subjects* |
|---|---|---|
| Inclusion and Exclusion | Any criterion | X |
| Inclusion | Any inclusion criterion | X |
| | [inclusion criterion 1] | X |
| | [inclusion criterion 2] | X |
| | [inclusion criterion 3] | Х |
| Exclusion | Any exclusion criterion | X |
| | [exclusion criterion 1] | X |
| | [exclusion criterion 2] | Х |
| | [exclusion criterion 3] | X |
| Declined Enrollment | Any Reason | X |
| | Time commitment | X |
| | Concern of potential risks | X |
| | Number of procedures | X |
| | Unable to contact subject | X |
| | Other | x |

Note: \*More than one criterion may be marked per subject.

Table 3: Intent-to-Treat and Modified Intent-to-Treat Analysis Populations by Treatment Group

| | | | | urin Vaginal<br>Gel<br>=X) | ( | icebo<br>Gel<br>I=X) | Sul | All<br>bjects<br>V=X) |
|---|---|---|---|---|---|---|---|---|
| Analysis Population | Eligibility Category | Reason Subjects Excluded | n | % | n | % | n | % |
| Intent-to-Treat (ITT) Analysis<br>Population | Eligible for ITT | | X | X | х | x | Х | х |
| | Eligible for mITT | | X | X | х | X | X | х |
| | | Any Reason | X | X | х | X | X | X |
| Modified Intent-to-Treat (mITT) | | Did not meet inclusion/exclusion criteria | Х | X | х | X | X | х |
| Analysis | Excluded from mITT | Nugent score < 4 from Visit 1 | Х | X | х | X | Х | х |
| | | Positive HIV, Chlamydia or Neisseria gonorrhoeae test | X | X | х | X | X | X |
| | | Positive for other concomitant vulvovaginal infections | Х | X | х | X | X | х |

Note: N=number of enrolled subjects

Treatment group is the treatment group to which a subject was randomized.

Table 4: Safety, Evaluable, and Per-Protocol Analysis Populations by Treatment Group

| | | | Va | Monolaurin<br>ginal Gel<br>(N=X) | ( | icebo<br>Gel<br>I=X) | Sul | All<br>ojects<br>(=X) |
|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Eligibility<br>Category | Reason Subjects Excluded | n | % | n | % | n | % |
| | Eligible for Safety | | х | X | X | х | х | Х |
| | Excluded from | Any Reason | X | X | X | X | Sul (N) | X |
| | Safety | Did not Receive Study product | X | X | X | X | Sub (N) | X |
| | Eligible for Evaluable | | X | X | X | X | X X X X | X |
| | | Any Reason | х | X | X | х | х | Х |
| | | Did not meet inclusion/exclusion criteria | х | Х | X | X | х | Х |
| | | Nugent score < 4 from Visit 1 | X | X | X | X | X | X |
| Evaluable Analysis<br>Population | Excluded from | Positive Chlamydia or Neisseria gonorrhoeae test | X | X | X | X | х | X |
| Population Safety Analysis Population Evaluable Analysis | Evaluable | Positive for other concomitant vulvovaginal infections | | х | Х | Х | х | X |
| | | Did not receive study product | | x | X | Х | х | X |
| | | Did not return for at least one post-<br>baseline visit | Х | X | Х | Х | N= N= N | X |
| | Eligible for PP | | х | X | X | X | X | Х |
| Population Safety Analysis Population Evaluable Analysis Population Per-Protocol (PP) Analysis | | Any Reason | X | X | X | X | X | X |
| | | Did not meet inclusion/exclusion criteria | X | X | X | X | X | X |
| | | Had significant protocol deviations | X | X | X | X | X | X |
| | | Received less than 5 doses of study product | X | X | X | X | Х | X |
| Per-Protocol (PP) Analysis | | Did Not Return for Test of Cure visit | X | X | X | X | X | X |
| | | Out of window Test of Cure visit | X | X | X | X | X | X |
| Analysis | | Discontinued early due to lack of treatment effect | x | X | X | X | х | X |
| Population Eligible for Safety | Excluded from PP | Received systemic antimicrobial therapy other than study drug | Х | х | Х | Х | х | X |
| | Grade 3 Lab Abnormality from Visit 1 | х | x | х | X | х | X | |
| | | Positive HIV, Chlamydia or Neisseria gonorrhoeae test | X | X | X | Х | х | X |
| | | Positive for other concomitant vulvovaginal infections | X | Х | X | X | х | X |
| | | PAP result consistent with HSIL, AGUS, or CIN2 or greater | X | Х | X | X | х | X |
| | | Nugent score < 4 from Visit 1 | Х | X | X | X | х | X |

Note: N=number of enrolled subjects; Treatment group is the actual treatment a subject received

**Subject Disposition by Treatment Group - All Enrolled Subjects** Table 5:

| Subject | ( | aurin Vaginal<br>Gel<br>I=X) | | bo Gel<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|
| Disposition | N | % | n | % | n | % |
| Screened | | | | | X | |
| Enrolled/Randomized | х | 100 | X | 100 | X | 100 |
| Received Treatment | Х | X | X | х | X | X |
| Complied with Treatment <sup>a, b</sup> | х | Х | х | х | X | х |
| Completed Test of Cure Visit,<br>Visit 2 (Study Day 8-15) | X | X | X | X | X | Х |
| Completed Test of Cure Visit Per<br>Protocol <sup>c</sup> | Х | X | Х | X | X | Х |
| Completed Visit 3 (Study Day 22-31) | X | X | X | X | X | Х |
| Completed Visit 3 Per Protocol <sup>c</sup> | X | X | X | X | X | X |

Notes: N=Number of enrolled subjects

aRefer to Listing 1 (16.2.1) for reasons subjects discontinued or terminated early.

b Refer to Listing 9 (16.2.5) for treatment compliance.

<sup>&</sup>lt;sup>c</sup>Refer to Listing 4 (16.2.3) for reasons subjects are excluded from the per protocol population.

Table 6: Distribution of Protocol Deviations by Category, Type, and Treatment Group - All Enrolled Subjects

| | | Vag | 5% Monolaurin<br>Vaginal Gel<br>(N=X) | | | | Gel<br>) | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. |
| Eligibility/enrollment | Any type | Х | Х | Х | Х | Х | Х | Х | х | Х |
| | Did not meet inclusion criterion | Х | х | Х | Х | х | х | Х | х | х |
| | Met exclusion criterion | Х | х | х | х | х | х | х | х | х |
| | ICF not signed prior to study procedures | х | Х | Х | Х | х | Х | Х | х | Х |
| | Other | Х | х | х | Х | х | х | х | х | х |
| Treatment administration schedule | Any type | Х | х | х | х | х | х | х | х | х |
| | Out of window visit | х | Х | Х | Х | х | х | Х | х | Х |
| | Missed visit/visit not conducted | Х | х | х | х | х | х | х | х | х |
| | Missed treatment administration | Х | х | х | х | х | х | х | х | х |
| | Delayed treatment administration | х | Х | Х | Х | х | х | х | х | Х |
| | Other | х | Х | Х | Х | х | х | х | х | Х |
| Follow-up visit schedule | Any type | х | Х | Х | Х | х | х | Х | х | Х |
| | Out of window visit | Х | х | х | х | х | х | х | х | х |
| | Missed visit/visit not conducted | Х | х | х | х | х | х | х | х | х |
| | Other | Х | х | х | х | х | х | х | х | х |
| Protocol procedure/assessment | Any type | Х | х | х | х | х | х | х | х | х |
| | Incorrect version of ICF signed | х | Х | Х | Х | х | х | Х | х | Х |
| | Blood not collected | Х | х | х | х | х | х | х | х | х |
| | Urine not collected | х | Х | Х | Х | х | х | х | х | Х |
| | Other specimen not collected | х | х | х | х | х | х | х | х | х |
| | Specimen result not obtained | х | х | х | Х | х | х | х | х | х |
| | Required procedure not conducted | X | х | Х | Х | х | Х | Х | х | Х |

Table 6: Distribution of Protocol Deviations by Category, Type and Treatment Group – All Enrolled Subjects (continued)

| | | Va | Ionola<br>ginal (<br>(N=X) | Gel | | cebo (<br>N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | Subject (N=X) | # of<br>Dev. |
| | Required procedure done incorrectly | Х | х | Х | Х | Х | х | Х | х | X |
| | Study product temperature excursion | Х | Х | Х | Х | Х | Х | Х | х | X |
| | Specimen temperature excursion | х | Х | Х | Х | Х | Х | Х | х | Х |
| | Other | Х | х | Х | Х | Х | Х | Х | х | X |
| Treatment administration | Any type | Х | Х | х | Х | Х | х | х | х | Х |
| | Required procedure done incorrectly | х | Х | Х | Х | Х | Х | Х | х | Х |
| | Study product temperature excursion | Х | х | х | х | Х | х | х | bj. | х |
| | Other | Х | х | х | х | Х | х | х | х | х |
| Blinding policy/procedure | Any type | Х | х | х | х | х | х | х | х | х |
| | Treatment unblinded | Х | х | х | х | Х | х | х | x x x x x | X |
| | Other | Х | Х | х | х | х | х | х | х | Х |

Notes: N=Number of enrolled subjects. Treatment group is the treatment the subject was randomized to.

Table 7: Summary of Categorical Demographic and Baseline Characteristics by Site - ITT Population

| | | Cincinnati Children's<br>Hospital<br>(N=X) | | University<br>(N= | | | niversity<br>=X) | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % |
| | Not Hispanic or Latino | х | Х | X | х | x | X | X | х |
| Ethnicity | Hispanic or Latino | X | х | х | х | X | X | X | х |
| | Not Reported/Unknown | X | х | х | х | X | X | X | х |
| | American Indian or Alaska Native | х | х | X | х | x | X | X | x |
| | Asian | X | х | х | х | X | X | X | х |
| | Native Hawaiian or Other Pacific Islander | х | X | X | х | X | X | x | x |
| Race | Black or African American | Х | X | X | X | X | X | x | x |
| | White | х | X | X | х | X | x | x | x |
| | Multi-Racial | х | X | X | х | X | x | x | x |
| | Unknown | х | х | х | х | x | X | X | X |

Note: N=number of enrolled subjects

Table 8: Summary of Continuous Demographic and Baseline Characteristic by Site - ITT Population

| Variable | Statistic | Cincinnati Children's<br>Hospital<br>(N=X) | University of Iowa<br>(N=X) | Duke University<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | Mean | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X |
| Age | Median | X.X | X.X | X.X | X.X |
| | Minimum | X | х | X | X |
| | Maximum | X | х | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| Episodes of BV (Including | Standard Deviation | X.X | X.X | X.X | X.X |
| Current Episode) in the | Median | X.X | X.X | X.X | X.X |
| previous 12 months | Minimum | X | х | X | х |
| | Maximum | X | X | X | X |

Notes: N=number of enrolled subjects

Protocol version 7.0 (May 11, 2017) removed exclusion for 6 or more episodes of vaginitis within the past year.

Table 9: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - ITT Population

| | | | in Vaginal Gel<br>=X) | Placebo<br>(N=2 | | All Su<br>(N= | |
|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % |
| | Not Hispanic or Latino | x | x | X | X | X | Х |
| Ethnicity | Hispanic or Latino | x | x | X | X | X | Х |
| | Not Reported/Unknown | X | X | X | X | X | Х |
| | American Indian or Alaska Native | x | x | X | X | X | Х |
| | Asian | x | x | X | X | X | Х |
| | Native Hawaiian or Other Pacific Islander | x | x | X | X | X | Х |
| Race | Black or African American | x | x | X | X | X | Х |
| | White | x | x | X | X | X | х |
| | Multi-Racial | x | х | X | X | X | х |
| | Unknown | x | x | X | X | X | х |

Note: N=number of enrolled subjects

**Table 10:** Summary of Continuous Baseline Characteristics by Treatment Group - ITT Population

| Variable | Statistic | 5% Monolaurin Vaginal Gel<br>(N=X) | Placebo Gel<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | Mean | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X |
| Age (Years) | Median | X | X | X |
| | Minimum | X | X | х |
| | Maximum | X | X | х |
| | Mean | X.X | X.X | X.X |
| Episodes of BV (Including | Standard Deviation | X.X | X.X | X.X |
| Current Episode) in the previous | Median | X.X | X.X | X.X |
| 12 months | Minimum | X | X | х |
| | Maximum | X | Х | Х |

Notes: N=number of enrolled subjects

Protocol version 7.0 (May 11, 2017) removed exclusion for 6 or more episodes of vaginitis within the past year.

**Table 11:** Baseline Sexual History by Site - ITT Population

| Sexual History Category | Value | Children | cinnati<br>'s Hospital<br>I=X) | Univer<br>Iov<br>(N= | va | Dul<br>Univer<br>(N=) | rsity | All Subj<br>(N=X | |
|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % |
| Subject has received treatment for previous episodes of BV in the | Yes | х | х | х | X | х | х | X | х |
| previous 12 months | No | X | X | x | X | х | х | X | х |
| Subject is sexually active | Yes | X | x | x | X | X | х | X | х |
| | No | X | X | X | X | X | X | X | x |
| | Unknown | X | X | X | X | X | X | X | X |
| Subject's sexual orientation* | Heterosexual | X | X | X | X | X | X | X | X |
| | Gay/Homosexual | X | X | X | X | X | X | X | X |
| | Bisexual | х | х | x | X | х | х | X | X |
| | Unknown | х | х | x | X | х | х | X | х |
| Subject has had sex with men or women in the past 12 months* | Men | х | х | x | X | х | х | X | х |
| | Women | х | х | x | X | х | х | X | х |
| | Both | х | х | x | X | х | х | X | х |
| | Neither | х | х | x | X | х | х | X | х |
| | Unknown | х | х | x | X | х | х | X | х |
| Subject has had vaginal intercourse in the past 12 months* | Yes | х | х | х | X | х | х | X | х |
| | No | х | х | x | X | х | х | X | х |
| | Unknown | х | х | х | X | х | х | X | х |
| Subject has had receptive oral intercourse in the past 12 months* | Yes | X | х | x | X | х | х | X | х |
| | No | x | x | x | X | х | X | X | X |
| | Unknown | X | х | x | X | х | х | X | х |
| Subject has had receptive anal intercourse in the past 12 months* | Yes | х | х | х | Х | х | х | X | х |
| | No | х | х | х | х | х | х | х | х |
| | Unknown | х | Х | х | X | Х | Х | Х | Х |

Notes: N=number of enrolled subjects. \*Denominator for percentages is the number of subjects who were sexually active in the respective site.

 Table 12:
 Baseline Sexual History by Treatment Group - ITT Population

| | | | urin Vaginal Gel<br>(N=X) | | ebo Gel<br>N=X) | | ubjects<br>N=X) |
|---|---|---|---|---|---|---|---|
| Sexual History Category | Value | n | % | n | % | n | % |
| Chief he was in the stand Committee with the CDV in the way in 12 words 2 | Yes | Х | х | х | Х | х | х |
| Subject has received treatment for previous episodes of BV in the previous 12 months? | No | Х | х | х | Х | х | х |
| | Yes | Х | х | х | Х | х | х |
| Subject is sexually active | No | Х | х | х | X | х | х |
| | Unknown | Х | х | х | X | х | х |
| | Heterosexual | Х | x | х | X | X | X |
| Cubication and animatetics.* | Gay/Homosexual | Х | х | х | X | х | X |
| Subject's sexual orientation* | Bisexual | Х | х | х | X | х | х |
| | Unknown | Х | х | х | X | х | х |
| | Men | Х | x | х | X | X | X |
| | Women | Х | x | х | X | х | X |
| Subject has had sex with men or women in the past 12 months* | Both | Х | x | х | X | X | X |
| | Neither | Х | x | х | X | х | X |
| | Unknown | Х | x | х | X | х | X |
| | Yes | Х | x | х | X | х | X |
| Subject has had vaginal intercourse in the past 12 months* | No | Х | x | х | X | х | X |
| | Unknown | Х | x | х | X | х | X |
| | Yes | Х | x | х | X | х | х |
| Subject has had receptive oral intercourse in the past 12 months* | No | X | х | х | Х | х | х |
| | Unknown | Х | х | х | Х | х | х |
| | Yes | Х | х | х | Х | х | х |
| Subject has had receptive anal intercourse in the past 12 months* | No | х | х | Х | Х | х | х |
| | Unknown | Х | х | х | Х | х | х |

Notes: N=number of enrolled subjects. \*Denominator for percentages is the number of subjects who were sexually active in the respective treatment group.

**Table 13:** Summary of Baseline Clinical Assessment of BV by Site - Safety Population

| | | Cinc | inna | | nildr<br>N=X) | en's Ho<br>) | spit | al | | | Un | | sity<br>N=3 | of Iowa<br>K) | | | | | D | | Unive<br>N=X) | rsity | | | | | 1 | | ubjec<br>=X) | ets | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | one | M | lild | Mo | derate | Se | vere | N | one | N | Iild | M | oderate | Se | evere | N | one | N | Iild | Mod | lerate | Se | vere | N | one | N | Iild | Mod | lerat | e Se | vere |
| Sign/Symptom | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Sign/Symptom <sup>1</sup> | x | x | X | x | x | x | x | x | x | x | x | x | X | X | х | X | x | X | X | x | x | X | X | x | x | х | х | х | х | х | х | х |
| Vaginal Odor | X | x | X | х | x | x | x | х | x | х | х | x | X | x | X | X | х | x | X | x | x | x | X | x | х | х | х | х | х | х | х | х |
| Vaginal Pain | x | x | X | x | x | x | x | x | x | x | x | x | X | X | х | X | x | X | X | x | x | X | X | x | x | х | х | х | х | х | х | х |
| Vaginal Tenderness | X | x | X | x | x | x | X | х | X | x | х | x | X | x | х | X | х | x | X | x | x | x | X | x | х | х | х | х | х | х | х | х |
| Vulvar/Vaginal<br>Itching | x | х | x | X | X | X | X | X | x | X | x | х | X | х | x | x | x | x | x | X | x | х | х | х | Х | X | Х | Х | X | х | х | х |
| Vaginal Dryness | x | x | x | x | x | x | x | x | x | x | x | x | X | X | x | X | x | х | x | x | x | x | X | x | x | х | x | х | х | х | х | х |
| Vaginal Discharge | x | x | x | x | x | x | X | x | X | x | x | X | x | X | x | x | х | x | X | x | x | x | X | X | х | х | х | х | х | x | х | х |
| Vulvar Inflammation | X | X | х | x | x | x | x | х | X | х | х | х | X | X | X | X | х | X | x | X | х | x | X | X | х | Х | х | х | х | х | Х | Х |

Notes: Denominator for percentages is the number of subjects in the Safety Population (N) for each Site.

Assessment is performed by the clinician.

¹The maximum severity of any sign or symptom is summarized. A subject is only counted once at the maximum severity.

Table 14: Summary of Baseline Clinical Assessment of BV by Treatment Group - Safety Population

| | | 59 | % Mo | | in Va<br>=X) | ginal G | Gel | | | | | | bo Ge<br>=X) | l | | | | | | All Su<br>(N: | ibjects<br>=X) | 3 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | one | M | lild | Mod | erate | Sev | vere | N | one | M | lild | Mod | lerate | Se | vere | N | one | M | ild | Mod | erate | Sev | vere |
| Sign/Symptom | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Sign/Symptom <sup>1</sup> | х | х | Х | х | X | х | X | х | Х | х | Х | х | Х | х | Х | х | Х | х | X | Х | Х | X | X | х |
| Vaginal Odor | х | х | X | x | X | х | X | х | Х | х | Х | х | Х | х | Х | х | Х | х | X | Х | X | x | Х | х |
| Vaginal Pain | х | х | X | х | X | x | X | х | X | х | Х | х | Х | х | Х | х | X | х | X | X | X | x | X | х |
| Vaginal Tenderness | х | х | X | x | X | х | X | х | Х | х | Х | х | Х | х | Х | х | Х | х | Х | Х | X | x | Х | х |
| Vulvar/Vaginal Itching | х | х | X | x | Х | х | X | х | Х | х | Х | х | Х | х | Х | х | Х | х | х | Х | Х | Х | X | х |
| Vaginal Dryness | х | х | Х | x | Х | х | X | х | Х | x | Х | x | Х | х | Х | x | Х | х | х | Х | Х | X | X | х |
| Vaginal Discharge | х | х | X | х | Х | х | X | х | Х | х | Х | х | х | х | х | х | Х | х | X | х | Х | х | X | х |
| Vulvar Inflammation | Х | х | Х | X | Х | x | X | Х | Х | x | Х | х | х | х | х | x | Х | х | X | Х | Х | X | X | х |

Notes: Denominator for percentages is the number of subjects in the Safety Population (N) for each treatment group. Assessment is performed by the clinician.

<sup>&</sup>lt;sup>1</sup>The maximum severity of any sign or symptom is summarized. A subject is only counted once at the maximum severity.

Table 15: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population - All Sites

| | 5% Mon<br>Vagina<br>(N= | al Gel | | bo Gel<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % |
| Any SOC | X | X | X | X | X | X |
| [SOC 1] | X | X | X | X | X | Х |
| [SOC 2] | X | X | X | X | Х | Х |

Notes: N=number of enrolled subjects.

A subject is only counted once per SOC.

#### Tables with Similar Format:

- Table 16: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group -ITT Population- Cincinnati Children's Hospital
- Table 17: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA
  System Organ Class and Treatment Group -ITT Population- University of
  Iowa
- Table 18: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group -ITT Population-Duke University

n = Number of subjects reporting medical history within the specified SOC.

**Table 19:** Dates of First Treatment by Site - Safety Population

[Note: Dates will be categorized by breaking the calendar year into quarters.]

| Dates of Dosing | Н | ati Children's<br>ospital<br>N = X) | | sity of Iowa<br>N = X) | | University<br>N = X) | | Subjects<br>N = X) |
|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % |
| DDMMMYYYY-DDMMMYYYY | Х | Х | Х | X | X | X | X | x |
| DDMMMYYYY-DDMMMYYYY | Х | Х | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | Х | Х | Х | X | X | X | X | x |
| DDMMMYYYY-DDMMMYYYY | Х | Х | Х | X | X | X | X | x |

Note: N=Number of subjects in the safety population

#### **Table 20:** Dates of First Treatment by Treatment Group - Safety Population

[Note: Dates will be categorized by breaking the calendar year into quarters.]

| Dates of Dosing | | laurin Vaginal Gel<br>(N = X) | | lacebo Gel<br>(N = X) | | l Subjects<br>(N = X) |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |

Note: N=Number of subjects in the safety population

Table 21: Dose Administration Schedule by Site and Number of Doses Administered - Safety Population

| | | | Number | of Doses Administe | ered n (%) | | |
|---|---|---|---|---|---|---|---|
| Dose Administration Schedule | 0<br>(N=X) | 1<br>(N=X) | 2<br>(N=X) | 3<br>(N=X) | 4<br>(N=X) | 5<br>(N=X) | 6<br>(N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| University of Iowa (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| Dose Administration Schedule | 0<br>(N=X) | 1<br>(N=X) | 2<br>(N=X) | 3<br>(N=X) | 4<br>(N=X) | 5<br>(N=X) | 6<br>(N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Duke University (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Dose Administration Schedule</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| Dose Administration Schedule | 0<br>(N=X) | 1<br>(N=X) | 2<br>(N=X) | 3<br>(N=X) | 4<br>(N=X) | 5<br>(N=X) | 6<br>(N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Site who received the specified number of doses.

**Table 22:** Dose Administration Schedule by Site and Dose Number - Safety Population

| Site | Dose Administration<br>Schedule | Dose 1<br>n (%) | Dose 2<br>n (%) | Dose 3<br>n (%) | Dose 4<br>n (%) | Dose 5<br>n (%) | Dose 6<br>n (%) |
|---|---|---|---|---|---|---|---|
| Cincinnati Children's Hospital | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| (N=X) | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| University of Iowa (N=X) | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Duke University (N=X) | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Site

Table 23: Dose Administration Schedule by Treatment Group and Number of Doses Administered - Safety Population

| 5% Monolaurin Vaginal Gel (N=X) | | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Number of Doses Administered n (%) | | | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Dose Administration Schedule</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Placebo Gel (N=X) | | | | | | | |
| | | | Number o | of Doses Administer | red n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Dose Administration Schedule</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | | | | | | | |
| | | | Number o | of Doses Administer | red n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Dose Administration Schedule</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Treatment Group who received the specified number of doses.

Table 24: Dose Administration Schedule by Treatment Group and Dose Number - Safety Population

| Site | Dose Administration<br>Schedule | Dose 1<br>n (%) | Dose 2<br>n (%) | Dose 3<br>n (%) | Dose 4<br>n (%) | Dose 5<br>n (%) | Dose 6<br>n (%) |
|---|---|---|---|---|---|---|---|
| 50/1/ | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| 5% Monolaurin Vaginal Gel (N=X) | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| (IV A) | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Placebo Gel (N=X) | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | As scheduled | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | Out of Window | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missed | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Treatment Group

Table 25: Product Administration Position by Site and Number of Doses Administered - Safety Population

| | Number of Doses Administered n (%) | | | | | | |
|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Product Administration Position</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| University of Iowa (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Product Administration Position</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Duke University (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Product Administration Position</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | | | | | | | |
| | | | Number | of Doses Administe | ered n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | ON NO | (N=X) | (N=X) | (N=X) | (N=X) |
| <b>Product Administration Position</b> | (N=X) | (N=X) | (N=X) | (IV-A) | (11 12) | (1, 12) | (-,) |
| Product Administration Position Recumbent | (N=X)<br>x (x) | (N=X)<br>x (x) | (N=X)<br>x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Site who received the specified number of doses.

**Table 26:** Product Administration Position by Site and Dose Number - Safety Population

| Site | Product Administration<br>Position | Dose 1<br>n (%) | Dose 2<br>n (%) | Dose 3<br>n (%) | Dose 4<br>n (%) | Dose 5<br>n (%) | Dose 6<br>n (%) |
|---|---|---|---|---|---|---|---|
| Cincinnati Children's Hospital | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| (N=X) | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| University of Iowa (N=X) | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Duke University (N=X) | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Site

Table 27: Product Administration Position and Number of Doses Administered - Safety Population

| 5% Monolaurin Vaginal Gel (N=X) | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Number of Doses Administered n (%) | | | | | | |
| Due due et Administration Decition | 0 | 1 | 2 | 3 | 4 | 5<br>(N. V) | 6 |
| Product Administration Position | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Placebo Gel (N=X) | | | | | | | |
| | | | Number ( | of Doses Administer | red n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Product Administration Position</b> | · · · | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | | | | | | | |
| | | | Number ( | of Doses Administer | red n (%) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <b>Product Administration Position</b> | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Treatment Group who received the specified number of doses.

**Table 28:** Product Administration Position by Treatment Group and Dose Number - Safety Population

| Site | Product Administration<br>Position | Dose 1<br>n (%) | Dose 2<br>n (%) | Dose 3<br>n (%) | Dose 4<br>n (%) | Dose 5<br>n (%) | Dose 6<br>n (%) |
|---|---|---|---|---|---|---|---|
| 50/3/ | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| 5% Monolaurin Vaginal Gel (N=X) | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| Placebo Gel (N=X) | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| All Subjects (N=X) | Not Recumbent | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Missing | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |

Note: Denominator for percentages is the number of subjects in the Safety Population for each Treatment Group

## **Section 14.2 Efficacy Data**

Table 29: Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group

| Analysis<br>Population | Treatment<br>Group | Number of<br>Subjects with<br>Clinical Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Clinical Cure | Proportion of<br>Subjects with<br>Clinical Cure<br>95% CI | Difference in Proportion<br>of Subjects with Clinical<br>Cure between 5%<br>Monolaurin Vaginal Gel<br>and Placebo Gel | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI | P-Value* |
|---|---|---|---|---|---|---|---|---|
| | 5% Monolaurin<br>Vaginal Gel | x | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| ITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | | |
| | 5% Monolaurin<br>Vaginal Gel | x | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| mITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | | |
| | 5% Monolaurin<br>Vaginal Gel | x | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Evaluable | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | | |
| | 5% Monolaurin<br>Vaginal Gel | х | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| PP | Placebo Gel | х | х | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | х | Х | 0.xx | 0.xx, 0.xx | | | |

Notes: The denominator for proportions is based on the number of subjects enrolled in the respective treatment group and analysis population.

<sup>\*</sup>P-value from the Fisher's exact two-sided test at the .05 level of significance.

Table 30: Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group

| Analysis<br>Population | Treatment Group | Number of<br>Subjects with<br>Clinical Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Clinical Cure | Proportion of<br>Subjects with<br>Clinical Cure<br>95% CI | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|---|
| | 5% Monolaurin<br>Vaginal Gel | x | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| ITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | X | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| mITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Evaluable | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | x | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| PP | Placebo Gel | х | Х | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |

Note: The denominator for proportions is based on the number of subjects enrolled in the respective treatment group and analysis population.

Table 31: Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group

| Analysis<br>Population | Treatment Group | Number of<br>Subjects with<br>Therapeutic<br>Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Therapeutic<br>Cure | Proportion of<br>Subjects with<br>Clinical Cure<br>95% CI | Difference in Proportion of<br>Subjects with Therapeutic Cure<br>between 5% Monolaurin Vaginal<br>Gel and Placebo Gel | Difference in Proportion of<br>Subjects with Therapeutic Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|---|
| | 5% Monolaurin<br>Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| ITT | Placebo Gel | х | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | x | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| mITT | Placebo Gel | X | x | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | х | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | X | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Evaluable | Placebo Gel | Х | Х | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | Х | Х | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | х | х | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| PP | Placebo Gel | х | х | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | Х | х | 0.xx | 0.xx, 0.xx | | |

Note: The denominator for proportions is based on the number of subjects enrolled in the respective treatment group and analysis population.

Table with similar format:

Table 32: Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group

Table 33: Summary of Amsel Criteria by Site and Study Visit - All Enrolled Subjects

| | | ( | Cincinnati Children's<br>Hospital<br>(N=X) | | | | | University of Iowa<br>(N=X) | | | | | | Duke University<br>(N=X) | | | | | | | All Subjects<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Amsel Criteria | | | sit 1<br>=X) | | sit 2<br>=X) | | sit 3<br>(=X) | | sit 1<br>=X) | | Visit 2<br>(N=X) | | Visit 3<br>(N=X) | | Visit 1<br>(N=X) | | sit 2<br>=X) | | sit 3<br>=X) | | sit 1<br>=X) | | | | sit 3<br>=X) |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | 0/4 | Х | Х | х | X | x | Х | х | Х | Х | X | Х | Х | х | Х | х | Х | X | X | Х | Х | Х | Х | X | Х |
| | 1/4 | X | Х | Х | х | Х | х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | X | Х | Х | Х | Х |
| Number of Amsel Criteria Present | 2/4 | X | X | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | X | Х | X | X | Х | Х | Х | Х | Х | Х | Х |
| | 3/4 | X | X | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | X | Х | X | X | Х | Х | Х | Х | Х | Х | Х |
| | 4/4 | X | X | X | х | X | х | X | Х | Х | Х | Х | Х | X | X | X | Х | X | Х | Х | Х | Х | Х | Х | Х |
| Vaginal Secretion pH | >4.5 | X | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | X | Х | Х | X | X | Х | Х | X | Х | Х | Х | Х |
| vaginal Secretion pri | ≤4.5 | X | Х | Х | х | Х | х | Х | х | Х | Х | Х | Х | Х | Х | Х | X | X | х | Х | Х | Х | х | Х | х |
| Clue Cells | ≥20% | X | Х | Х | х | X | х | X | Х | Х | Х | Х | Х | X | Х | Х | Х | X | Х | Х | Х | Х | х | Х | Х |
| Cide Cells | <20% | X | Х | Х | х | Х | х | Х | х | Х | Х | Х | Х | Х | Х | Х | X | X | х | Х | Х | Х | х | Х | х |
| Amine ("whiff") test on KOH wet | Positive | X | Х | Х | х | X | х | X | Х | Х | Х | Х | Х | X | Х | Х | Х | X | Х | Х | Х | Х | х | Х | Х |
| mount | Negative | X | Х | Х | х | X | х | X | Х | Х | х | Х | Х | X | Х | Х | Х | X | х | Х | х | Х | Х | Х | Х |
| Off-white (milky or gray), thin, | Yes | X | Х | Х | х | X | х | X | Х | Х | Х | Х | Х | X | Х | Х | Х | X | Х | Х | Х | Х | х | Х | Х |
| homogenous discharge | No | X | Х | Х | Х | X | Х | X | Х | Х | Х | Х | Х | X | Х | Х | X | X | Х | Х | Х | Х | Х | Х | Х |

Note: Denominator for percentages is the number of subjects enrolled (N) in the study for each Site.
Table 34: Summary of Amsel Criteria by Treatment Group and Study Visit - ITT Population

| | | 59 | % Moi | | rin Va<br>=X) | ginal | Gel | | ] | | bo Ge<br>=X) | el | | | A | | ubject<br>=X) | S | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Amsel Criteria | | | sit 1<br>=X) | | sit 2<br>=X) | | sit 3<br>(=X) | | sit 1<br>=X) | | sit 2<br>=X) | | sit 3<br>=X) | | sit 1<br>=X) | | sit 2<br>(=X) | | sit 3<br>=X) |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | 0/4 | Х | X | Х | X | Х | Х | X | X | Х | X | Х | Х | X | Х | Х | Х | X | Х |
| | 1/4 | Х | Х | Х | Х | Х | Х | Х | X | Х | X | Х | Х | Х | X | х | Х | Х | Х |
| Number of Amsel Criteria Present | 2/4 | Х | Х | Х | Х | Х | Х | Х | X | Х | X | Х | Х | Х | X | х | Х | X | Х |
| | 3/4 | Х | X | Х | X | Х | х | X | X | X | X | X | X | X | X | Х | Х | X | Х |
| | 4/4 | Х | X | Х | X | Х | X | Х | X | Х | X | Х | X | Х | X | X | Х | X | Х |
| Vaginal Secretion pH | >4.5 | Х | X | Х | х | Х | Х | Х | X | Х | X | Х | Х | Х | Х | Х | Х | X | Х |
| vaginar secretion pri | ≤4.5 | Х | X | Х | Х | Х | X | X | X | X | X | X | X | X | X | X | Х | X | Х |
| Clue Cells | ≥20% | Х | X | Х | Х | Х | X | X | X | X | X | X | X | X | X | X | Х | X | Х |
| Cide Celis | <20% | Х | X | Х | Х | Х | Х | Х | X | Х | X | Х | Х | Х | Х | х | Х | X | Х |
| Amine ("whiff") test on KOH wet mount | Positive | Х | X | Х | х | Х | Х | Х | X | Х | X | Х | Х | Х | Х | Х | Х | X | Х |
| Annue (winn ) test on Korr wet mount | Negative | х | X | Х | Х | Х | Х | Х | X | х | Х | Х | Х | Х | Х | Х | Х | х | Х |
| Off-white (milky or gray), thin, homogenous discharge | Yes | Х | X | Х | X | Х | Х | Х | X | Х | X | Х | Х | Х | X | X | Х | Х | Х |
| On-write (minky or gray), that, nonlogenous discharge | No | Х | X | Х | X | Х | Х | Х | X | х | X | х | Х | х | X | X | Х | X | Х |

Note: Denominator for percentages is the number of subjects enrolled (N) in the study for each treatment group.

#### Tables with similar format:

Table 35: Summary of Amsel Criteria by Treatment Group and Study Visit - mITT Population

Table 36: Summary of Amsel Criteria by Treatment Group and Study Visit - Evaluable Population

Table 37: Summary of Amsel Criteria by Treatment Group and Study Visit - PP Population

Table 38: Nugent Scores by Category, Study Visit, Analysis Population, and Site – All Subjects

| | | | | | | All Subjects<br>(N = X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Nugent Score | | Visit 1 (N = X) | | | Visit 2<br>(N = X) | | | Visit 3<br>(N = X) | |
| Population | Category | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI |
| | 0-3 (Normal) | х | 0.xx | 0.xx, 0.xx | х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| ITT | 4-6 (Intermediate) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| mITT | 4-6 (Intermediate) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| Evaluable | 4-6 (Intermediate) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| PP | 4-6 (Intermediate) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |

Note: Denominator for percentages is the number of subjects enrolled (N) in the study for each Site.

## Tables with Similar Format:

Table 39: Nugent Scores by Category, Study Visit, Analysis Population, and Site—Cincinnati Children's Hospital

Table 40: Nugent Scores by Category, Study Visit, Analysis Population, and Site—University of Iowa

Table 41: Nugent Scores by Category, Study Visit, Analysis Population, and Site—Duke University

Table 42: Nugent Scores by Category, Study Visit, Analysis Population, and Treatment Group - 5% Monolaurin Vaginal Gel

| | | | | | 5% I | Monolaurin Vag<br>(N = X) | inal Gel | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Nugent Score | | Visit 1 (N = X) | | | Visit 2 (N = X) | | | Visit 3 (N = X) | |
| Population | Category | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI | Number<br>of<br>Subjects<br>n | Proportion of Subjects | Proportion<br>of Subjects<br>95% CI |
| | 0-3 (Normal) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| ITT | 4-6 (Intermediate) | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | Х | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx |
| mITT | 4-6 (Intermediate) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| Evaluable | 4-6 (Intermediate) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 0-3 (Normal) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| PP | 4-6 (Intermediate) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |
| | 7-10 (BV) | X | 0.xx | 0.xx, 0.xx | X | 0.xx | 0.xx, 0.xx | Х | 0.xx | 0.xx, 0.xx |

Note: Denominator for percentages is the number of subjects enrolled (N) in the study for each treatment group.

Tables with Similar Format:

Table 43: Nugent Scores by Category, Study Visit, Analysis Population, and Treatment Group - Placebo Gel

Continuous Nugent Score Characteristics by Study Visit, Analysis Population, and Treatment Group **Table 44:** 

| | | 5% Mon | olaurin Va<br>(N=X) | ginal Gel | I | Placebo Ge<br>(N=X) | l | A | All Subject<br>(N = X) | s |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Population | Statistic | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) |
| | Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| ITT | Standard Deviation of Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| 11 1 | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | x.xx |
| mITT | Standard Deviation of Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | x.xx |
| mii i | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | x.xx |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Evaluable | Standard Deviation of Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Evaluable | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| рр | Standard Deviation of Mean | x.xx | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| rr | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |

Nugent Scores by Category, Study Visit, Clinical Cure Status, and Treatment Group -ITT Population **Table 45:** 

| | | | 5% M | | urin Va<br>N=X) | ginal G | el | | | | cebo Ge<br>N=X) | l | | | | | Subjects<br>= xxx) | S | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Nugent Score<br>Category | C | nical<br>ure<br>= X) | Fai | nical<br>ilure<br>= X) | Eva | Not<br>luable<br>= X) | C | nical<br>ure<br>= X) | Fai | nical<br>ilure<br>= X) | Eva | Not<br>luable<br>= X) | C | nical<br>ure<br>= X) | Fa | nical<br>ilure<br>= X) | Eva | Not<br>luable<br>= X) |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| *** | 0-3 (Normal) | X | X | X | X | Х | X | X | Х | X | Х | X | Х | Х | X | Х | Х | Х | Х |
| Visit 2<br>Test of Cure | 4-6 (Intermediate) | X | X | X | X | X | X | X | X | X | X | X | Х | х | X | Х | X | X | X |
| | 7-10 (BV) | X | X | X | X | X | X | X | X | X | X | X | Х | х | X | Х | X | X | X |
| | 0-3 (Normal) | X | X | X | X | X | X | X | X | X | X | X | Х | х | X | Х | X | X | X |
| Visit 3 | 4-6 (Intermediate) | X | X | Х | X | X | X | Х | Х | Х | X | X | Х | Х | X | Х | X | Х | X |
| | 7-10 (BV) | X | X | Х | Х | X | X | X | Х | X | Х | Х | Х | X | X | Х | Х | Х | X |

Note: Denominator for percentages is the number of subjects in the ITT population for each treatment group.

Table 46: Continuous Nugent Score Characteristics by Study Visit, Clinical Cure Status, and Treatment Group-ITT Population

| | | 5% M | onolaurin Vag<br>(N=X) | ginal Gel | | Placebo Gel<br>(N=X) | | | All Subjects (N = X) | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Visit | Statistic | Clinical<br>Cure<br>(N = X) | Clinical<br>Failure<br>(N = X) | Not<br>Evaluable<br>(N = X) | Clinical<br>Cure<br>(N = X) | Clinical<br>Failure<br>(N = X) | Not<br>Evaluable<br>(N = X) | Clinical<br>Cure<br>(N = X) | Clinical<br>Failure<br>(N = X) | Not<br>Evaluable<br>(N = X) |
| | Mean | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Visit 2<br>Test of | Standard Deviation of<br>Mean | x.xx | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx | X.XX | X.XX |
| Cure | Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of<br>Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Visit 3 | Standard Deviation of<br>Mean | x.xx | X.XX | X.XX | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX |
| v 151t 3 | Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of<br>Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |

Table 47: Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group - First Time BV

| Analysis<br>Population | Treatment Group | Number of<br>Subjects with<br>Clinical Cure<br>n | Number of<br>Subjects<br>N | Proportion<br>of Subjects<br>with Clinical<br>Cure | Proportion of<br>Subjects with<br>Clinical Cure<br>95% CI | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin Vaginal<br>Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|---|
| | 5% Monolaurin<br>Vaginal Gel | х | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| ITT | Placebo Gel | x | X | 0.xx | 0.xx, 0.xx | 1 | 1 |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | х | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| mITT | Placebo Gel | x | X | 0.xx | 0.xx, 0.xx | 1 | 1 |
| | All Subjects | x | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | x | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Evaluable | Placebo Gel | х | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | х | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin<br>Vaginal Gel | х | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| PP | Placebo Gel | х | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | Х | X | 0.xx | 0.xx, 0.xx | | |

Note: The denominator for proportions is based on the number of subjects with first time BV enrolled in the respective treatment group and analysis population.

## Tables with similar format:

Table 48: Clinical Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group - Recurrent BV

Table 49: Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group - First Time BV

Table 50: Clinical Cure Results at Visit 3 by Analysis Population and Treatment Group - Recurrent BV

Table 51: Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group - First Time BV

| Analysis<br>Population | Treatment Group | Number of<br>Subjects with<br>Therapeutic<br>Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Therapeutic<br>Cure | Proportion of<br>Subjects with<br>Therapeutic<br>Cure<br>95% CI | Difference in Proportion of<br>Subjects with Therapeutic<br>Cure between 5%<br>Monolaurin Vaginal Gel and<br>Placebo Gel | Difference in Proportion of<br>Subjects with Therapeutic Cure<br>between 5% Monolaurin Vaginal<br>Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|---|
| | 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| ITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| mITT | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Evaluable | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
| | 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| PP | Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| N. T. I | All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |

Note: The denominator for proportions is based on the number of subjects with first time BV enrolled in the respective treatment group and analysis population.

#### Tables with similar format:

Table 52: Therapeutic Cure Results at the Test of Cure Visit, Visit 2 by Analysis Population and Treatment Group - Recurrent BV

Table 53: Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group - First Time BV

Table 54: Therapeutic Cure Results at Visit 3 by Analysis Population and Treatment Group - Recurrent BV

Table 55: Clinical Cure Results at the Test of Cure Visit, Visit 2 by Treatment Group- Recumbent Subjects - PP Population

| Treatment Group | Number of<br>Subjects with<br>Clinical Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Clinical Cure | Clinical Cure | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo<br>Gel | Difference in Proportion of Subjects with<br>Clinical Cure between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|
| 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| All Subjects | x | X | 0.xx | 0.xx, 0.xx | | |

Notes: The denominator for proportions is based on the number of subjects enrolled in the PP population\* in the respective treatment group.

In this analysis, the PP population, has the additional stipulation that the subject remain in the recumbent position for 5 of 6 doses to be considered compliant with study product

Table 56: Clinical Cure Results at the Test of Cure Visit, Visit 2 by Treatment Group Using Imputation - mITT Population

| Treatment Group | Number of<br>Subjects with<br>Clinical Cure<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Clinical Cure | Proportion of<br>Subjects with<br>Clinical Cure<br>95% CI | Difference in Proportion of<br>Subjects with Clinical Cure<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel | Difference in Proportion of Subjects with<br>Clinical Cure between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|
| 5% Monolaurin Vaginal Gel | х | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| All Subjects | X | Х | 0.xx | 0.xx, 0.xx | | |

Notes: The denominator for proportions is based on the number of subjects enrolled in the mITT population\* in the respective treatment group.

<sup>\*</sup>In this analysis, subjects in the 5% Monolaurin Vaginal Gel arm who are not evaluable for clinical cure will have their cure status imputed as a clinical failure and subjects in the placebo arm who are not evaluable for clinical cure will have their cure status imputed as a clinical cure.

Table 57: Mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.* by Study Visit, and Treatment Group - ITT Population

| | | 5% Mon | olaurin Va<br>(N=X) | ginal Gel | ] | Placebo Ge<br>(N=X) | el | 1 | All Subject<br>(N = X) | s |
|---|---|---|---|---|---|---|---|---|---|---|
| Species | Statistic | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3 (N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3 (N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3 (N = X) |
| | Mean | x.xx | x.xx | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX |
| Lastabasillua ann | Standard Deviation of Mean | x.xx | x.xx | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX |
| Lactobacillus spp. | Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | x.xx |
| | Mean | x.xx | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX |
| C d 11 | Standard Deviation of Mean | x.xx | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX |
| Gardnerella spp | Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | X.XX | X.XX | | x.xx | X.XX | | x.xx | X.XX |
| | Mean | x.xx | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX |
| Makilonana | Standard Deviation of Mean | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| Mobiluncus spp | Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | x.xx |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | X.XX |

#### Tables with similar format:

- Table 58: Mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.* by Study Visit, and Treatment Group mITT Population
- Table 59: Mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.* by Study Visit, and Treatment Group Evaluable Population
- Table 60: Mean count of *Lactobacillus spp.*, *Gardnerella spp.*, and *Mobiluncus spp.* by Study Visit, and Treatment Group PP Population

Table 61: Mean fungal colony count of *Candida Spp.* by Study Visit, Analysis Population, and Treatment Group in Subjects with Candida spp. Identified at Screening

| | | 5% Mon | olaurin Va<br>(N=X) | ginal Gel | ] | Placebo Ge<br>(N=X) | l | A | All Subject<br>(N = X) | s |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Population | Statistic | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) | Visit 1 (N = X) | Visit 2 (N = X) | Visit 3<br>(N = X) |
| | Mean | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx |
| ITT | Standard Deviation of Mean | X.XX | x.xx | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX |
| 111 | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx |
| mITT | Standard Deviation of Mean | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx |
| miii | Mean Change from Visit 1 | | x.xx | x.xx | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX | X.XX |
| Evaluable | Standard Deviation of Mean | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx |
| Evaluable | Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | x.xx | | X.XX | x.xx |
| | Standard Deviation of Mean Change from Visit 1 | | X.XX | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Mean | x.xx | x.xx | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX |
| PP | Standard Deviation of Mean | X.XX | x.xx | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| rr | Mean Change from Visit 1 | | x.xx | X.XX | | X.XX | X.XX | | X.XX | X.XX |
| | Standard Deviation of Mean Change from Visit 1 | | x.xx | x.xx | | x.xx | x.xx | | x.xx | x.xx |

## **Section 14.3 Safety Data**

Table 62: Number and Percentage of Subjects Experiencing Treatment Emergent Solicited Urogenital Adverse Events with 95% Confidence Intervals by Symptom and Treatment Group - Safety Population

| | 5% Mo | onolaurin<br>(N=X | Vaginal Gel<br>) | | Placeb<br>(N= | | All Subjects (N=X) | | |
|---|---|---|---|---|---|---|---|---|---|
| Solicited Urogenital Adverse Event | n | n % 95% CI | | | | 95% CI | n | % | 95% CI |
| Any Solicited Adverse Event | х | Х | x, x | х | Х | х, х | X | X | x, x |
| Vaginal Odor | Х | Х | X, X | х | Х | x, x | x x | | x, x |
| Vaginal Pain | х | Х | X, X | x x x, x | | х | X | x, x | |
| Vaginal Tenderness | х | Х | X, X | х | X | x, x | х | X | x, x |
| Vulvar/Vaginal Itching | х | Х | X, X | х | X | x, x | х | X | x, x |
| Vaginal Dryness | х | Х | X, X | х | X | x, x | х | X | x, x |
| Vaginal Discharge | х | Х | X, X | x x x, x | | x, x | X | X | x, x |
| Vulvar Inflammation | х | Х | X, X | x | Х | x, x | X | X | x, x |

Notes: N = number of subjects in the Safety Analysis Population who received the specified treatment.

A subject is only counted once per solicited adverse event.

This table presents number and percentage of subjects.

Table 63: Comparison of the Proportion of Subjects Experiencing Treatment Emergent Solicited Urogenital Adverse Events through the Test of Cure Visit, Visit 2 by Treatment Group - Safety Population

| Solicited<br>Urogenital<br>Adverse Event | Treatment<br>Group | Proportion of<br>Subjects<br>Experiencing<br>Solicited Event | Proportion of<br>Subjects<br>Experiencing<br>Solicited Event<br>95% CI | Difference in Proportion of Subjects<br>Experiencing Solicited Event between<br>5% Monolaurin Vaginal Gel and<br>Placebo Gel<br>% | Difference in Proportion of Subjects<br>Experiencing Solicited Event between<br>5% Monolaurin Vaginal Gel and<br>Placebo Gel<br>95% CI | P-Value |
|---|---|---|---|---|---|---|
| Any Solicited | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Adverse event | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vaginal Odor | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| v agiliai Odoi | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vaginal Pain | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| v agillai i alli | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vaginal | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Tenderness | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vulvar/Vaginal | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Itching | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |

Table 63 Comparison of the Proportion of Subjects Experiencing Treatment Emergent Solicited Urogenital Adverse Events through the Test of Cure Visit, Visit 2 by Treatment Group- Safety Population (continued)

| Solicited<br>Urogenital<br>Adverse Event | Treatment<br>Group | Proportion of<br>Subjects<br>Experiencing<br>Solicited Event | Proportion of<br>Subjects<br>Experiencing<br>Solicited Event<br>95% CI | Difference in Proportion of Subjects<br>Experiencing Solicited Event between<br>5% Monolaurin Vaginal Gel and<br>Placebo Gel<br>% | Difference in Proportion of Subjects<br>Experiencing Solicited Event between<br>5% Monolaurin Vaginal Gel and<br>Placebo Gel<br>95% CI | P-Value |
|---|---|---|---|---|---|---|
| Vaginal Dryness | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| v aginai Di yness | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vaginal | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Discharge | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |
| Vulvar | 5%<br>Monolaurin<br>Vaginal Gel | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Inflammation | Placebo Gel | 0.xx | 0.xx, 0.xx | | | |
| | All Subjects | 0.xx | 0.xx, 0.xx | | | |

Table 64: Number and Percentage of Subjects Experiencing Treatment Emergent Solicited Urogenital Adverse Events by Symptom, Maximum Severity, and Treatment Group - Safety Population

| Solicited Urogenital<br>Adverse Event | Severity | 5% | Monolaurin V<br>(N=X) | | | Placebo (N=X) | | | All Subj<br>(N=X | |
|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event | | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| | None | х | Х | x,x | X | х | x,x | х | X | x,x |
| | Mild | Х | X | x,x | X | Х | x,x | X | X | x,x |
| Any Solicited Urogenital | Moderate | X | X | x,x | X | Х | x,x | X | X | x,x |
| Adverse Event | Severe | X | X | x,x | X | Х | x,x | X | X | x,x |
| | Not Reported | X | X | x,x | X | х | x,x | x | X | x,x |
| | Total | X | X | x,x | X | Х | x,x | X | X | x,x |
| | None | X | X | x,x | X | X | x,x | X | X | x,x |
| | Mild | X | X | x,x | X | Х | x,x | X | X | x,x |
| Vaginal Odor | Moderate | X | X | x,x | X | Х | x,x | X | X | x,x |
| Vaginai Odoi | Severe | X | X | x,x | x | X | x,x | X | X | x,x |
| | Not Reported | X | X | x,x | X | X | x,x | X | X | x,x |
| | Total | X | X | x,x | x | X | x,x | X | X | x,x |
| | None | X | X | x,x | x | X | x,x | X | X | x,x |
| | Mild | X | X | x,x | X | X | x,x | X | X | x,x |
| Vaginal Pain | Moderate | X | X | x,x | X | X | x,x | X | X | x,x |
| v agillai Falli | Severe | X | X | x,x | X | X | x,x | X | X | x,x |
| | Not Reported | X | X | x,x | X | x | x,x | X | X | x,x |
| | Total | X | X | x,x | X | X | x,x | X | X | x,x |
| | None | X | X | x,x | X | X | x,x | X | X | x,x |
| | Mild | X | X | x,x | X | Х | x,x | х | X | x,x |
| Vacinal Tandarnass | Moderate | Х | Х | x,x | X | х | x,x | х | X | x,x |
| Vaginal Tenderness | Severe | X | Х | x,x | X | Х | x,x | х | X | x,x |
| | Not Reported | X | X | x,x | X | Х | x,x | X | X | x,x |
| | Total | x | X | x,x | X | x | x,x | X | X | x,x |

Table 64 Number and Percentage of Subjects Experiencing Treatment Emergent Solicited Urogenital Adverse Events by Symptom,
Maximum Severity, and Treatment Group- Safety Population (continued)

| Solicited Urogenital<br>Adverse Event | Severity | 5% | Monolaurin (N=X) | | | Placebo (N=X) | | | All Subj<br>(N=X | |
|---|---|---|---|---|---|---|---|---|---|---|
| Auverse Event | | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| | None | X | X | x,x | X | x | x,x | х | x | x,x |
| | Mild | X | X | x,x | x | х | x,x | X | х | x,x |
| Valuen/Vasinal Habina | Moderate | x | X | x,x | X | x | x,x | Х | x | x,x |
| Vulvar/Vaginal Itching | Severe | x | X | x,x | x | x | x,x | х | x | x,x |
| | Not Reported | X | X | x,x | X | X | x,x | X | X | x,x |
| | Total | x | X | x,x | X | x | x,x | Х | x | x,x |
| | None | x | X | x,x | X | x | x,x | Х | x | x,x |
| | Mild | X | X | x,x | X | X | x,x | Х | X | x,x |
| Vaginal Dryness | Moderate | x | X | x,x | x | x | x,x | х | х | x,x |
| | Not Reported | x | X | x,x | X | x | x,x | Х | x | x,x |
| | Total | x | X | x,x | X | x | x,x | Х | x | x,x |
| | None | x | X | x,x | x | x | x,x | х | x | x,x |
| | Mild | X | X | x,x | X | X | x,x | Х | х | x,x |
| Vaginal Discharge | Moderate | x | X | x,x | X | x | x,x | Х | x | x,x |
| | Not Reported | x | X | x,x | X | x | x,x | Х | x | x,x |
| | Total | x | X | x,x | x | x | x,x | х | x | x,x |
| | None | x | X | x,x | x | x | x,x | х | х | x,x |
| | Mild | х | X | x,x | х | х | x,x | х | х | x,x |
| X 1 | Moderate | х | X | x,x | х | х | x,x | х | х | x,x |
| Vulvar Inflammation | Severe | х | X | x,x | X | X | x,x | х | х | x,x |
| | Not Reported | х | X | x,x | х | х | x,x | х | х | x,x |
| | Total | х | X | x,x | x | х | x,x | х | х | x,x |

Notes: Denominator for percentages is the number of subjects in the Safety Population (N) with treatment emergent solicited urogenital adverse event data available for the specific solicited urogenital adverse event for each treatment group.

<sup>1</sup>Each subject's maximum severity is reported for each treatment emergent solicited urogenital adverse event across all doses. Table includes solicited urogenital adverse events reported from the first dose of study product through Visit 2.

Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Maximum Severity, and **Table 65: Treatment Group - Safety Population** 

| Solicited Symptom | Severity | 5% | Monolaurin V<br>(N=X) | | | Placebo (N=X) | | | All Subj<br>(N=X | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| | None | X | X | x,x | X | х | x,x | х | X | x,x |
| | Mild | X | X | x,x | x | X | x,x | X | X | x,x |
| Am. Caliaita d Commtan | Moderate | X | X | x,x | X | х | x,x | x | X | x,x |
| Any Solicited Symptom | Severe | X | X | x,x | x | х | x,x | x | X | x,x |
| | Not Reported | X | X | x,x | X | X | x,x | х | X | x,x |
| | Total | X | X | x,x | x | х | x,x | x | X | x,x |
| | None | X | X | x,x | X | х | x,x | х | X | x,x |
| | Mild | X | X | x,x | X | X | x,x | х | X | x,x |
| Vocinal Odon | Moderate | X | X | x,x | X | х | x,x | х | X | x,x |
| Vaginal Odor | Severe | X | X | x,x | X | х | x,x | х | X | x,x |
| | Not Reported | X | X | x,x | X | х | x,x | х | X | x,x |
| | Total | X | X | x,x | X | х | x,x | x | X | x,x |
| | None | X | X | x,x | X | х | x,x | x | X | x,x |
| | Mild | X | X | x,x | x | х | x,x | x | X | x,x |
| Vaginal Pain | Moderate | X | X | x,x | X | х | x,x | х | X | x,x |
| vaginai Pain | Severe | X | X | x,x | X | х | x,x | X | X | x,x |
| | Not Reported | X | X | x,x | x | X | x,x | X | X | x,x |
| | Total | X | X | x,x | x | X | x,x | X | X | x,x |
| | None | X | X | x,x | X | х | x,x | х | X | x,x |
| | Mild | X | X | x,x | X | х | x,x | х | X | x,x |
| Vacinal Tandarnasa | Moderate | X | Х | x,x | X | х | x,x | х | X | x,x |
| Vaginal Tenderness | Severe | х | Х | x,x | X | х | x,x | х | X | x,x |
| | Not Reported | X | X | x,x | X | х | x,x | х | х | x,x |
| | Total | X | X | x,x | X | Х | x,x | Х | Х | x,x |

Table 65 Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Maximum Severity, and Treatment Group-Safety Population (continued)

| Solicited Symptom | Severity | 5% | Monolaurin \( (N=X) | | | Placebo (N=X) | | All Subjects (N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| | None | X | X | x,x | X | х | x,x | х | X | x,x |
| | Mild | X | X | x,x | X | х | x,x | х | X | x,x |
| Violence/Violence I Hobins | Moderate | X | X | x,x | X | x | x,x | x | X | x,x |
| Vulvar/Vaginal Itching | Severe | X | X | x,x | X | x | x,x | x | X | x,x |
| | Not Reported | X | X | x,x | X | X | x,x | X | X | x,x |
| | Total | X | X | x,x | X | x | x,x | x | X | x,x |
| | None | X | X | x,x | X | x | x,x | x | X | x,x |
| | Mild | X | X | x,x | X | x | x,x | x | X | x,x |
| Vaginal Dryness | Moderate | X | X | x,x | X | X | x,x | х | X | x,x |
| | Not Reported | X | X | x,x | X | x | x,x | x | X | x,x |
| | Total | X | X | x,x | X | x | x,x | x | X | x,x |
| | None | X | X | x,x | X | x | x,x | X | X | x,x |
| | Mild | X | X | x,x | X | X | x,x | X | X | x,x |
| Vaginal Discharge | Moderate | X | X | x,x | X | x | x,x | x | X | x,x |
| | Not Reported | X | X | x,x | X | x | x,x | x | X | x,x |
| | Total | X | X | x,x | X | X | x,x | х | X | x,x |
| | None | X | X | x,x | X | X | x,x | х | X | x,x |
| | Mild | X | X | x,x | Х | X | x,x | х | X | x,x |
| X 1 Tr Q time | Moderate | х | х | x,x | х | х | x,x | х | х | x,x |
| Vulvar Inflammation | Severe | х | X | x,x | Х | х | x,x | х | х | x,x |
| | Not Reported | x | X | x,x | Х | х | x,x | х | х | x,x |
| | Total | X | X | x,x | Х | х | x,x | Х | X | x,x |

Notes: Denominator for percentages is the number of subjects in the Safety Population (N) with solicited symptom data available for the specific symptom for each treatment group. Each subject's maximum severity is reported for each solicited symptom across all doses. Table includes solicited symptoms reported from the first dose of study product through Visit 2.

Table 66: Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Severity, Study Day, and Treatment Group - All Treatment Groups - Safety Population

| | | | Dose=X) | | ny 1<br>=X) | | ny 2<br>=X) | | y 3<br>=X) | | y 4<br>=X) | Da<br>(N: | ny 5<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Solicited Symptom | Severity <sup>1</sup> | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Solicited Symptom | None | X | x | X | x | X | x | x | X | X | x | X | X |
| | Mild | X | X | X | X | X | X | x | X | X | X | X | X |
| | Moderate | X | X | X | X | X | X | x | X | X | X | X | X |
| | Severe | X | X | X | X | X | X | x | X | X | X | X | X |
| | Not Reported | x | X | X | x | X | x | x | x | х | x | x | X |
| | Total | X | x | X | x | X | x | x | X | X | x | X | X |
| Vaginal Odor | None | x | X | X | x | X | x | x | x | х | x | x | X |
| | Mild | x | x | X | x | X | x | x | x | X | x | x | X |
| | Moderate | X | x | X | x | X | x | x | X | х | x | X | X |
| | Severe | x | x | X | x | X | x | x | x | X | x | x | X |
| | Not Reported | x | x | X | x | X | x | x | x | X | x | x | X |
| | Total | X | x | X | x | X | x | x | X | х | x | X | X |
| Vaginal Pain | None | x | x | X | x | X | x | x | x | X | x | x | X |
| | Mild | x | х | X | X | X | X | X | х | х | x | X | X |
| | Moderate | X | x | X | x | X | x | x | X | х | x | X | X |
| | Severe | x | x | X | x | X | x | x | x | X | x | x | X |
| | Not Reported | x | X | X | x | X | x | x | x | х | x | x | X |
| | Total | x | x | X | x | X | x | x | x | X | x | х | X |
| Vaginal Tenderness | None | х | х | х | х | Х | х | х | х | х | х | Х | х |
| | Mild | X | x | X | x | X | x | x | X | х | x | X | X |
| | Moderate | х | х | X | х | Х | х | х | х | х | х | х | х |
| | Severe | х | х | X | х | Х | х | х | х | х | х | х | х |
| | Not Reported | х | х | X | х | Х | х | х | х | х | х | х | х |
| | Total | х | Х | X | Х | X | Х | х | х | Х | X | х | х |

Table 66 Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Severity, Study Day, and Treatment Group-All Treatment Groups - Safety Population (continued)

| | | | Dose<br>=X) | | ny 1<br>=X) | | ny 2<br>=X) | | y 3<br>=X) | | y 4<br>=X) | | ay 5<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Solicited Symptom | Severity <sup>1</sup> | n | % | n | % | n | % | n | % | n | % | n | % |
| Vulvar/Vaginal Itching | None | X | x | X | x | X | X | x | X | х | x | X | X |
| | Mild | x | x | X | x | X | X | x | X | X | x | х | X |
| | Moderate | X | x | X | x | X | X | x | X | X | x | X | X |
| | Severe | X | x | X | x | X | X | x | X | X | x | X | X |
| | Not Reported | X | x | X | x | X | X | x | X | x | x | X | X |
| | Total | X | x | X | x | X | X | x | X | X | x | X | X |
| Vaginal Dryness | None | x | x | X | x | X | X | x | x | x | x | x | X |
| | Mild | X | X | X | X | X | X | X | X | X | x | X | X |
| | Moderate | x | x | X | x | X | X | x | x | x | x | x | X |
| | Not Reported | X | x | X | x | X | X | x | X | x | x | X | X |
| | Total | X | x | X | x | X | X | x | X | X | x | X | X |
| Vaginal Discharge | None | x | x | X | x | X | X | x | x | x | x | x | X |
| | Mild | X | x | X | X | X | X | x | X | X | x | X | X |
| | Moderate | x | x | X | x | X | X | x | x | x | x | x | X |
| | Not Reported | X | x | X | x | X | X | x | X | x | x | X | X |
| | Total | x | x | X | x | X | X | x | x | x | x | x | X |
| Vulvar Inflammation | None | X | x | X | x | X | X | x | X | х | x | X | X |
| | Mild | X | x | X | x | X | X | x | X | x | x | X | X |
| | Moderate | X | x | X | X | X | X | x | X | X | X | X | X |
| | Severe | X | Х | X | х | X | х | Х | Х | х | X | Х | X |
| | Not Reported | X | Х | X | x | Х | Х | Х | Х | х | X | Х | X |
| | Total | x | x | X | X | x | x | x | x | x | x | x | X |

Notes: Denominator for percentages is the number of subjects in the Safety Population (N) with solicited event data available reporting a solicited adverse event at the day being summarized for each treatment group.

<sup>1</sup>The maximum severity of any solicited adverse event is summarized. A subject is only counted once at the maximum severity.

## Tables with similar format:

- Table 67: Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Severity, Study Day, and Treatment Group-5% Monolaurin Vaginal Gel Safety Population
- Table 68: Number and Percentage of Subjects Experiencing Solicited Symptoms by Symptom, Severity, Study Day, and Treatment Group-Placebo Gel Safety Population

Table 69: Proportion of Subjects Reporting Non-Solicited Non-Laboratory Adverse Events Following the First Dose of Study Product through Visit 3 by Treatment Group - Safety Population

| Treatment Group | Number of<br>Subjects<br>with AEs<br>n | Number of<br>Subjects<br>N | Proportion<br>of Subjects<br>with AEs | Proportion of<br>Subjects with<br>AEs<br>95% CI | Difference in Proportion of<br>Subjects with AEs between<br>5% Monolaurin Vaginal Gel<br>and Placebo Gel | Difference in Proportion of Subjects<br>with AEs between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|
| 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |

Table 70: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Events with 95% Confidence Intervals by MedDRA System Organ Class, and Preferred Term, and Treatment Group - Safety Population

| | | 5% Mono | laurin V<br>(N=X) | Vaginal Gel | | Placeb<br>(N= | | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | MedDRA Preferred Term | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any SOC | Any PT | х | х | x, x | х | х | X, X | Х | х | X, X |
| [SOC 1] | Any PT | х | х | x, x | Х | Х | x, x | Х | X | X, X |
| | [PT 1] | х | х | x, x | Х | Х | x, x | Х | X | X, X |
| | [PT 2] | х | х | x, x | Х | Х | x, x | Х | X | X, X |
| [SOC 2] | Any PT | х | х | x, x | Х | Х | x, x | Х | X | X, X |
| | [PT 1] | х | х | x, x | Х | х | x, x | Х | х | X, X |
| | [PT 2] | х | х | x, x | X | х | X, X | X | х | X, X |

Notes: N = number of subjects in the Safety Analysis Population who received the specified treatment.

This table presents number and percentage of subjects.

A subject is only counted once per PT/timepoint.

Table 71: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - Safety Population

| | | | All Subje | cts (N= | X) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Severity [1] | | | | | | | | Relationship to Treatment [2 | | |
| | | Any In | cidence | M | ild | Mod | erate | Sev | ere | Not Related | | Related | |
| MedDRA System Organ Class | MedDRA Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | Х | Х | X | Х | х | х | х | Х | х | Х | Х | Х |
| [SOC 1] | Any PT | X | X | X | X | х | х | X | X | х | Х | Х | х |
| | [PT 1] | X | X | X | X | Х | Х | X | X | X | X | X | х |
| | [PT 2] | Х | Х | X | Х | х | х | Х | х | х | х | х | Х |
| [SOC 2] | Any PT | Х | Х | X | X | х | х | X | X | х | Х | х | Х |
| | [PT 1] | х | Х | X | х | х | х | X | X | х | Х | х | Х |
| | [PT 2] | Х | Х | X | х | Х | х | Х | х | х | Х | х | х |

Notes: N = Number of subjects in the Safety Analysis Population.

#### Tables with Similar Format:

Table 72: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - 5% Monolaurin Vaginal Gel - Safety Population

Table 73: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group-Placebo Gel - Safety Population

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity,

<sup>[2]</sup> For relationship, a subject is only counted once per preferred term and is summarized according to their closest relationship.

Table 74: Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment Group - Safety Population - All Subjects

| All Subjects (N=X) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Severity [1] | | | | | |
| | | Any In | cidence | M | ild | Moderate | | Severe | |
| MedDRA System Organ Class | MedDRA Preferred Term | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | х | Х | X | X | Х | X | Х | Х |
| [SOC 1] | Any PT | х | X | X | X | X | X | Х | Х |
| | [PT 1] | х | X | X | X | X | X | Х | X |
| | [PT 2] | х | х | Х | X | Х | Х | Х | Х |
| [SOC 2] | Any PT | х | х | X | X | Х | X | Х | X |
| | [PT 1] | х | х | Х | X | Х | Х | Х | Х |
| | [PT 2] | х | х | х | X | X | х | Х | Х |

Notes: N = Number of subjects in the Safety Analysis Population This table presents number and percentage of subjects.

[1] For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

#### Tables with Similar Format:

- Table 75: Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment Group-5% Monolaurin Vaginal Gel Safety Population
- Table 76: Number and Percentage of Subjects Experiencing Related Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, and Treatment Group-Placebo Gel-Safety Population

Table 77: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group - Safety Population - All Subjects

| All Subjects (N=X) | | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Visit 1 (Day 1) – TOC Visit 2<br>(Day 8-15) | | | 2 (Day 8-15) –<br>(Day 22-31) | Any Study Day | |
| MedDRA System Organ Class | MedDRA Preferred Term | n | % | n | % | n | % |
| Any SOC | Any PT | х | Х | Х | Х | Х | X |
| [SOC 1] | Any PT | х | Х | Х | Х | Х | X |
| | [PT 1] | х | Х | х | х | Х | X |
| | [PT 2] | х | X | х | Х | Х | X |
| [SOC 2] | Any PT | х | X | х | Х | Х | X |
| | [PT 1] | х | х | х | х | х | X |
| | [PT 2] | х | X | х | Х | Х | X |

Notes: N = Number of subjects in the Safety Analysis Population

This table presents number and percentage of subjects.

For each time period, a subject is only counted once per PT.

#### Tables with Similar Format:

Table 78: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-5% Monolaurin Vaginal Gel - Safety Population

Table 79: Number and Percentage of Subjects Experiencing Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-Placebo Gel - Safety Population

Table 80: Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group - Safety Population - All Subjects

| All Subjects (N=X) | | | | |
|---|---|---|---|---|
| | | Visit 1 (Day 1) – TOC Visit 2<br>(Day 8-15) | TOC Visit 2 (Day 8-15) –<br>Visit 3 (Day 22-31) | Any Study Day |
| MedDRA System Organ Class | MedDRA Preferred Term | # of Events | # of Events | # of Events |
| Any SOC | Any PT | X | X | X |
| [SOC 1] | Any PT | X | X | X |
| | [PT 1] | X | Х | X |
| | [PT 2] | X | Х | X |
| [SOC 2] | Any PT | X | Х | X |
| | [PT 1] | x | х | X |
| | [PT 2] | X | Х | х |

Notes: N = Number of subjects in the Safety Analysis Population.

This table presents number of events; a subject may be counted multiple times.

#### Tables with Similar Format:

Table 81: Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-5% Monolaurin Vaginal Gel - Safety Population

Table 82: Number of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Preferred Term, Study Day, and Treatment Group-Placebo Gel - Safety Population

Table 83: Number of Non-Solicited Non-Laboratory Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| Preferred Term | Preferred Term MedDRA System Organ Class | 5% Monolaurin Vaginal Gel | Placebo Gel | All Treatment Groups |
|---|---|---|---|---|
| xxxxxx | XXXXXX XXXXXXXX | XX | XX | XX |

Table 84: Subjects Reporting Non-Solicited Non-Laboratory Adverse Events occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| Preferred Term | ferred Term MedDRA System Organ Class Med | | 5% Monolaurin Vaginal Gel | Placebo Gel | All Treatment Groups |
|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | XX.X | XX | XX | XX |

## **Table 85:** Summary of Halting Rules - Safety Population

| Halting Rules | Number of<br>Subjects |
|---|---|
| One or more subjects experiences a treatment-related SAE | x |
| One or more subjects experiences vulvar and/or vaginal ulceration, abscess, or necrosis associated with study product administration | x |
| Two or more subjects experience a treatment-related severe (Grade 3) unsolicited adverse event | X |
| Three or more subjects who received at least one treatment dose experience the same_severe (Grade 3) solicited AE as evaluated by a licensed clinician | х |
| Three or more subjects who received at least one treatment dose experience a severe (Grade 3) study related laboratory abnormality in the same laboratory parameter | х |
| An overall pattern of symptomatic, clinical, or laboratory events that the DMID Medical Monitor or DSMB consider associated with study drug and that may appear minor in terms of individual events, but that may collectively represent a serious potential concern for safety | х |

Table 86: Number and Percentage of Subjects Experiencing Serious Adverse Events Related to Study Product with 95% Confidence Intervals by Treatment Group - Safety Population

| Treatment Group | Number of<br>Subjects with<br>Related SAEs<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Related<br>SAEs | Related<br>SAE<br>95% CI | Difference in Proportion of<br>Subjects with Related SAEs<br>between 5% Monolaurin<br>Vaginal Gel and Placebo Gel | Difference in Proportion of Subjects with<br>Related SAEs between 5% Monolaurin<br>Vaginal Gel and Placebo Gel<br>95% CI | P-Value |
|---|---|---|---|---|---|---|---|
| 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Placebo Gel | x | X | 0.xx | 0.xx, 0.xx | | | |
| All Subjects | x | X | 0.xx | 0.xx, 0.xx | | | |

**Table 87:** Listing of Serious Adverse Events - Safety Population

| Adverse<br>Event | Study Day the<br>Event Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship to<br>Study<br>Treatment | In Not Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject ID: , Treatment Group: , AE Number: | | | | | | | | | |
| xxxxxxx | xx | xxxxxx | xxxxxx | XXXXXX | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments | Comments: xxxxxxxxxxxx | | | | | | | | | |
| Subject ID | : , Treatment Gr | oup: , AE Nui | nber: | | | | | | | |
| xxxxxxx | xx | xxxxxx | xxxxxx | XXXXXX | XXXXX | XXXXXX | Y/N | xxxxx | xxxxx | xxxxx |
| Comments | Comments: xxxxxxxxxxx | | | | | | | | | |

Table 88: Listing of Non-Serious, Non-Solicited, Non-Laboratory, Moderate or Severe Adverse Events - Safety Population

| Adverse<br>Event | Study<br>Day | Severity | Relationship to<br>Study Treatment | In Not Related,<br>Alternative<br>Etiology | Action Taken with<br>Study Treatment | Subject<br>Discontinued Due<br>to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID:, | Treatment | Group: , Al | E Number: | | | | | | |
| xxxxxxx | XX | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | XXXXX | xxxxx |
| Comments:x | XXXXXXXX | XX | | | | | | | |
| Subject ID:, | Subject ID: , Treatment Group: , AE Number: | | | | | | | | |
| xxxxxxx | XX | xxxxxx | xxxxxx | XXXXX | xxxxxx | Y/N | xxxxx | XXXXX | XXXXX |
| Comments:x | Comments:xxxxxxxxxx | | | | | | | | |

# Section 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, placeholder for the CSR)

Table 89: Proportion of Subjects Reporting Laboratory Adverse Events Following the First Dose of Study Product through the Test of Cure Visit, Visit 2 by Treatment Group - Safety Population

| Treatment Group | Number of<br>Subjects with<br>Laboratory AEs<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with<br>Laboratory AEs | Proportion of<br>Subjects with<br>Laboratory AEs<br>95% CI | Difference in Proportion of<br>Subjects with Laboratory<br>AEs between 5% Monolaurin<br>Vaginal Gel and Placebo Gel | Difference in Proportion of Subjects<br>with Laboratory AEs between 5%<br>Monolaurin Vaginal Gel and<br>Placebo Gel<br>95% CI |
|---|---|---|---|---|---|---|
| 5% Monolaurin Vaginal Gel | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx |
| Placebo Gel | X | X | 0.xx | 0.xx, 0.xx | | |
| All Subjects | X | X | 0.xx | 0.xx, 0.xx | | |
Table 90: Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group - Hematology - Safety Population

| | | 5 | 5% Monolaurin Vaginal Gel<br>(N=X) | | | | el | | | Placel<br>(N= | bo Gel<br>=X) | | | | | | bjects<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>y 1<br>=X) | Da | sit 2<br>y 8<br>=X) | Visi<br>Day<br>(N= | <b>28</b> | Da | sit 1<br>y 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Day | it 3*<br>y 28<br>=X) |
| Laboratory Parameter | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | None | Х | х | х | х | х | х | X | х | х | х | х | х | х | х | Х | х | х | х |
| | Any | X | X | X | X | х | X | X | X | X | X | X | X | X | X | X | х | x | X |
| Hemoglobin | Mild | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | Moderate | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | x | X |
| | Severe | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | None | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | Any | Х | х | X | х | х | х | X | Х | X | х | X | X | X | X | х | х | х | х |
| Neutrophils | Mild | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | Moderate | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | X |
| | Severe | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | X |
| | None | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | X |
| | Any | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | x | X |
| Platelets | Mild | Х | х | х | х | х | х | X | х | х | х | х | х | х | х | Х | х | х | х |
| | Moderate | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | x |
| | Severe | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | X |
| | None | X | х | X | Х | Х | х | X | Х | X | X | X | X | X | X | Х | X | х | х |
| | Any | X | х | X | Х | Х | х | X | Х | X | X | X | X | X | X | Х | X | х | х |
| White Blood Cell Count,<br>Decreased | Mild | Х | х | X | х | Х | х | X | Х | X | Х | Х | X | X | х | Х | х | х | х |
| | Moderate | Х | х | X | х | Х | х | X | Х | X | X | х | X | X | X | Х | х | х | х |
| | Severe | Х | х | X | х | х | х | X | Х | X | х | X | X | X | X | х | х | х | х |

Table 90 Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group- Hematology - Safety Population (continued)

| | | 5 | 5% Monolaurin Vaginal Gel<br>(N=X) | | | | | | | | bo Gel<br>=X) | | | | | | bjects<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Da | Day 1 Day 8 1 (N=X) | | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>sy 1<br>=X) | Da | sit 2<br>y 8<br>=X) | Day | it 3* y 28 =X) | |
| Laboratory Parameter | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | None | х | х | X | х | х | х | x | х | х | х | х | х | х | х | x | х | X | х |
| | Any | Х | X | X | х | х | X | x | Х | х | х | х | х | х | х | X | х | X | х |
| White Blood Cell Count,<br>Increased | Mild | х | X | X | х | х | X | X | х | х | х | х | х | х | X | X | X | X | х |
| | Moderate | х | X | X | х | х | X | X | х | х | х | х | х | х | X | X | X | X | х |
| | Severe | х | X | X | х | х | X | X | х | х | х | х | х | х | X | X | X | X | х |
| | None | х | X | X | х | х | X | X | х | х | х | х | х | х | X | X | X | X | х |
| | Any | X | X | X | х | х | X | X | X | х | х | х | х | х | X | X | X | X | х |
| Max of Hematology Parameters | Mild | х | х | X | х | х | x | х | х | х | х | Х | х | х | х | X | x | x | х |
| | Moderate | х | х | X | х | х | x | х | х | х | х | х | х | х | х | Х | x | X | х |
| | Severe | х | X | X | х | х | X | X | х | х | х | х | х | х | х | X | X | Vising Day (No. 2) No. 2 | X |

Notes: N=number of subjects in the Safety Population reporting at least one laboratory measurement at the visit. Denominator for percentages is the number of subjects with the specific laboratory value at the visit.

#### Tables with Similar Format:

Table 91: Laboratory Results Related to Study Product by Parameter, Maximum Severity, Study Visit, and Treatment Group - Hematology - Safety Population

<sup>\*</sup>Laboratory abnormalities that were stable at Visit 2 will not be repeated at Visit 3. Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 will be repeated at Visit 3.

A laboratory abnormality is considered an adverse event if there is a worsening of the laboratory value from the baseline value and it meets the laboratory toxicity grading.

Table 92: Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group – Biochemistry - Safety Population

| | | 5 | 5% Mo | | in Vag<br>=X) | ginal G | el | | | | bo Gel<br>=X) | | | | | | erapies<br>=X) | } | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Day | it 3*<br>y 28<br>=X) |
| Laboratory Parameter | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | None | х | X | X | X | х | х | х | х | X | х | Х | х | х | х | X | X | х | х |
| | Any | х | х | х | х | х | х | х | х | х | х | Х | х | х | х | х | х | х | х |
| Alanine Aminotransferase | Mild | X | X | X | X | X | х | x | х | X | х | X | X | X | X | X | X | X | X |
| | Moderate | X | X | X | X | X | х | x | х | X | х | X | X | X | X | X | X | X | X |
| | Severe | Х | X | X | X | х | х | X | х | х | х | х | х | х | х | х | X | Х | х |
| | None | Х | X | X | X | х | х | X | х | х | х | х | х | х | х | х | X | Х | х |
| | Any | х | X | X | X | X | х | X | X | X | х | х | х | X | х | X | X | X | x |
| Aspartate Aminotransferase | Mild | х | X | X | X | X | х | X | X | X | х | х | х | X | х | X | X | X | x |
| | Moderate | Х | X | X | X | х | х | х | х | х | х | х | х | х | х | х | X | Х | х |
| | Severe | Х | X | X | X | х | х | х | х | х | х | х | х | х | х | х | X | Х | х |
| | None | х | x | x | X | X | х | X | х | x | х | X | х | x | х | x | x | X | х |
| | Any | х | X | х | X | X | х | x | х | х | х | х | х | х | х | х | X | х | х |
| Bilirubin | Mild | х | X | X | X | х | х | х | х | X | х | Х | х | х | х | X | X | х | х |
| | Moderate | х | x | x | X | X | х | X | х | x | х | X | х | x | х | x | x | X | х |
| | Severe | х | X | X | X | X | х | X | X | X | х | х | х | X | х | X | X | X | x |
| | None | х | X | X | X | X | х | X | х | X | х | Х | х | X | Х | X | х | х | х |
| | Any | х | X | X | X | X | х | X | х | X | х | Х | х | X | Х | X | х | х | х |
| Creatinine | Mild | X | X | X | х | X | х | X | х | X | х | Х | X | X | х | X | X | х | X |
| | Moderate | X | X | X | X | X | х | х | х | х | х | х | х | Х | х | х | X | х | х |
| | Severe | х | X | X | X | X | х | X | X | х | х | х | х | X | х | X | X | X | x |

Table 92 Laboratory Results by Parameter, Maximum Severity, Study Visit, and Treatment Group- Biochemistry - Safety Population (continued)

| | | 5 | 5% Mo | | rin Vag<br>=X) | ginal G | el | | | | bo Gel<br>=X) | | | | | | erapie:<br>=X) | S | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Da | sit 1<br>ny 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | sit 1<br>sy 1<br>=X) | Da | sit 2<br>y 8<br>=X) | Da | it 3*<br>y 28<br>=X) | Da | it 1<br>y 1<br>=X) | Da | sit 2<br>ny 8<br>=X) | Da | it 3*<br>y 28<br>=X) |
| Laboratory Parameter | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | None | X | х | Х | х | X | х | х | х | х | х | х | х | x | x | X | X | х | х |
| | Any | X | х | X | х | х | х | х | X | х | х | х | х | X | x | X | X | х | х |
| Glucose, Hypoglycemia | Mild | X | х | X | х | х | х | х | X | х | х | х | х | X | x | X | X | х | х |
| | Moderate | х | х | X | х | х | х | х | х | х | х | х | х | х | х | x | x | х | Х |
| | Severe | х | х | X | х | x | х | х | х | х | х | х | х | х | х | x | x | х | Х |
| | None | х | х | X | х | x | х | х | х | х | х | х | х | х | х | x | x | х | Х |
| | Any | X | х | X | Х | X | х | х | X | х | х | х | х | X | x | X | X | х | х |
| Glucose, Hyperglycemia | Mild | X | х | X | Х | X | X | х | х | х | х | x | x | х | х | X | X | х | х |
| | Moderate | х | х | X | х | x | х | х | х | х | х | х | х | х | х | x | x | х | Х |
| | Severe | X | х | X | Х | X | X | х | х | х | х | x | X | х | х | х | X | х | х |
| | None | X | х | X | Х | X | X | х | х | х | х | x | X | х | х | х | X | х | х |
| | Any | Х | х | х | х | x | х | х | х | х | х | х | x | х | х | х | x | х | х |
| Max of Biochemistry<br>Parameters | Mild | Х | х | х | х | x | х | х | х | х | х | х | x | х | х | х | x | х | х |
| T didilionis | Moderate | X | х | X | х | x | x | x | х | х | х | x | x | х | Х | x | x | x | X |
| | Severe | X | х | Х | х | х | х | х | х | х | х | х | X | х | X | х | X | х | х |

Notes: N=number of subjects reporting at least one laboratory measurement at the visit.

A laboratory abnormality is considered an adverse event if there is a worsening of the laboratory value from the baseline value and it meets the laboratory toxicity grading.

Denominator for percentages is the number of subjects with the specific laboratory value at the visit.

<sup>\*</sup>Laboratory abnormalities that were stable at Visit 2 will not be repeated at Visit 3. Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 will be repeated at Visit 3.

Tables with Similar Format:

Table 93: Laboratory Results Related to Study Product by Parameter, Maximum Severity, Study Visit, and Treatment Group - Biochemistry - Safety Population

Table 94: Laboratory Summary Statistics by Parameter, Study Visit, and Treatment Group - Safety Population

| | | 5% Mo | nolaurin Vaş<br>(N=X) | ginal Gel | | Placebo Gel<br>(N=X) | | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter (unit) | Statistic | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹<br>Day 28<br>(N=X) |
| | n | х | X | X | X | X | X | X | X | х |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| II | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Hemoglobin (g/dL) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | х | x | X | X | x | X | x | x | x |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| N 1.1 (109/L) | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Neutrophils (10 <sup>9</sup> /L) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | x | X | x | X | X | x | x | X | x |
| | Mean | x.x | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| DI ( 1 ( (10 <sup>9</sup> /L) | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| Platelets (10 <sup>9</sup> /L) | Median | x.x | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | x.x |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | x | x | x | X | x | X | x | x | x |
| WI: DI 10 II (1007) | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| White Blood Cells (10 <sup>9</sup> /L) | Standard Deviation | x.x | X.X | x.x | X.X | X.X | X.X | X.X | X.X | x.x |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |

Table 94 Laboratory Summary Statistics by Parameter, Study Visit, and Treatment Group - Safety Population (continued)

| | | 5% Mo | nolaurin Vag<br>(N=X) | ginal Gel | | Placebo Gel<br>(N=X) | | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter (unit) | Statistic | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3 <sup>1</sup> Day 28 (N=X) |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | х | X | X | X | х | x | X | x | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Alanine Aminotransferase | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| (U/L) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | х | X | X | X | х | X | X | x | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Aspartate | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Aminotransferase (U/L) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | х | X | X | X | x | x | x | х | Х |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Dilimakin (m. c/JI.) | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Bilirubin (mg/dL) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | x.x |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | x.x |
| | n | х | X | x | X | х | X | x | х | х |
| Creatinine (mg/dL) | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | x.x |

Table 94 Laboratory Summary Statistics by Parameter, Study Visit, and Treatment Group - Safety Population (continued)

| | | 5% Mo | nolaurin Vag<br>(N=X) | ginal Gel | | Placebo Gel<br>(N=X) | | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter (unit) | Statistic | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹ Day 28 (N=X) | Visit 1<br>Day 1<br>(N=X) | Visit 2<br>Day 8<br>(N=X) | Visit 3¹<br>Day 28<br>(N=X) |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | n | х | X | X | X | X | X | X | X | Х |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Chasse (mg/dL) | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Glucose (mg/dL) | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Mean Change from Visit 1 | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |
| | Standard Deviation | - | X.X | X.X | - | X.X | X.X | - | X.X | X.X |

Notes: N = number of subjects in the Safety Population completing each visit;

n = number of subjects with a laboratory test at the visit specified.

<sup>&</sup>lt;sup>1</sup>Laboratory abnormalities that were stable at Visit 2 will not be repeated at Visit 3. Laboratory abnormalities that occurred between Visit 1 and Visit 2 or worsened at Visit 2 will be repeated at Visit 3. A laboratory abnormality is considered an adverse event if there is a worsening of the laboratory value from the baseline value and it meets the laboratory toxicity grading.

Table 95: Listing of Abnormal Laboratory Results - Hematology - Safety Population

| Subject<br>ID | Treatment<br>Group | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | XX | xx | xx | xxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | Y/N |

Table 96: Listing of Abnormal Laboratory Results - Biochemistry - Safety Population

| Subject<br>ID | Treatment<br>Group | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | XX | xx | xx | xxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | Y/N |

Table 97: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - All Subjects

| All Subjects (N=X) | | | | | | | |
|---|---|---|---|---|---|---|---|
| WHO Drug Code | WHO Drug Code | | ırin Vaginal Gel<br>N=X) | | bo Gel<br>=X) | | ubjects<br>=X) |
| Level 1, Anatomic Group | Level 2, Therapeutic Subgroup | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | x | X | X | X | Х |
| ATC Level 1 - 1] | Any | X | х | X | X | х | Х |
| | [ATC 2 - 1] | X | X | X | X | X | Х |
| | [ATC 2 - 2] | X | X | X | X | X | Х |
| | [ATC 2 - 3] | X | X | X | X | X | Х |
| [ATC Level 1 – 2] | Any | X | x | X | X | х | Х |
| | [ATC 2 - 1] | X | x | X | X | X | Х |
| | [ATC 2 - 2] | X | х | X | X | х | Х |
| | [ATC 2 - 3] | X | х | х | X | х | Х |

Notes: N= Number of subjects in the Safety population

n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

## Tables with Similar Format:

- Table 98: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group-Safety Population-Cincinnati Children's Hospital
- Table 99: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group-Safety Population-University of Iowa
- Table 100: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group-Safety Population-Duke University

| Appendix I | I: Figure Mock-Ups |
|---|---|
| Figure 1: | CONSORT Flow Diagram - All Subjects |
| Figure 2: | Nugent Scores by Visit and Treatment Group - ITT Population 123 |
| Figure 3: | Nugent Scores by Visit and Treatment Group - mITT Population |
| Figure 4: | Nugent Scores by Visit and Treatment Group - Evaluable Population |
| Figure 5: | Nugent Scores by Visit and Treatment Group - PP Population |
| Figure 6: | Maximum Severity of Treatment Emergent Solicited Urogenital Adverse Events by |
| | Treatment Group - Safety Population |
| Figure 7: | Maximum Severity of Solicited Symptoms by Symptom and Treatment Group - Safety |
| Population | 124 |
| Figure 8: | Maximum Severity of Solicited Symptoms by Study Day and Treatment Group - Safety |
| Population | 125 |
| Figure 9: | Frequency of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| Class and Seve | rity - Safety Population 126 |
| Figure 10: | Incidence of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| Class and Seve | rity - Safety Population 127 |
| Figure 11: | Frequency of Non-Solicited Non-Laboratory Adverse Events by Severity - Safety |
| Population | 128 |
| Figure 12: | Incidence of Non-Solicited Non-Laboratory Adverse Events by Severity - Safety Population 129 |
| Figure 13: | Frequency of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| | tionship to Treatment - Safety Population |
| Figure 14: | Incidence of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ |
| Class and Rela | tionship to Treatment - Safety Population |
| Figure 15: | Frequency of Non-Solicited Non-Laboratory Adverse Events by Relationship to Treatment |
| - Safety Popula | tion |
| Figure 16: | Incidence of Non-Solicited Non-Laboratory Adverse Events by Relationship to Treatment |
| - Safety Popula | tion |
| Figure 17: | Laboratory Results by Parameter, Severity, Visit - All Subjects |
| Figure 18: | Laboratory Results by Parameter, Severity, Visit - All Subjects - 5% Monolaurin Vaginal |
| Gel | 134 |
| Figure 19: | Laboratory Results by Parameter, Severity, Visit - All Subjects - Placebo Gel |
| Figure 20: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| Alanine Amino | otransferase (U/L) |
| Figure 21: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| | notransferase (U/L) |
| Figure 22: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| | 136 |
| Figure 23: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| ` • | /dL) |
| Figure 24: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| | L) |
| Figure 25: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| | /dL) |
| Figure 26: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| | 0 <sup>9</sup> /L) |
| Figure 27: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| , | L) |
| Figure 28: | Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - |
| White Blood C | $^{136}$ ells ( $^{10}$ /L) |

Figure 1: CONSORT Flow Diagram - All Subjects





Figure 2: Nugent Scores by Visit and Treatment Group - ITT Population

Figures with similar Format:

Figure 3: Nugent Scores by Visit and Treatment Group - mITT Population

Figure 4: Nugent Scores by Visit and Treatment Group - Evaluable Population

Figure 5: Nugent Scores by Visit and Treatment Group - PP Population

Figure 6: Maximum Severity of Treatment Emergent Solicited Urogenital Adverse Events by Symptom and Treatment Group - Safety Population



Figures with similar format:

Figure 7: Maximum Severity of Solicited Symptoms by Symptom and Treatment Group - Safety Population

#### Implementation Note:

Figures will be paneled in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 8: Maximum Severity of Solicited Symptoms by Study Day and Treatment Group - Safety Population



### Implementation Note:

Figures will be paneled in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 9: Frequency of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Severity - Safety Population



Figure 10: Incidence of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Severity - Safety Population



Figure 11: Frequency of Non-Solicited Non-Laboratory Adverse Events by Severity - Safety Population



### Implementation Note:

Figures will be presented in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 12: Incidence of Non-Solicited Non-Laboratory Adverse Events by Severity - Safety Population



Implementation Note: Figures will be presented in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 13: Frequency of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Relationship to Treatment - Safety Population



Figure 14: Incidence of Non-Solicited Non-Laboratory Adverse Events by MedDRA System Organ Class and Relationship to Treatment - Safety Population



Frequency of Non-Solicited Non-Laboratory Adverse Events by Relationship to Treatment - Safety Population Figure 15:



Implementation Note:

Figures will be presented in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 16: Incidence of Non-Solicited Non-Laboratory Adverse Events by Relationship to Treatment - Safety Population



Implementation Note:

Figures will be presented in the following order: 5% Monolaurin Vaginal Gel, Placebo Gel, All Subjects

Figure 17: Laboratory Results by Parameter, Severity, Visit - All Subjects



Figures with Similar Format:

Figure 18: Laboratory Results by Parameter, Severity, Visit - All Subjects - 5% Monolaurin Vaginal Gel

Figure 19: Laboratory Results by Parameter, Severity, Visit - All Subjects - Placebo Gel

Figure 20: Summary of Mean Change from Baseline Clinical Laboratory Result - Safety Population - Alanine Aminotransferase (U/L)



### Figures with Similar format:

- Figure 21: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Aspartate Aminotransferase (U/L)
- Figure 22: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Bilirubin (mg/dL)
- Figure 23: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Creatinine (mg/dL)
- Figure 24: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Glucose (mg/dL)
- Figure 25: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Hemoglobin (g/dL)
- Figure 26: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Neutrophils (10<sup>9</sup>/L)
- Figure 27: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population Platelets (10<sup>9</sup>/L)
- Figure 28: Summary of Mean Change from Baseline Clinical Laboratory Result Safety Population White Blood Cells (10<sup>9</sup>/L)

| Appendix | III: Listings Mock-Ups | |
|---|---|---|
| Listing 1: | 16.2.1 Early Terminations or Discontinued Subjects – All Enrolled Subjects | 138 |
| Listing 2: | 16.2.2.1 Subject-Specific Protocol Deviations- All Enrolled Subjects | |
| Listing 3: | 16.2.2.2 Non-Subject-Specific Protocol Deviations | |
| Listing 4: | 16.2.3 Subjects Excluded from Analysis Populations | 141 |
| Listing 5: | 16.2.4.1 Demographics Data - All Enrolled Subjects | 142 |
| Listing 6: | 16.2.4.2 Pre-Existing Medical Conditions – All Enrolled Subjects | 143 |
| Listing 7: | 16.2.4.3 Baseline Sexual History – All Enrolled Subjects | |
| Listing 8: | 16.2.4.4 Follow-up Sexual History - Safety Population | 145 |
| Listing 9: | 16.2.5 Compliance Data - Safety Population | 146 |
| Listing 10: | 16.2.6 Individual Efficacy Response Data | 147 |
| Listing 11: | 16.2.7.1 Clinical Assessment - Safety Population | 148 |
| Listing 12: | 16.2.7.2 Solicited Symptoms - Safety Population | |
| Listing 13: | 16.2.7.3 Unsolicited Adverse Event - Safety Population | 150 |
| Listing 14: | 16.2.8.1 Clinical Laboratory Results – Hematology - Safety Population | 151 |
| Listing 15: | 16.2.8.2 Clinical Laboratory Results – Biochemistry - Safety Population | 152 |
| Listing 16: | 16.2.9.1 Physical Exam Findings | 153 |
| Listing 17: | 16.2.9.2 Pelvic Exam Findings | 154 |
| Listing 18: | 16.2.9.3 Additional Gynecological Test Results | 155 |
| Listing 19: | 16.2.10.1 Concomitant Medications - Safety Population | 156 |
| Listing 20: | 16.2.10.2 Subjects Whose Assigned Treatment Group Does Not Match Their Rand | lomized |
| Treatment G | roup | |
| Listing 21: | 16.2.10.3 Subjects Product Administration Position- Safety Population | 158 |
| Listing 22: | 16.2.10.4 Amsel Criteria - mITT population | |
| Listing 23: | 16.2.10.5 Nugent Scores, Bacterial Morphotypes, and Yeast - mITT Population | 160 |
| Listing 24 | 16.2.10.6 Clinical Failures-Safety Population | |
| Listing 25 | 16.2.10.7 BV Infection Status - Safety Population | |
| Listing 26 | 16.2.11.1 Pregnancy Reports – Maternal Information - Safety Population | 163 |
| Listing 27 | 16.2.11.2 Pregnancy Reports – Gravida and Para | |
| Listing 28 | 16.2.11.3 Pregnancy Reports – Live Birth Outcomes | |
| Listing 29 | 16.2.11.4 Pregnancy Reports – Still Birth Outcomes | |
| Listing 30 | 16.2.11.5 Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Ou<br>165 | itcomes |

## **Programming Notes:**

The following notes should be implemented on all listings:

- 1. If the actual treatment is not the same as the randomized treatment, then have a column for Randomized Treatment Group and Actual Treatment Group on all listings. If actual treatment equals randomized treatment, then will have one column labeled "Treatment Group".
- 2. For missing data, '-' will be used in blank cells.

**Listing 1:** 16.2.1 Early Terminations or Discontinued Subjects – All Enrolled Subjects

| Subject<br>ID | Randomized<br>Treatment Group | Actual Treatment<br>Group | Category | Study Day Corresponding to Early Termination/Treatment Discontinuation/Completion | Reason for Early<br>Termination/ Treatment<br>Discontinuation |
|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | Early Termination/Treatment Discontinuation/Completion | XX | xxxxxxxxxxxxx |
| xxxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | Early Termination/Treatment Discontinuation/Completion | XX | |

- 1. Sort order will be by Subject ID, Category
- 2. Category will be "Early Termination", "Completion" or "Treatment Discontinuation". If a subject discontinued treatment, they will have two records.
- 3. In the "Reason" column, concatenate any "specify" fields, including AE number and DV number.

Listing 2: 16.2.2.1 Subject-Specific Protocol Deviations- All Enrolled Subjects

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Deviation<br>Number | Study<br>Day | Deviation<br>Description | Deviation<br>Category | Reason<br>for<br>Deviation | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Xxxxxx | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xx | xx | xxxxxx | xxxxxxxxxx | xxxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | xxxxxxxxxx |
| Xxxxxx | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xx | xx | xxxxxxx | xxxxxxxxx | xxxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |

Note: Deviation description column will contain all subfields concatenated together

- 1. Sort order will be by Subject ID, Deviation Number
- 2. In the Deviation Category column concatenate any specify fields
- 3. In the Reason for Deviation column concatenate any specify fields.

**Listing 3:** 16.2.2.2 Non-Subject-Specific Protocol Deviations

| Site | Deviation | Start Day | End Day | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | XX | XX | XXXX | Yes/No | Yes/No/NA | XXXX | xxxx | XXXX |
| xxxx | xxxx | XX | XX | XXXX | Yes/No | Yes/No/NA | XXXX | XXXX | XXXX |

Note: Deviation column will contain all subfields concatenated together

- 1. Sort order will be by Site Name, Start Date
- 2. In the Deviation Category column concatenate any specify fields
- 3. In the Reason for Deviation column concatenate any specify fields.

Listing 4: 16.2.3 Subjects Excluded from Analysis Populations

| Randomized<br>Treatment Group | Actual<br>Treatment<br>Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason(s) Subject<br>Excluded |
|---|---|---|---|---|---|---|
| 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xxxxxx | [e.g., Safety, ITT, mITT,<br>Evaluable, PP] | [e.g., Safety, ITT, mITT, Evaluable, PP, Visit x] | Yes/No | xxxxx |
| 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xxxxx | [e.g., Safety, ITT, mITT,<br>Evaluable, PP] | [e.g., Safety, ITT, mITT, Evaluable, PP, Visit x] | Yes/No | xxxxx |
| 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xxxxxx | [e.g., Safety, ITT, mITT,<br>Evaluable, PP] | [e.g., Safety, ITT, mITT, Evaluable, PP, Visit x] | Yes/No | xxxxx |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. If "Yes" the population in which data were removed will be listed in parenthesis. "No" indicates that no data were available for inclusion in the analysis.

- 1. Sort order will be randomized treatment group, Subject ID
- 2. Reasons Subject Excluded should match the same verbiage that is used on the Analysis population tables (Tables 3 and 4)
- 3. For subjects excluded from the Per Protocol population, specify which visit's PP population (Visit 2 or Visit 3) the subject is excluded from

**Listing 5:** 16.2.4.1 Demographics Data - All Enrolled Subjects

| Subject ID | Randomized Treatment<br>Group | Actual Treatment Group | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | xx | xxxxxx | xxxxxx |
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | xx | xxxxxx | xxxxxx |
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | XX | xxxxxx | xxxxxx |

- 1. Sort order will be by Subject ID
- 2. For the Race column, if a subject is Multi-Racial, all races will be listed, separated by a comma

# **Listing 6:** 16.2.4.2 Pre-Existing Medical Conditions – All Enrolled Subjects

| Subject<br>ID | Randomized Treatment Group | Actual Treatment Group | MH<br>Number | Medical<br>History Term | Condition<br>Start Day | Condition<br>End Day | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | xxx | xxxxxx | xx | xx | xxxxxx | xxxxxx |
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | xxx | xxxxxx | xx | xx | xxxxxx | xxxxxx |

- 1. Sort order is Subject ID, MH Number.
- 2. "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). Rather than use exact study days, categorize as follows:
- > 5 years prior to enrollment
- 1-5 years prior to enrollment
- -1-12 months prior to enrollment
- -Within 1 month of enrollment
- -During Study
- -If Ongoing at the end of the study, display "Ongoing' in the "Condition End Day" column.
- -If ending is unknown at the end of the study, display "Unknown" in the "Condition End Day" column.

**Listing 7:** 16.2.4.3 Baseline Sexual History – All Enrolled Subjects

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Number of<br>episodes of<br>BV in last<br>12 months | Received<br>treatment for<br>previous episodes<br>of BV in the<br>previous 12<br>months? | Sexually active? | Sexual<br>Orientation | Sex with men or<br>women in the past 12<br>months? | Vaginal<br>intercourse in<br>the past 12<br>months? | Receptive oral<br>intercourse in<br>the past 12<br>months? | Receptive anal intercourse in the past 12 months? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xx | Yes/No | Yes/No/Unknown | Heterosexual/<br>Gay/<br>Homosexual/<br>Bisexual/<br>Unknown | Men/Women/Both/<br>Neither/Unknown | Yes/No/<br>Unknown | Yes/No/<br>Unknown | Yes/No/<br>Unknown |
| xxxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | xx | Yes/No | Yes/No/Unknown | Heterosexual/<br>Gay/<br>Homosexual/<br>Bisexual/<br>Unknown | Men/Women/Both/<br>Neither/Unknown | Yes/No/<br>Unknown | Yes/No/<br>Unknown | Yes/No/<br>Unknown |

- 1. Sort order is Subject ID.
- 2. If answer to Sexually Active is 'No', then the remaining columns ('Sexual Orientation' through 'Receptive anal intercourse in the past 12 months?" should be blank. Fill with a '-'.
**Listing 8:** 16.2.4.4 Follow-up Sexual History - Safety Population

| | | | S | ince First Dose of T | Treatment | | 48 Hours Prior to Vis | it 3 |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Randomized<br>Treatment Group | Actual<br>Treatment<br>Group | Engaged in<br>vaginal<br>intercourse? | Received oral intercourse? | Inserted any intravaginal substances or objects other than the study treatment? | Engaged in<br>vaginal<br>intercourse? | Received oral intercourse? | Inserted any intravaginal substances or objects other than the study treatment? |
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | Yes/No/<br>Unknown<br>[Condom:<br>xxx] | Yes/No/Unknown<br>[Barrier: xxx] | Yes/No/<br>Unknown<br>[Substance(s): xxx] | Yes/No/Unknown<br>[Condom: xxx] | Yes/No/Unknown<br>[Barrier: xxx] | Yes/No/Unknown<br>[Substance(s): xxx] |
| XXXXXX | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | Yes/No/<br>Unknown<br>[Condom:<br>xxx] | Yes/No/Unknown<br>[Barrier: xxx] | Yes/No/<br>Unknown<br>[Substance(s): xxx] | Yes/No/Unknown<br>[Condom: xxx] | Yes/No/Unknown<br>[Barrier: xxx] | Yes/No/Unknown<br>[Substance(s): xxx] |

Note: If Condoms, barriers, or substances were used, they will be listed in the cell

- 1. Sort order is Subject ID.
- 2. If answer to 'Engaged in vaginal intercourse?' is 'Yes', then concatenate answer to whether a condom was used 'Yes/No' (i.e. Yes [Condom: Yes]). If answer is 'No' or 'Unknown', there will be no answer to condom usage.
- 3. If answer to 'Received oral intercourse?' is 'Yes', then concatenate answer to whether a barrier was used 'Yes/No' (i.e. Yes [Barrier: No]). If answer is 'No' or 'Unknown', there will be no answer to barrier usage.
- 4. If answer to 'Inserted any intravaginal substances or objects other than the study treatment?' is 'Yes', then concatenate answer to the substances that were inserted: Tampons, Spermicide, Douche, Diaphragm, Feminine deodorant product, Other: Other, specify. For example, if a subject marked Yes to Tampons, Douche and Other, where other specify is metronidazole gel, this column would be: Yes [Substances: Tampons, Douche, Other: metronidazole gel]. If answer is 'No' or 'Unknown', there will be no answer to substances.

**Listing 9:** 16.2.5 Compliance Data - Safety Population

| | | | | Subject Report | | Clinic Assessment of | Product Accountability |
|---|---|---|---|---|---|---|---|
| Subject ID | Randomized<br>Treatment Group | Actual Treatment<br>Group | Number of Doses<br>Taken as<br>Scheduled | Number of Doses<br>Taken Out of<br>Window | Number of Doses<br>Not Taken | Returned Used<br>Applicators | Returned Unused<br>Applicators |
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | x | x | x | x | x |
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | X | x | x | x | x |
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | x | x | x | x | x |

- 1. Sort order is Subject ID.
- 2. Total number of doses is 6. Number of doses not taken will be calculated as 6 Number of doses taken as scheduled Number of doses taken out of window.
- 3. A dose will be considered 'Taken as Scheduled' on a given day if there are 2 doses taken on the same day at least 8 hours a part. The doses should be taken within 72 hours from first dose at least 8 hours apart and not more than 2 doses in a 24 hour period to be counted as all 6 being 'Taken as Scheduled'. If only one dose is taken on a day, then the first dose will be considered 'Taken as Scheduled'. If the first dose is taken after 3 pm, then only 1 dose will be taken on Day 1 and 1 dose on Day 4. Otherwise, a subject should have 2 doses taken on Day 1, 2 doses taken on Day 2 and 2 doses taken on Day 3. Any doses taken outside these time limits will be considered to be 'Taken Out of Window'.
- 4. If a subject does not have a record for 'Returned Used Applicators' or 'Returned Unused Applicators', then an 'Unknown' will be placed in those columns.

### **Listing 10:** 16.2.6 Individual Efficacy Response Data

| Subject ID | Randomized Treatment Group | Actual Treatment<br>Group | Analysis Population | Visit<br>Number | Study<br>Day | Clinical Cure | Bacteriologic<br>Cure | Therapeutic<br>Cure |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal Gel/Placebo<br>Gel | | ITT, mITT,<br>Evaluable, PP | XX | xx | Y/N | Y/N | Y/N |
| xxxxxx | 5% Monolaurin Vaginal Gel/Placebo<br>Gel | | ITT, mITT,<br>Evaluable, PP | XX | XX | Y/N | Y/N | Y/N |
| xxxxxx | 5% Monolaurin Vaginal Gel/Placebo<br>Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | ITT, mITT,<br>Evaluable, PP | XX | xx | Y/N | Y/N | Y/N |

- 1. Sort order is Subject ID, Analysis Population, Visit Number.
- 2. For Analysis Population, sort in the following order (will have to create a dummy sort variable): ITT, mITT, Evaluable, PP.
- 3. A subject will have one row for each analysis population/visit combination. So if a subject is in all 4 populations, that subject will have 8 rows in this table. One for ITT Visit 2, ITT Visit 3, mITT Visit 3, Evaluable Visit 2, Evaluable Visit 3, PP Visit 3.

**Listing 11: 16.2.7.1 Clinical Assessment - Safety Population** 

| Study Day | Study Day Vaginal Odor | | Vaginal<br>Tenderness | Vulvar/Vaginal<br>Itching | Vaginal Dryness | Vaginal Discharge | Vulvar<br>Inflammation |
|---|---|---|---|---|---|---|---|
| Subject ID: , Randomized Treatment Group: , Actual Treatment Group: | | | | | | | |
| XX | [severity] | [severity] | [severity] | [severity] [severity] | | [severity] | [severity] |
| XX | [severity] | [severity] | [severity] | [severity] [severity] | | [severity] | [severity] |
| XX | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] |

Note: Vaginal Dryness and Vaginal Discharge are graded on a two-point scale (mild, moderate).

- 1. Sort order is Subject ID.
- 2. Data from Visits 1, 2, and 3 will be listed

**Listing 12:** 16.2.7.2 Solicited Symptoms - Safety Population

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Study Day | Vaginal<br>Odor | Vaginal<br>Pain | Vaginal<br>Tenderness | Vulvar/Vaginal<br>Itching | Vaginal<br>Dryness | Vaginal<br>Discharge | Vulvar Inflammation |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | xx | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] |
| xxxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | xx | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] | [severity] |

Note: \* means symptom qualifies as a treatment emergent solicited adverse event.

- 1. Sort order is Subject ID, Study Day.
- 2. If a symptom is ongoing after day 5, add a row for Day 6 and for each day until the end date of the symptom. The severity will be the maximum severity reported for that symptom.
- 3. Mark all severities with an asterisk, \*, that are considered treatment emergent solicited adverse events.

**Listing 13: 16.2.7.3 Unsolicited Adverse Event - Safety Population** 

| Adverse<br>Event | Study<br>Day | Severity | SAE? | Relationship to<br>Study Treatment | In Not Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued Due<br>to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Randomized Treatment Group: , Actual Treatment Group: , AE Number: | | | | | | | | | | |
| XXXXXXX | XX | xxxxxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | XXXXX | XXXXX |
| Comments: | Comments: xxxxxxxxxxx | | | | | | | | | |
| Subject ID | :, Randor | nized Treat | ment Gro | up: , Actual Treatme | ent Group: , AE Num | ber: | | | | |
| xxxxxxx | xx | xxxxxx | xxxxxx | XXXXXX | XXXXX | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments: | XXXXXXXX | xxxxx | | | 1 | ı | ' | 1 | 1 | 1 |

Note: For additional details about SAEs, see Table 79.

- 1. Sort order is Subject ID, AE Number.
- 2. Shaded rows will be in the SAS color LTGRAY light gray #C0C0C0

Listing 14: 16.2.8.1 Clinical Laboratory Results – Hematology - Safety Population

| Subject ID | Randomized Treatment<br>Group | Actual Treatment<br>Group | Age<br>(years) | Study<br>Day | Hemoglobin<br>(g/dL) | Neutrophils<br>(10 <sup>9</sup> /L) | Platelets (10 <sup>9</sup> /L) | White Blood Cell Count (109/L) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | XX | XX | XX.X | XX.XX | XXX | XX.XX |
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | XX | XX | XX.X | XX.XX | XXX | XX.XX |

- 1. Sort order is Subject ID, Study Day.
- 2. Toxicity grades can be found in Appendix B of the Protocol. If a lab has a toxicity Grade of 1, 2, or 3, then put grade in parenthesis after the result. (i.e. 90 (Gr 3). If the toxicity grade is an increase, then add a "+" to the grade (i.e. +Gr 3). If a toxicity grade is a decrease, then add a '-' to the grade (i.e. -Gr 3). Note: all of the above hematology labs have a toxicity grading scale.

**Listing 15:** 16.2.8.2 Clinical Laboratory Results – Biochemistry - Safety Population

| Subject ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Age<br>(years) | Study<br>Day | Alanine<br>Aminotransferase<br>(U/L) | Aspartate<br>Aminotransferase<br>(U/L) | Bilirubin<br>(mg/dL) | Creatinine (mg/dL) | Glucose<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | XX | xx | XXXX | XXXX | X.X | X.XX | XXX |
| xxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | 5% Monolaurin<br>Vaginal<br>Gel/Placebo Gel | XX | xx | XXXX | XXXX | X.X | X.XX | XXX |

- 1. Sort order is Subject ID, Study Day.
- 2. Toxicity grades can be found in Appendix B of the Protocol. If a lab has a toxicity Grade of 1, 2, or 3, then put grade in parenthesis after the result. (i.e. 90 (Gr 3). If the toxicity grade is an increase, then add a "+" to the grade (i.e. +Gr 3). If a toxicity grade is a decrease, then add a '-' to the grade (i.e. -Gr 3). Note: all of the above biochemistry labs have a toxicity grading scale.

# Listing 16: 16.2.9.1 Physical Exam Findings

| Subject ID | Randomized Treatment<br>Group | Actual Treatment Group | | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; AE Number) |
|---|---|---|---|---|---|---|
| xxxxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | XXX | xxxxxxx | xxxxxxx | Yes/No<br>xxxxxx; xx |

- 1. Sort order is Subject ID, Study Day.
- 2. Only abnormal findings will be presented.
- 3. If the physical exam was reported as an AE, then concatenate the Physical exam with the Adverse Events by AENUM and report the AETERM, plus the AE Number.

**Listing 17:** 16.2.9.2 Pelvic Exam Findings

| | | | | | | | Objectiv | Objective Signs of Inflammation | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Cervix | | | Vagina | | | Vulva | | | Vaginal Discharge | | | |
| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Study<br>Day | Edema | Erythema | Excoriation | Edema | Erythema | Excoriation | Edema | Erythema | Excoriation | Quantity | Color | Consistency | Odor |
| xxxxxxxx | 5% Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | XXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | xxxxx | xxxxx | xxxxx | xxxxx |

- 1. Sort order is Subject ID, Study Day.
- 2. If Discharge is not present, populate cells with '-'.

# Listing 18: 16.2.9.3 Additional Gynecological Test Results

| Subject<br>ID | Randomized Treatment<br>Group | <b>Actual Treatment Group</b> | Study<br>Day | Motile flagellated protozoa on saline wet mount? | Rapid Trichomonas<br>test result | Pseudohyphae or budding spores on KOH wet mount? |
|---|---|---|---|---|---|---|
| xxxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | XX | Negative/Positive | Negative/Positive | Negative/Positive |

- 1. Sort order is Subject ID, Study Day.
- 2. 'Rapid Trichomonas test' was only collected on Day 1 and only conducted if the 'Motile flagellated protozoa' test was negative. Put a 'N/A' if test was not collected .

**Listing 19: 16.2.10.1 Concomitant Medications - Safety Population** 

| Subject<br>ID | Randomized<br>Treatment Group | Actual Treatment<br>Group | Concomitant<br>Medication<br>Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Taken for an AE? (AE Description; AE Number) | Taken for a<br>condition on<br>Medical History?<br>(MH Description;<br>MH Number) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | XX | xxxxxx | XX | XX | xxxxxx | Yes/No<br>xxxxx; xx | Yes/No<br>xxxxx; xx |
| xxxxxx | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | 5% Monolaurin<br>Vaginal Gel/Placebo<br>Gel | xx | xxxxxx | XX | xx | xxxxxx | Yes/No<br>xxxxx; xx | Yes/No<br>xxxxx; xx |

- 1. Sort order is Subject ID, concomitant medication number.
- 2. 'Medication Start Day' and 'Medication End Day' are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact days, categorize as follows:
- > 5 years prior to enrollment
- 1- 5 years prior to enrollment
- 1-12 months prior to enrollment.
- For 'Medication End Day', if medication is Ongoing, display 'Ongoing' in the Medication End Day' column.
- For 'Medication End Day', if end of medication is unknown, display 'Unknown' in the 'Medication End Day' column.
- 3. If a Medication is taken for an AE, then concatenate the conmed with the Adverse Events by AENUM and report the AETERM, plus the AE Number.
- 4. If a Medication is taken for an MH, then concatenate the conmed with the Medical History event by MHNUM and report the MHTERM, plus the MH Number.
- 5. Include the birth control information in this dataset. The birth control information is coming from the RP/SUPPRP or BC1 dataset.

# Listing 20: 16.2.10.2 Subjects Whose Assigned Treatment Group Does Not Match Their Randomized Treatment Group

| Subject ID | Treatment Group at Randomization | Treatment Actually Received |
|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal Gel/Placebo Gel | 5% Monolaurin Vaginal Gel/Placebo Gel |
| xxxxxx | 5% Monolaurin Vaginal Gel/Placebo Gel | 5% Monolaurin Vaginal Gel/Placebo Gel |

### Implementation Note:

1. Sort order is Subject ID.

Listing 21: 16.2.10.3 Subjects Product Administration Position- Safety Population

| Subje<br>ct ID | Randomize<br>d<br>Treatment<br>Group | Actual<br>Treatmen<br>t Group | Dose 1 Status | Dose 2 Status | Dose 3 Status | Dose 4 Status | Dose 5 Status | Dose 6 Status | Total Number of Doses Taken in the Recumbe nt Position n (%) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx<br>x | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placeb<br>o Gel | 5%<br>Monolauri<br>n Vaginal<br>Gel/Placeb<br>o Gel | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | xx (xx) |
| XXXXX<br>X | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placeb<br>o Gel | 5%<br>Monolauri<br>n Vaginal<br>Gel/Placeb<br>o Gel | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | Recumbent/Not<br>Recumbent/Missi<br>ng | xx (xx) |

1. Sort order is Subject ID.

Listing 22: 16.2.10.4 Amsel Criteria - mITT population

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Visit | Study<br>Day | Amine ("whiff") test<br>on KOH wet<br>mount | Off-white<br>(milky or gray),<br>thin,<br>homogenous<br>discharge | Percentage of<br>clue cells on<br>saline wet<br>mount | Vaginal<br>pH | Number<br>of Amsel<br>Criteria<br>Met | Clinical Cure<br>Determination |
|---|---|---|---|---|---|---|---|---|---|---|
| | 5% Monolaurin | 5%<br>Monolaurin | 01 | XX | Positive/Negative/Not<br>Assessed | Yes/No/Not<br>Assessed | x/Not<br>Assessed | xx.x/Not<br>Assessed | xx | |
| xxxxxx | Vaginal<br>Gel/Placebo | Vaginal<br>Gel/Placebo<br>Gel | 02 | XX | Positive/Negative/Not<br>Assessed | Yes/No/Not<br>Assessed | x/Not<br>Assessed | xx.x/Not<br>Assessed | xx | Cure/Failure/Not<br>Evaluable |
| | Gel | | 03 | XX | Positive/Negative/Not<br>Assessed | Yes/No/Not<br>Assessed | x/Not<br>Assessed | xx.x/Not<br>Assessed | xx | Cure/Failure/Not<br>Evaluable |

- 1. Sort order is Subject ID, Study Day.
- 2, Unscheduled visits will be included
- 3. Clinical Cure Determination will be based on the mITT population

Listing 23: 16.2.10.5 Nugent Scores, Bacterial Morphotypes, and Yeast - mITT Population

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Visit | Study Day | Lactobacillus<br>Culture<br>Count | Gardnerella<br>Culture<br>Count | Mobiluncus<br>Culture<br>Count | Candida<br>Culture<br>Count | Budding<br>Yeast | Nugent<br>Score | Bacteriological<br>Cure<br>Determination |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5% | 5%<br>Monolaurin<br>Vaginal | 01 | xx | xxxxxxx | xxxxxxx | xxxxxxx | xxxxxxxx | Few/Moderate/<br>Many/No<br>organisms seen | 0-10 | |
| xxxxxx | Monolaurin<br>Vaginal<br>Gel/Placebo | Gel/Placebo<br>Gel | 02 | xx | xxxxxxx | xxxxxxx | xxxxxxx | xxxxxxxx | Few/Moderate/<br>Many/No<br>organisms seen | 0-10 | Cure/Failure |
| | Gel | | 03 | xx | xxxxxxx | xxxxxxx | xxxxxxx | xxxxxxx | Few/Moderate/<br>Many/No<br>organisms seen | 0-10 | Cure/Failure |

- 1. Sort order is Subject ID, Study Day.
- 2, Unscheduled visits will be included
- 3. Bacteriological Cure Determination will be based on the mITT population

Listing 24 16.2.10.6 Clinical Failures-Safety Population

| | | | | | | Re | ason for Clinical Failu | ire | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Visit | Study<br>Day | Lack of resolution<br>of one or more<br>signs or symptoms<br>in the Amsel<br>criteria | Presentation of<br>new signs or<br>symptoms<br>meeting the Amsel<br>criteria | Early discontinuation of study therapy due to lack of treatment effect | Use of any vaginosis<br>therapy or systemic<br>antimicrobial<br>therapy other than<br>study product | Requires<br>additional<br>treatment for<br>vaginosis |
| | 5% Monolaurin | 5%<br>Monolaurin | 02 | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| xxxxxx | Vaginal<br>Gel/Placebo<br>Gel | Vaginal Gel/Placebo Gel | 03 | xx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

- 1. Sort order is Subject ID, Study Day.
- 2. These reasons come from the eCRF and are not calculated (GYN) dataset.

# **Listing 25** 16.2.10.7 BV Infection Status - Safety Population

| Subject ID | Randomized Treatment Group | Actual Treatment Group | BV Infection Subgroup | If Recurrent, Number of Episodes in previous 12 months |
|---|---|---|---|---|
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | First time Infection | NA |
| xxxxxx | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | 5% Monolaurin Vaginal<br>Gel/Placebo Gel | Recurrent Infection | xx |

- 1. Sort order is Subject ID.
- 2. The infection status comes from Question 1 of the Sexual History CRF. If a subject answers 1, then they have 'First time infection'. If they answer 2 or more, then they have Recurrent Infection.

**Listing 26** 16.2.11.1 Pregnancy Reports – Maternal Information - Safety Population

| Subject<br>ID | Randomized<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal Complications During Labor, Delivery, or Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | 5%<br>Monolaurin<br>Vaginal<br>Gel/Placebo<br>Gel | XXX | xxx | xxx | XXX | xxx | xxx | Y/N | Y/N | Y/N | Y Y/N /N |

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Implementation Notes:

1. Sort order is Subject ID, Pregnancy Number

Listing 27 16.2.11.2 Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subje<br>ct ID | Pregnan<br>cy<br>Number | Gravid<br>a | Extreme<br>ly<br>Preterm<br>Births | Very<br>Preter<br>m<br>Births | Early<br>Preter<br>m<br>Births | Late<br>Preter<br>m<br>Births | Earl<br>y<br>Ter<br>m<br>Birth | Full<br>Ter<br>m<br>Birth<br>s | Late<br>Ter<br>m<br>Birth<br>s | Post<br>Ter<br>m<br>Birth<br>s | Still<br>Birth<br>s | Spontaneo<br>us<br>Abortion/<br>Miscarriag<br>e | Elective<br>Abortio<br>ns | Therapeut ic Abortions | Major<br>Congenita<br>I Anomaly<br>with<br>Previous<br>Pregnanc<br>y? |
| xxxxx<br>x | xxx | xxx | xxx | xxx | xxx | XXX | xxx | xxx | xxx | xxx | xxx | xxx | xxx | xxx | Y/N |

Note: Gravida includes the current pregnancy, para events do not.

**Listing 28** 16.2.11.3 Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Y/N | XXX |

Note: Congenital Anomalies are included in the Adverse Event listing.

**Listing 29** 16.2.11.4 Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Day of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord<br>pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XX | XXX | xxxxxxx | Y/N | xxxxxxx | XXX | XXX | XX | Y/N | Y/N | xxxxxxx |

# **Listing 30** 16.2.11.5 Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Day of Initial<br>Report | Fetus Number | Pregnancy<br>Outcome (for this<br>Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|
| XXXXXX | xx | XXX | XXXXX | XXXX | Y/N | xxxxxxx |

**Appendix IV: Clinical Lab Reference Ranges** 

| Site | Test | Sex | Age (yrs) | Lower<br>Limit | Upper<br>Limit | Units |
|---|---|---|---|---|---|---|
| Cincinnati Children's Hospital | Alanine Aminotransferase | Female | All | 12 | 78 | U/L |
| Cincinnati Children's Hospital | Aspartate Aminotransferase | Female | All | 9 | 37 | U/L |
| Cincinnati Children's Hospital | Bilirubin | Both | All | 0.1 | 1.1 | mg/dL |
| Cincinnati Children's Hospital | Creatinine | Female | All | 0.51 | 0.95 | mg/dL |
| Cincinnati Children's Hospital | Glucose | Female | All | 65 | 106 | mg/dL |
| Cincinnati Children's Hospital | Hemoglobin | Female | All | 11.7 | 15.7 | g/dL |
| Cincinnati Children's Hospital | Neutrophils | Both | 10 - 20 | 1.8 | 8 | 10 <sup>9</sup> /L |
| Cincinnati Children's Hospital | Neutrophils | Both | 21+ | 1.8 | 7.7 | 10 <sup>9</sup> /L |
| Cincinnati Children's Hospital | Platelets | Both | All | 135 | 466 | 10 <sup>9</sup> /L |
| Cincinnati Children's Hospital | White Blood Cell Counts | Both | 16 - 20 | 4.5 | 13 | 10 <sup>9</sup> /L |
| Cincinnati Children's Hospital | White Blood Cell Counts | Both | 21+ | 4.5 | 11 | 10 <sup>9</sup> /L |
| University of Iowa | Alanine Aminotransferase | Female | 10 - 18 | 5 | 20 | U/L |
| University of Iowa | Alanine Aminotransferase | Female | 19+ | 0 | 33 | U/L |
| University of Iowa | Aspartate Aminotransferase | Both | 13 - 18 | 10 | 35 | U/L |
| University of Iowa | Aspartate Aminotransferase | Female | 19+ | 0 | 32 | U/L |
| University of Iowa | Bilirubin | Both | 18+ | | 1.2 | mg/dL |
| University of Iowa | Creatinine | Female | 16+ | 0.5 | 1 | mg/dL |
| University of Iowa | Glucose | Both | All | 65 | 99 | mg/dL |
| University of Iowa | Hemoglobin | Female | 18+ | 11.9 | 15.5 | g/dL |
| University of Iowa | Neutrophils | Both | 5 - 18 | 1.7 | 7.5 | 10 <sup>9</sup> /L |
| University of Iowa | Neutrophils | Both | 19+ | 2.188 | 7.8 | 10 <sup>9</sup> /L |
| University of Iowa | Platelets | Both | All | 150 | 400 | 10 <sup>9</sup> /L |
| University of Iowa | White Blood Cell Counts | Both | 18+ | 3.7 | 10.5 | 10 <sup>9</sup> /L |
| Duke University | Alanine Aminotransferase | Female | 12+ | 14 | 54 | U/L |
| Duke University | Aspartate Aminotransferase | Female | 2+ | 15 | 41 | mg/dL |
| Duke University | Bilirubin | Female | All | 0.4 | 1.5 | mg/dL |
| Duke University | Creatinine | Female | 16+ | 0.4 | 1.0 | mg/dL |
| Duke University | Glucose | Female | All | 70 | 140 | mg/dL |
| Duke University | Hemoglobin | Female | 12-18 | 12.0 | 16.0 | g/dL |
| Duke University | Hemoglobin | Female | 19+ | 12.0 | 15.5 | g/dL |
| Duke University | Neutrophils | Female | 12-18 | 1.8 | 7.2 | 10 <sup>9</sup> /L |
| Duke University | Neutrophils | Female | 19+ | 2.0 | 8.6 | 10 <sup>9</sup> /L |
| Duke University | Platelets | Female | 12-18 | 150 | 400 | 10 <sup>9</sup> /L |
| Duke University | Platelets | Female | 19+ | 150 | 450 | 10 <sup>9</sup> /L |
| Duke University | White Blood Cell Counts | Female | 18+ | 3.2 | 9.8 | 10 <sup>9</sup> /L |